CLINICAL TRIAL: NCT01972841
Title: A Randomized, Double-Blind, Parallel-Group, Placebo- and Active-Controlled, Multi-center Study to Evaluate the Efficacy, Safety and Tolerability of Combinations of Solifenacin Succinate and Mirabegron Compared to Solifenacin Succinate and Mirabegron Monotherapy in the Treatment of Overactive Bladder
Brief Title: This Was a Multinational Study Comparing the Efficacy and Safety of Two Medicines , Solifenacin Succinate and Mirabegron Taken Together, or Separately, or a Mock Treatment (Placebo) in Subjects With Symptoms of Overactive Bladder
Acronym: SYNERGY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 178-CL-101; 2012-005735-91 (EudraCT Number); U1111-1153-9095 (Other: World Health Organization)
Record Dates: First submitted 2013-10-25; First posted 2013-10-31 (Estimated); Results first posted 2018-06-12 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Urinary Bladder Overactive; Urinary Bladder Diseases\Urologic Diseases; Overactive Bladder; Urgency Incontinence
Keywords: Combination Therapy; Mirabegron; Overactive Bladder; Urgency; Urinary Incontinence; Nocturia; Solifenacin Succinate
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence; Nocturia | interventions — Solifenacin Succinate; mirabegron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1: Solifenacin 5 mg + Mirabegron 25 mg (Experimental): Participants who received solifenacin 5 mg and mirabegron 25 mg once a day for 12 weeks.
  Interventions: Drug: Solifenacin succinate; Drug: Mirabegron; Drug: Placebo to match mirabegron
- 2: Solifenacin 5 mg + Mirabegron 50 mg (Experimental): Participants who received solifenacin 5 mg and mirabegron 50 mg once a day for 12 weeks.
  Interventions: Drug: Solifenacin succinate; Drug: Mirabegron; Drug: Placebo to match mirabegron
- 3: Placebo (Placebo Comparator): Participants who received matching placebo once a day for 12 weeks.
  Interventions: Drug: Placebo to match solifenacin succinate; Drug: Placebo to match mirabegron
- 4: Solifenacin 5 mg (Active Comparator): Participants who received solifenacin 5 mg once a day for 12 weeks.
  Interventions: Drug: Solifenacin succinate; Drug: Placebo to match mirabegron
- 5:Mirabegron 25 mg (Active Comparator): Participants who received mirabegron 25 mg once a day for 12 weeks.
  Interventions: Drug: Mirabegron; Drug: Placebo to match solifenacin succinate; Drug: Placebo to match mirabegron
- 6: Mirabegron 50 mg (Active Comparator): Participants who received mirabegron 50 mg once a day for 12 weeks.
  Interventions: Drug: Mirabegron; Drug: Placebo to match solifenacin succinate; Drug: Placebo to match mirabegron

INTERVENTIONS:
Drug: Solifenacin succinate — Oral tablet
  Other Names: Vesikur; Vesitrim; YM905; Vesicare
  Arms: 1: Solifenacin 5 mg + Mirabegron 25 mg; 2: Solifenacin 5 mg + Mirabegron 50 mg; 4: Solifenacin 5 mg
Drug: Mirabegron — Oral tablet
  Other Names: YM178; Betmiga; Betanis; Myrbetriq
  Arms: 1: Solifenacin 5 mg + Mirabegron 25 mg; 2: Solifenacin 5 mg + Mirabegron 50 mg; 5:Mirabegron 25 mg; 6: Mirabegron 50 mg
Drug: Placebo to match solifenacin succinate — Oral tablet
  Arms: 3: Placebo; 5:Mirabegron 25 mg; 6: Mirabegron 50 mg
Drug: Placebo to match mirabegron — Oral tablet

SUMMARY:
The purpose of this study was to examine how well two medicines (solifenacin succinate and mirabegron) combined work compared to each medicine alone in the treatment of bladder problems.

ELIGIBILITY:
Inclusion Criteria:

* Subject was willing and able to complete the micturition diary and questionnaires correctly and able to measure his/her vital signs at home at stipulated time points, using the device provided by the study personnel, and to adequately record the readings;
* Subject had symptoms of "wet" OAB (urinary frequency and urgency with incontinence) for at least 3 months;

Exclusion Criteria:

* Subject had significant PVR volume (> 150 mL);
* Subject had a neurological cause for detrusor overactivity (e.g. neurogenic bladder, diabetic neuropathy with autonomic component or bladder involvement, or systemic or central neurological disease such as multiple sclerosis and Parkinson's disease with autonomic component or bladder involvement). An autonomic component could be inferred when autonomic functions were affected, including heart rate, blood pressure, perspiration and digestion.
* Subject had an indwelling catheter or practices intermittent self catheterization.
* Subject had chronic inflammation such as bladder pain syndrome /interstitial cystitis, symptomatic bladder stones or any previous or current radiation cystitis.
* Subject had received intravesical treatment in the past 12 months with e.g., botulinum toxin, resiniferatoxin, capsaicin.
* Subject had moderate to severe hepatic impairment
* Subject had severe renal impairment
* Subject had a clinically significant abnormal ECG
* Subject had a concurrent malignancy or history of cancer (except noninvasive skin cancer) within the last 5 years prior to screening.
* Subject had an average QTcF interval > 450 ms for males or > 470 ms for females based on the triplicate ECGs completed at Screening or is at risk of QT prolongation (e.g., family history of long QT syndrome, hypokalaemia).
* Subject had severe hypertension, which is defined as a sitting average systolic blood pressure ≥ 180 mmHg and/or average diastolic blood pressure ≥ 110 mmHg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3527 (Actual)
Dates: Start 2013-11-05 (Actual); Primary Completion 2015-10-22 (Actual); Study Completion 2015-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Europe B.V.
Locations (435):
- United States (121):
  - Site US10049 Coastal Clinical Research, Inc., Mobile, Alabama
  - Site US10112 TFI, LLC, Mobile, Alabama
  - Site US10104 Clinical Research Advantage, Inc., Chandler, Arizona
  - Site US10021 Beach Clinical Studies, Phoenix, Arizona
  - Site US10122 Orange County Research Institute, Anaheim, California
  - Site US10098 Skyline Research, Cerritos, California
  - Site US10539 Citrus Valley Medical Research, Glendora, California
  - Site US10082 American Clinical Trials, Hawaiian Gardens, California
  - Site US10132 Axis Clinical Trials, Los Angeles, California
  - Site US10133 Axis Clinical Trials, Los Angeles, California
  - Site US10536 Stanford School of Medicine, Palo Alto, California
  - Site US10149 Bayview Research Group, Paramount, California
  - Site US10559 UC Davis Medical Center, Sacramento, California
  - Site US10003 San Diego Clinical Trials, San Diego, California
  - Site US10545 San Diego Institute for Sexual Medicine, San Diego, California
  - Site US10106 West Coast Clinical Research, Tarzana, California
  - Site US10595 Bayview Research Group, Valley Village, California
  - Site US10034 Urology Center of Colorado, Denver, Colorado
  - Site US10070 Physicians' Research Options/Red Rocks OB/GYN, Lakewood, Colorado
  - Site US10053 Western Clinical Research, Inc., Wheat Ridge, Colorado
  - Site US10128 Clinical Research Center of CT, Danbury, Connecticut
  - Site US10018 Grove Hill Clinical Research, New Britain, Connecticut
  - Site US10170 Yale - New Haven Hospital West Haven VAMC, New Haven, Connecticut
  - Site US10123 Chase Medical Research, LLC, Waterbury, Connecticut
  - Site US10060 Meridien Research, Bradenton, Florida
  - Site US10097 A.G.A. Clinical Trials DBA Neostart Group, Hialeah, Florida
  - Site US10148 Best Quality Research, Inc., Hialeah, Florida
  - Site US10153 Palmetto Professional Research, Hialeah, Florida
  - Site US10159 Urological Research Network, Hialeah, Florida
  - Site US10534 South Florida Medical Research, Hialeah, Florida
  - Site US10535 South Florida Medical Research, Homestead, Florida
  - Site US10165 East Coast Institute for Research, Jacksonville, Florida
  - Site US10091 Health Awareness, Jupiter, Florida
  - Site US10150 Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Site US10158 Renstar Medical Research, Ocala, Florida
  - Site US10124 Winter Park Urology Associates, Orlando, Florida
  - Site US10134 Compass Research, LLC, Orlando, Florida
  - Site US10009 South Broward Research, Pembroke Pines, Florida
  - Site US10540 Demaur Clinical Research, INC, Pembroke Pines, Florida
  - Site US10554 Private Practice, Plantation, Florida
  - Site US10095 Florida Urology Specialists, Sarasota, Florida
  - Site US10010 Southeastern Research Group, Inc, Tallahassee, Florida
  - Site US10014 Private Practice, Wellington, Florida
  - Site US10037 Atlanta Medical Research Institute, Alpharetta, Georgia
  - Site US10127 Perimeter North Medical Research, Inc., Roswell, Georgia
  - Site US10120 WR-Mount Vernon Clinical Research, Sandy Springs, Georgia
  - Site US10024 GTC Research, Shawnee Mission, Kansas
  - Site US10078 Heartland Research Associates, LLC, Wichita, Kansas
  - Site US10088 Centex Studies, Inc., Lake Charles, Louisiana
  - Site US10074 Medpharmics, LLC, Metairie, Louisiana
  - Site US10025 Regional Urology, LLC, Shreveport, Louisiana
  - Site US10558 Chesapeake Urology Research Associates, Glen Burnie, Maryland
  - Site US10560 Chesapeake Urology Research Associates, Owings Mills, Maryland
  - Site US10282 Boston Clinical Trials, Boston, Massachusetts
  - Site US10114 Bay State Clinical Trials, Inc., Watertown, Massachusetts
  - Site US10152 Female Pelvic Medicine & Urogynecology Institute, Grand Rapids, Michigan
  - Site US10542 Adult & Pediatric Urology Group, Sartell, Minnesota
  - Site US10110 Montana Health Research Institute, Inc., Billings, Montana
  - Site US10154 Montana Medical Research Inc, Missoula, Montana
  - Site US10553 Women's Clinic of Lincoln, Lincoln, Nebraska
  - Site US10140 IVCTLV, Las Vegas, Nevada
  - Site US10002 Urology Center Research Institute, Englewood, New Jersey
  - Site US10051 AdvancedMed Research, Lawrenceville, New Jersey
  - Site US10047 Lawrence OBGYN Associates, Lawrenceville, New Jersey
  - Site US10162 Phoenix OB-GYN Associates, LLC, Moorestown, New Jersey
  - Site US10011 Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - Site US10015 Urology Group of New Mexico, Albuquerque, New Mexico
  - Site US10077 Northeast Urogynecology, Albany, New York
  - Site US10089 Maimonides Medical Center, Brooklyn, New York
  - Site US10026 AccuMed Research Associates, Garden City, New York
  - Site US10040 Premier Medical Group Of The Hudson Valley, Kingston, New York
  - Site US10073 Manhattan Medical Research Practice, PLLC, New York, New York
  - Site US10249 New York Clinical Trials, New York, New York
  - Site US10168 Weill Cornell Medical College, New York, New York
  - Site US10126 Premier Medical Group, Newburgh, New York
  - Site US10028 Premier Medical Group of the Hudson Valley, Poughkeepsie, New York
  - Site US10593 Upstate Clinical Research Associates LLC, Williamsville, New York
  - Site US10076 Carolina Clinical Trials, Concord, North Carolina
  - Site US10129 PMG Research of Raleigh, Raleigh, North Carolina
  - Site US10549 Associated Urologists of North Carolina, Raleigh, North Carolina
  - Site US10062 Piedmont Medical Research, Winston-Salem, North Carolina
  - Site US10050 Rapid Medical Research, Inc., Cleveland, Ohio
  - Site US10033 Ohio Clinical Research, Lyndhurst, Ohio
  - Site US10067 Family Practice Center of Wadsworth, Wadsworth, Ohio
  - Site US10551 The Christ Hospital, West Chester, Ohio
  - Site US10109 Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Site US10541 Sunstone Medical Research, Medford, Oregon
  - Site US10008 Urologic Consultants of Southeastern Pennsylvania, Bala-Cynwyd, Pennsylvania
  - Site US10045 Lancaster Urology, Lancaster, Pennsylvania
  - Site US10017 Philadelphia Clinical Research, LLC, Philadelphia, Pennsylvania
  - Site US10167 University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Site US10250 Preferred Primary Care Physicians Inc., Pittsburgh, Pennsylvania
  - Site US10248 Preferred Primary Care Physicians, Inc, Pittsburgh, Pennsylvania
  - Site US10063 Preferred Primary Care Physician Research, Uniontown, Pennsylvania
  - Site US10012 Advanced Clinical Concepts, West Reading, Pennsylvania
  - Site US10166 Medical University of South Carolina, Charleston, South Carolina
  - Site US10094 University Medical Group, Greer, South Carolina
  - Site US10046 Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Site US10079 PMG Research of Charleston, LLC, Mt. Pleasant, South Carolina
  - Site US10117 Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Site US10023 Hillcrest Clinical Research, LLC, Simpsonville, South Carolina
  - Site US10101 Palmetto Clinical Research, Summerville, South Carolina
  - Site US10006 Holston Medical Group, Kingsport, Tennessee
  - Site US10084 Dynamed Clinical Research of Austin,LLC dba DM Clinical Resc, Austin, Texas
  - Site US10066 Texas Urology PA, Carrollton, Texas
  - Site US10065 Advanced Research Associates, Corpus Christi, Texas
  - Site US10085 Centex Studies, Inc., Houston, Texas
  - Site US10108 Clinical Trial Network, Houston, Texas
  - Site US10219 Methodist Urology Associates, Houston, Texas
  - Site US10093 Pioneer Research Solutions, Inc., Houston, Texas
  - Site US10090 Protenium Clinical Research, LLC, Hurst, Texas
  - Site US10105 Clinical Trials of Texas, San Antonio, Texas
  - Site US10111 Clinical Trials of Texas, San Antonio, Texas
  - Site US10092 Physicians' Research Options/Salt Lake Women's Center, Sandy City, Utah
  - Site US10032 National Clinical Research Inc., Richmond, Virginia
  - Site US10064 The Group for Women, Virginia Beach, Virginia
  - Site US10083 Urology of Virginia, PLLC., Virginia Beach, Virginia
  - Site US10013 Seattle Urology Research Center, Burien, Washington
  - Site US10004 Integrity Medical Research, LLC, Mountlake Terrace, Washington
  - Site US10155 Seattle Women's Health, Research, Gynecology, Seattle, Washington
  - Site US10135 Walla Walla Clinic, Walla Walla, Washington
- Argentina (5):
  - Site AR54005 IUBA - Instituto Urologico de Buenos Aires, Buenos Aires
  - Site AR54003 Hospital Italiano de Buenos Aires, Buenos Aires
  - Site AR54006 Hospital Italiano de Buenos Aires, Buenos Aires
  - Site AR54001 CDU - Centro de Urología, Ciudad Autónoma Buenos Aires
  - Site AR54004 Instituto de Investigaciones Clnicas Rosario, Rosario Provincia de Santa Fe
- Australia (15):
  - Site AU61026 Ballarat Urology, Ballarat
  - Site AU61022 Brisbane South Clinical Research Centre, Brisbane
  - Site AU61005 Hunter Clinical Research, Broadmeadow
  - Site AU61015 Repatriation General Hospital, Daw Park
  - Site AU61025 Western Health, Footscray
  - Site AU61012 Cabrini Hospital, Malvern
  - Site AU61010 Nambour General Hospital, Nambour
  - Site AU61002 The Royal Womens Hospital, Parkville
  - Site AU61004 Keogh Institute for Medical Research, Perth
  - Site AU61007 Prince of Wales Hospital, Randwick
  - Site AU61008 Epworth Healthcare, Richmond
  - Site AU61019 AusTrialsSherwood, Sherwood
  - Site AU61017 Healthpac Medical Centre, Sydney
  - Site AU61021 Royal Hospital for Women, Sydney
  - Site AU61011 Illawarra Health and Medical Research Institute, Wollongong
- Belgium (4):
  - Site BE32004 Gent University Hospital, Ghent
  - Site BE32011 Universitaire Ziekenhuizen Leuven, Leuven
  - Site BE32014 Hart Ziekenhuis, Roeselare
  - Site BE32012 Sint-Trudo Ziekenhuis, Campus Sint Jozef/Sint-Anna, Sint-Truiden
- Bulgaria (7):
  - Site BG35904 University Hospital (UMHAT) - George Stranski, Pleven
  - Site BG35908 MHAT Plovdiv AD, Plovdiv
  - Site BG35902 MHAT Ruse, Rousse
  - Site BG35905 MHAT Alexandrovska Hospital, Sofia
  - Site BG35903 MHATEM Pirogov, Sofia
  - Site BG35906 UMHAT Varna, Varna
  - Site BG35910 MHAT, Veliko Tarnovo
- Canada (26):
  - Site CA15029 Royal Alexandra Hospital, Edmonton, Alberta
  - Site CA15035 Glenrose Rehabilitation Hospital, Edmonton, Alberta
  - Site CA15033 Prohealth, Vancouver, British Columbia
  - Site CA15008 Private Practice, Saint John, New Brunswick
  - Site CA15001 The Male/Female Health & Research Centre, Barrie, Ontario
  - Site CA15006 Bramalea Medical Centre, Brampton, Ontario
  - Site CA15003 Brantford Urology Research, Brantford, Ontario
  - Site CA15042 G. Kenneth Jansz Medicine Professional Corporation, Burlington, Ontario
  - Site CA15044 McMaster Institute of Urology, Hamilton, Ontario
  - Site CA15031 Centre for Applied Urology Research (CAUR), Kingston, Ontario
  - Site CA15007 Eunoia2 Incorporated, Kitchener, Ontario
  - Site CA15034 Oxford/Richmond Medical, London, Ontario
  - Site CA15032 Stanley Flax Medical Prof Corp, North York, Ontario
  - Site CA15013 Sunnybrook Health Sciences Center, Toronto, Ontario
  - Site CA15004 Primehealth Clinical Research, Toronto, Ontario
  - Site CA15002 Toronto Western Hospital, Toronto, Ontario
  - Site CA15026 Rhodin Recherche Clinique, Drummondville, Quebec
  - Site CA15015 Recherches Cliniques Theradev, Inc., Granby, Quebec
  - Site CA15021 Urology South Shore Research, Greenfield Park, Quebec
  - Site CA15030 UroLaval, Laval, Quebec
  - Site CA15040 RechercheGCP Research, Montreal, Quebec
  - Site CA15020 Diex Research Montreal, Montreal, Quebec
  - Site CA15010 Ultra Med Research, Inc., Point-Claire, Quebec
  - Site CA15025 Clinique RSF Inc., Québec, Quebec
  - Site CA15039 Pro-recherche, Saint Romuald, Quebec
  - Site CA15027 Diex Research Sherbrooke Inc, Sherbrooke, Quebec
- China (22):
  - Site CN86017 Affiliated Union Hospital of Fujian Medical Uni., Fuzhou, Fujian
  - Site CN86025 Beijing Friendship Hospital, Beijing
  - Site CN86009 Peking University 3rd Hospital, Beijing
  - Site CN86013 Beijing Hospital, Beijing
  - Site CN86014 The First Hospital Bethune of Jilin University, Changchun
  - Site CN86002 Changsha Central Hospital, Changsha
  - Site CN86028 General Hospital of Chengdu Military Region of PLA, Chengdu
  - Site CN86029 Southwest Hospital (Chongqing), Chongqing
  - Site CN86016 Guangzhou First People's Hospital, Guangzhou
  - Site CN86027 Second Hospital of Lanzhou University, Lanzhou
  - Site CN86030 Lanzhou University First Hospital, Lanzhou
  - Site CN86020 The First Affiliated Hospital of NanChang Univers, Nanchang
  - Site CN86023 Nanjing First Hospital, Nanjing
  - Site CN86021 HuaDong Hosipital Affiliated to Fudan University, Shanghai
  - Site CN86003 Shanghai Renji Hospital, Shanghai
  - Site CN86012 The Fifth People's Hospital of Shanghai, Shanghai
  - Site CN86011 The Second Affiliated Hospital of Soochow Universi, Suzhou
  - Site CN86010 1st Affiliated Hosptital of Suchow University, Suzhou
  - Site CN86026 The First Affiliated Hospital of Wenzhou Medical C, Wenzhou
  - Site CN86022 Tongji Hospital, Tongji Medical College of Hust, Wuhan
  - Site CN86015 Zhongnan Hospital of Wuhan University, Wuhan
  - Site CN86018 Wuxi People's Hospital, Wuxi
- Colombia (2):
  - Site CO57003 Hospital Pablo Tobón Uribe, Medellín, Antioquia
  - Site CO57004 Instituto de Coloproctologia ICO SAS, Medellín
- Czechia (12):
  - Site CZ42015 Centrum ambulantni gynekologie a primarni pece, Brno
  - Site CZ42003 SANUS, Hradec Králové
  - Site CZ42001 Fakultni Nemocnice Hradec Kralove, Hradec Králové
  - Site CZ42002 Hospital Jihlava, Jihlava
  - Site CZ42011 Hospital Novy Jicin, Nový Jičín
  - Site CZ42010 G-centrum Olomouc S.R.O., Olomouc
  - Site CZ42014 Private Practice, Ostrava
  - Site CZ42005 Research Site s.r.o., Pilsen
  - Site CZ42007 Uro-Santé/Nová Brumlovka, Prague
  - Site CZ42013 Urology Clinic, Sternberk
  - Site CZ42009 Hospital Uherské Hradiště a.s., Uherské Hradiště
  - Site CZ42006 Private Practice, Ústí nad Labem
- Denmark (2):
  - Site DK45012 Aalborg Sygehus Nord, Aalborg
  - Site DK45013 University Hospital of Aarhus, Skejby, Aarhus
- Estonia (3):
  - Site EE37201 Parnu Hospital, Pärnu
  - Site EE37205 West Tallinn Central Hospital, Tallinn
  - Site EE37202 Tartu University Hospital, Tartu
- Finland (3):
  - Site FI35801 Kouvolan Lääkäriasema, Kouvola
  - Site FI35803 Oulu University Hospital, Oulu
  - Site FI35802 Meilahti Hospital, Vantaa
- France (10):
  - Site FR33007 Centre Hospitalier Louis Pasteur, Colmar
  - Site FR33010 CHU Hopital du Bocage, Dijon
  - Site FR33008 CHU Nantes, Nantes
  - Site FR33002 CHU Carémeau, Nîmes
  - Site FR33013 Hopital Saint Louis, Paris
  - Site FR33001 Hopital Tenon, Paris
  - Site FR33024 Hopital Tenon, Paris
  - Site FR33011 Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Site FR33012 Hopital Foch, Suresnes
  - Site FR33005 Hopital Bretonneau, Tours
- Germany (13):
  - Site DE49008 Private Practice, Bad Ems
  - Site DE49031 Urologisches Zentrum Refrath, Bergisch Gladbach
  - Site DE49033 Universitsy Clinic Bonn, Bonn
  - Site DE49002 Private Practice, Duisburg
  - Site DE49032 Urologicum Duisburg, Duisburg
  - Site DE49003 Private Practice, Eisleben Lutherstadt
  - Site DE49010 Private Practice, Ganderkesee
  - Site DE49011 Private Practice, Halle
  - Site DE49013 Private Practice, Leipzig
  - Site DE49034 LMU Muenchen, Munich
  - Site DE49001 Private Practice, Neustadt in Sachsen
  - Site DE49026 Zentrum fuer Onkologie und Urologie Rostock, Rostock
  - Site DE49014 Private Practice, Sangerhausen
- Site GR30009 Aretaieio/Maginio, Athens, Greece
- Hong Kong (3):
  - Site HK85204 The Chinese Uni of HK, Prince of Wales Hospital, Hong Kong
  - Site HK85201 Kwong Wah Hospital, Kowloon
  - Site HK85203 The Chinese Uni of HK, Prince of Wales Hospital, Shatin
- Hungary (6):
  - Site HU36003 Dr.Szarka Ödön Kistérségi Egészségügyi Szolgáltató Kft, Csongrád
  - Site HU36007 Mediroyal Prevention Center, Kecskemét
  - Site HU36005 Uro-clin Ltd, Pécs
  - Site HU36013 Sopron Erzsébet Hospital, Sopron
  - Site HU36001 Donatella 99BT, Szentes
  - Site HU36012 Veszprém County Cholnoky Ferenc Hospital, Veszprém
- Italy (5):
  - Site IT39022 Azienda Ospedale Umberto I (Ancona), Ancona
  - Site IT39007 Azienda Ospedaliera San Giuseppe Moscati, Avellino
  - Site IT39001 U.O. Dip. di Neuro-Urologia; Univ. di Roma La Sapienza, Latina
  - Site IT39003 Ospedale San Raffaele, Milan
  - Site IT39020 Ospedale San Raffaele IRCCS, U.O. di Ginecologia e Ostetricia, Unità Funzionale di Uroginecologia, Milan
- Latvia (3):
  - Site LV37102 Private Practice, Liepāja
  - Site LV37103 Health Centre "Olaine", Olaine
  - Site LV37105 P.Stradins Clinical University Hospital, Riga
- Lithuania (9):
  - Site LT37008 Kaunas 2nd Clinical Hospital, Kaunas
  - Site LT37004 KHospital of Lithuanian University of Health Science, Kaunas
  - Site LT37011 Saules Family Medicine Centre, Kaunas
  - Site LT37012 Klaipeda University Hospital, Klaipėda
  - Site LT37005 Public Institution Vilnius City University Hospital, Vilnius
  - Site LT37010 Public Institution Vilnius City University Hospital, Vilnius
  - Site LT37003 Family Medical Centre Seimos gydytojas, Vilnius
  - Site LT37007 Vilnius University Hospital Santariskiu Klinikos, Vilnius
  - Site LT37009 Clinics Privatus gydytojas, Vilnius
- Malaysia (6):
  - Site MY60006 Hospital Pulau Pinang, George Town
  - Site MY60001 Hospital Kuala Lumpur, Kuala Lumpur
  - Site MY60004 University Malaya Medical Centre, Kuala Lumpur
  - Site MY60005 Universiti Kebangsaan Malaysia Medical Centre, Kuala Lumpur
  - Site MY60003 Hospital Ummum Sarawak, Kuching
  - Site MY60002 Sime Darby Medical Centre, Petaling Jaya
- Mexico (4):
  - Site MX52004 Consultorio de Especialidad en Urologia, Durango
  - Site MX52001 Centro de Investigacin Basica y Clnica, Guadalajara
  - Site MX52003 Clinstile, Sociedad Anonima de Capital Variable, Mexico City
  - Site MX52002 Accelerium Clinical Research/ Hospital San Jorge, Monterrey
- Netherlands (5):
  - Site NL31002 Academic Medical Center (AMC), Amsterdam
  - Site NL31006 Medisch Spectrum Twente, Enschede
  - Site NL31005 Canisius-Wilhelmina Ziekenhuis, Nijmegen
  - Site NL31010 Antonius Ziekenhuis Sneek, Sneek
  - Site NL31001 University Medical Centre Utrecht, Utrecht
- New Zealand (6):
  - Site NZ64004 John A Tuckey Ltd Ascot Central, Auckland
  - Site NZ64001 Canterbury Urology Research Trust, Christchurch
  - Site NZ64005 Waikato Urology Research Limited, Hamilton
  - Site NZ64002 Roundhay Medical Centre, Nelson
  - Site NZ64003 Tauranga Urology Research Ltd, Tauranga
  - Site NZ64006 Cardinal Point Specialist Centre, Whangarei
- Norway (3):
  - Site NO47007 Medi3 Clinic AS, Ålesund, Ålesund
  - Site NO47006 M3 Helse AS, Hamar
  - Site NO47008 Norsk Helseklinikk (Heiaklinikken), Lierskogen
- Peru (6):
  - Site PE51006 Hospital Nacional Guillermo Almenara Irigoyen EsSalud, La Victoria, Lima region
  - Site PE51007 Clínica Anglo Americana, San Isidro, Lima region
  - Site PE51001 Instituto de Ginecologia y Reproduccion, Lima
  - Site PE51002 Clinica San Borja, Lima
  - Site PE51004 Clinica San Pablo, Lima
  - Site PE51005 Hospital Nacional Hipolito Unanue, Lima
- Philippines (6):
  - Site PH63008 Dr. Pablo O. Torre Memorial Hospital, Bacolod City
  - Site PH63005 Davao Doctor's Hospital, Davao City
  - Site PH63010 Davao Doctor's Hospital, Davao City
  - Site PH63003 University of Santo Tomas Hospital (USTH), Manila
  - Site PH63009 Chinese General Hospital and Medical Center, Manila
  - Site PH63004 East Avenue Medical Center, Quezon City
- Poland (12):
  - Site PL48018 Gastromed, Bialystok
  - Site PL48013 Urovita Ltd., Chorzów
  - Site PL48014 Synexus Polska, Gdynia
  - Site PL48004 NZOZ Szpital Sw.Rodziny Centrum Medyczne, Lodz
  - Site PL48010 Nzoz Novita, Lublin
  - Site PL48011 Nzoz Centrum Urologiczne sp. z o.o., Mysłowice
  - Site PL48016 Prywatny Gabinet Urologiczny, Opole
  - Site PL48005 HEUREKA Hanna Szalecka, Piaseczno
  - Site PL48012 Military Institute of Medicine, Warsaw
  - Site PL48003 CSKMSW, Warsaw
  - Site PL48001 Specjalistyczny Gabinet Lekarski, Warsaw
  - Site PL48019 Synexus Polska sp. z o. o., Wroclaw
- Romania (8):
  - Site RO40015 Spitaul Clinic Judetean de Urgenta Brasov, Brasov
  - Site RO40004 Spitalul Clinic de Urgenta Sfantul Ioan, Bucharest
  - Site RO40001 Spiatlul Clinic Th. Burghele, Bucharest
  - Site RO40005 Spiatlul Clinic Th. Burghele, Bucharest
  - Site RO40014 E-URO Cabinet, Cluj-Napoca
  - Site RO40007 Spital Clinic, Iași
  - Site RO40010 Spitalul Clinic Judetan de Urgenta Sibiu, Sibiu
  - Site RO40002 Spitalul Clinic Judetean de Urgenta Timisoara, Timișoara
- Russia (7):
  - Site RU70015 LLC Clinical Research Medical Complex, Kazan'
  - Site RU70023 Penza Regional Clinical Hospatal n. a. N.N. Burdenko, Penza
  - Site RU70019 City Multidisciplinary Hospital No. 2, Saint Petersburg
  - Site RU70002 Pavlov St. Petersburg State Medical University, Saint Petersburg
  - Site RU70022 St. Petersburg State Public Health Institution, Saint Petersburg
  - Site RU70014 OOO Hospital Orkli, Saint Petersburg
  - Site RU70018 Bashkirsky State Medical University of Roszdrav, Ufa
- Singapore (3):
  - Site SG65001 National University Hospital, Singapore
  - Site SG65002 Singapore General Hospital, Singapore
  - Site SG65003 KK Women's and Children's Hospital, Singapore
- Slovakia (8):
  - Site SK42105 Ruzinovska poliklinika a.s., Bratislava
  - Site SK42107 Zeleznicne zdravotnictvo Kosice, s.r.o., Košice
  - Site SK42101 Andrologicka a Urologicka Ambulancia, Košice
  - Site SK42103 UroExam s.r.o., Nitra
  - Site SK42108 BrenCare, s. r. o., Poprad
  - Site SK42104 Urology Outpatient Department, Prešov
  - Site SK42106 Private Urological Care Center, Trenčín
  - Site SK42102 CeGys, s.r.o., Trenčín
- Slovenia (2):
  - Site SI38604 General Hospital Murska Sobota, Murska Sobota
  - Site SI38602 General Hospital Novo Mesto, Novo Mesto
- South Africa (6):
  - Site ZA27005 Grootte Schuur Hospital, Cape Town
  - Site ZA27001 Private Practice, Centurion
  - Site ZA27006 Parklands Hospital, Durban
  - Site ZA27013 Synexus Clinical Research SA (Pty) Ltd, Meyerspark
  - Site ZA27007 Paarl Medical Centre, Paarl
  - Site ZA27002 Mayo Clinic, Roodepoort
- South Korea (26):
  - Site KR82014 Soon Chun Hyang University Hospital, Bucheon-si
  - Site KR82006 Dong-A University Medical Center, Busan
  - Site KR82016 Pusan National University Hospital, Busan
  - Site KR82024 Chungbuk National University Hospital, Cheongju-si
  - Site KR82032 Kyungpook National University Hospital, Daegu
  - Site KR82005 Yeungnam University Hospital, Daegu
  - Site KR82029 Daegu Catholic Univ. Medical Center, Daegu
  - Site KR82019 Chungnam National University Hospital, Daejeon
  - Site KR82011 Eulji University Hospital, Daejeon
  - Site KR82031 Chonnam National University Hospital, Gwangju
  - Site KR82009 Wonkwang University Hospital, Iksan -Si
  - Site KR82023 Gachon University Gil Hospital, Incheon
  - Site KR82010 Chonbuk National University Hospital, Jeonju
  - Site KR82025 Seoul National University Bundang Hospital, Seongnam-si
  - Site KR82021 Cheil General Hospital & Women's Healthcare Center, Seoul
  - Site KR82020 Seoul National University Hospital, Seoul
  - Site KR82030 Severance Hospital, Seoul
  - Site KR82013 Hallym University Kangdong Sacred Heart Hospital, Seoul
  - Site KR82017 Kyung Hee University Medical Center, Seoul
  - Site KR82002 Samsung Medical Center, Seoul
  - Site KR82008 Gangnam Severance Hospital, Seoul
  - Site KR82015 Korea University Medical Center, Seoul
  - Site KR82001 Seoul Saint Mary's Hospital, Seoul
  - Site KR82003 Asan Medical Center, Seoul
  - Site KR82012 Konkuk University Medical Center, Seoul
  - Site KR82004 Ajou University Hospital, Suwon
- Spain (11):
  - Site ES34010 Hospital del Henares, Coslada
  - Site ES34024 Hospital San Juan de Dios, Esplugues de Llobregat-Barcelo
  - Site ES34001 Hospital Universitario de Getafe, Getafe (Madrid)
  - Site ES34006 Hospital San Rafael, Madrid
  - Site ES34004 Hospital Infanta Leonor, Madrid
  - Site ES34015 Hospital 12 de Octubre, Madrid
  - Site ES34009 Hospital Universitario La Paz, Madrid
  - Site ES34005 Hospital de Fuenlabrada, Madrid
  - Site ES34003 Hospital Universitario Nuestra Señora de Valme, Seville
  - Site ES34007 Hospital Virgen del Rocio, Seville
  - Site ES34002 H. U. Politecnico La Fe, Valencia
- Sweden (9):
  - Site SE46007 Ladulaas Clinical Studies, Borås
  - Site SE46025 Pharmasite, Helsingborg
  - Site SE46005 Center för Läkemedelsstudier, Malmo
  - Site SE46016 Citydiabetes - Stockholm, Stockholm
  - Site SE46008 Bragée Medect AB, Stockholm
  - Site SE46012 Karolinska University Hospital Huddinge, Stockholm
  - Site SE46003 Danderyds Hospital, Stockholm
  - Site SE46009 Encia AB, Uppsala Hälsomottagning, Uppsala
  - Site SE46017 S3 Clinical Research Centers, Vällingby
- Taiwan (4):
  - Site TW88605 Taichung Veteran General Hospital, Taichung
  - Site TW88611 Chung Shan Medical University Hospital, Taichung
  - Site TW88612 Chi Mei Medical Center, Yong Kang, Tainan
  - Site TW88614 Tri-Service General Hospital, Taipei
- Thailand (8):
  - Site TH66002 Chulalongkorn Hospital, Bangkok
  - Site TH66008 Phramongkutklao Hospital, Bangkok
  - Site TH66005 Siriraj Hospital, Bangkok
  - Site TH66010 Maharaj Nakorm Chiangmai Hosp, Chiang Mai
  - Site TH66006 Songklanagarind Hospital, Prince of Songkla University, Hat Yai
  - Site TH66009 Srinagarind Hospital, Khon Kaen
  - Site TH66007 Thammasat University Hospital, Pathum Thani
  - Site TH66011 Ramathibodi Hospital, Ratchathewi
- Turkey (Türkiye) (4):
  - Site TR90019 Ankara University Medical Faculty Ibni Sina Hospital, Ankara
  - Site TR90013 Uludag University Faculty of Medicine, Bursa
  - Site TR90001 Pamukkale University Faculty of Medicine, Denizli
  - Site TR90017 Bilim University Sisli Florence Nightingale Hospital, Istanbul
- Ukraine (10):
  - Site UA38002 City Hospital No 2, Chernihiv
  - Site UA38015 Regional Municipal Institution, Urology Department, Chernivtsi
  - Site UA38013 Dnipropetrovsk State Medical Academy, Mechnikov Dnipropetrov, Dnipropetrovsk
  - Site UA38006 Shapoval Regional Clinical Centre of Urology and Nephrology, Kharkiv
  - Site UA38007 Central Outpatient Hospital of Deanyanskyy Distric, Kiev
  - Site UA38003 Urology Dpt of Kyiv City Clinical Hospital #3, Kyiv
  - Site UA38010 Academy of Medical Sciences of Ukraine, Kyiv
  - Site UA38014 Uzhgorod City Polyclinic, Uzhhorod
  - Site UA38004 Vinnitsa Endocrinology Dispens, Vinnytsia
  - Site UA38008 Medical Academy of Postgraduate Education, Urology Clinic, Zaporizhzhya
- United Kingdom (9):
  - Site GB44009 Sheepcot Medical Centre, Garston, Watfort
  - Site GB44003 Leighton Hospital, Crewe
  - Site GB44021 Medway Hospital, Gillingham
  - Site GB44005 North West London Hosp Menopause Clinic, Harrow
  - Site GB44024 St James's University Hospital, Leeds
  - Site GB44025 Kings College Hospital, London
  - Site GB44006 Derriford Hospital, Plymouth
  - Site GB44022 The Royal Berkshire Hospital, Reading
  - Site GB44001 Royal Hallamshire Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Stoniute A, Madhuvrata P, Still M, Barron-Millar E, Nabi G, Omar MI. Oral anticholinergic drugs versus placebo or no treatment for managing overactive bladder syndrome in adults. Cochrane Database Syst Rev. 2023 May 9;5(5):CD003781. doi: 10.1002/14651858.CD003781.pub3. PMID 37160401
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=254

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who had symptoms of "wet" overactive bladder (OAB) (urgency, urinary frequency and urgency incontinence) for ≥ 3 months were enrolled at 435 centers in 42 countries. Eligible participants went into a single-blind, 4-week placebo run-in period and completed a micturition diary the last 7 days prior to each study visit.
Pre-assignment Details: A total of 6991 participants were screened, 6275 participants received placebo run-in treatment and 3527 participants were randomized into 1 of 6 treatment arms in a 1:1:1:1:2:2 ratio in the 12-week double-blind treatment period. A total of 953 participants were also enrolled in an ambulatory blood pressure monitoring (ABPM) substudy.
Groups:
- Placebo: Participants who received matching placebo once a day for 12 weeks.
- Mirabegron 25 mg: Participants who received mirabegron 25 mg once a day for 12 weeks.
- Mirabegron 50 mg: Participants who received mirabegron 50 mg once a day for 12 weeks.
- Solifenacin 5 mg: Participants who received solifenacin 5 mg once a day for 12 weeks.
- Solifenacin 5 mg + Mirabegron 25 mg: Participants who received solifenacin 5 mg and mirabegron 25 mg once a day for 12 weeks.
- Solifenacin 5 mg + Mirabegron 50 mg: Participants who received solifenacin 5 mg and mirabegron 50 mg once a day for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Started | 447 | 441 | 437 | 434 | 885 | 883
Completed | 404 | 397 | 387 | 397 | 802 | 798
Not Completed | 43 | 44 | 50 | 37 | 83 | 85
Not completed — Randomized but Never Received Treatment | 2 | 5 | 4 | 2 | 6 | 13
Not completed — Adverse Event | 13 | 8 | 12 | 9 | 21 | 26
Not completed — Lack of Efficacy | 1 | 0 | 0 | 2 | 4 | 1
Not completed — Lost to Follow-up | 4 | 2 | 4 | 2 | 9 | 3
Not completed — Protocol Violation | 2 | 2 | 3 | 5 | 9 | 4
Not completed — Withdrawal by participants | 21 | 27 | 23 | 16 | 33 | 34
Not completed — Miscellaneous | 0 | 0 | 4 | 1 | 0 | 4
Not completed — Did not have end of treatment page | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Randomized analysis set (RAS), comprised all randomized patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg | Total
Number analyzed (Participants) | 447 | 441 | 437 | 434 | 885 | 883 | 3527
Age, Continuous [Mean (Standard Deviation); unit: Year] | 57.46 (13.2) | 56.77 (13.46) | 56.69 (13.28) | 57.88 (12.92) | 56.94 (13.78) | 57.3 (13.46) | 57.16 (13.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 345 | 343 | 338 | 342 | 686 | 684 | 2738
  Male | 102 | 98 | 99 | 92 | 199 | 199 | 789
Mean number of incontinence episodes/24 h [Mean (Standard Deviation); unit: incontinence episodes] — An incontinence episode was defined as the complaint of any involuntary leakage of urine. The mean number of incontinence episodes per 24 hours was calculated from data recorded by the participant per day on valid diary days during the 7-day micturition diary period. Population: Full analysis set (FAS) comprised all RAS patients who took ≥ 1 dose of double-blind treatment after randomization, reported ≥ 1 micturition in the baseline diary and ≥ 1 micturition postbaseline, reported ≥ 1 incontinence episode in the baseline diary and excluded participants from one site. Participants with available data were included.
  incontinence episodes
    number analyzed (Participants) | 418 | 409 | 411 | 415 | 827 | 826 | 3306
    (all) | 3.41 (3.37) | 3.42 (3.40) | 3.18 (3.47) | 3.58 (3.51) | 3.22 (3.17) | 3.16 (3.08) | 3.29 (3.29)
Mean number of micturitions/24 h [Mean (Standard Deviation); unit: micturitions] — A micturition was defined as any voluntary micturition (excluding incontinence only episodes). The mean number of micturitions per 24 hours was calculated from data recorded by the participant per day on valid diary days during the 7-day micturition diary period. Population: FAS participants with available data were included in the analysis.
  micturitions
    number analyzed (Participants) | 418 | 409 | 411 | 415 | 827 | 826 | 3306
    (all) | 10.97 (2.86) | 10.81 (2.63) | 11.19 (3.27) | 10.76 (2.47) | 10.73 (2.88) | 10.74 (2.36) | 10.84 (2.73)
Mean volume voided per micturition [Least Squares Mean (Standard Deviation); unit: mL] — The mean volume voided per micturition was calculated from the data recorded by the participant during 3 consecutive days with volume measurements during the 7-day micturition diary period. Population: FAS participants with available data were included in the analysis.
  mL
    number analyzed (Participants) | 414 | 407 | 409 | 413 | 823 | 824 | 3290
    (all) | 157.94 (58.78) | 152.46 (60.96) | 155.31 (60.78) | 151.94 (59.29) | 159.32 (58.29) | 153.57 (59.67) | 155.43 (59.49)
Number of incontinence episodes/week [Mean (Standard Deviation); unit: incontinence episodes] — The number of incontinence episodes was calculated from total number of incontinence episodes recorded by the participant per day on valid diary days during the 7-day micturition diary period. Population: FAS participants with available data were included in the analysis.
  incontinence episodes
    number analyzed (Participants) | 418 | 409 | 411 | 415 | 827 | 826 | 3306
    (all) | 23.6 (23.6) | 23.5 (23.6) | 21.7 (23.8) | 24.8 (24.5) | 22.1 (21.7) | 21.7 (21.3) | 22.7 (22.7)
Mean number of urgency incontinence episodes/24 h [Mean (Standard Deviation); unit: urgency incontinence episodes] — An urgency incontinence episode was defined as the involuntary leakage of urine accompanied by or immediately preceded by urgency. The mean number of urgency incontinence episodes per 24 hours was calculated from number of times a participant recorded an urgency incontinence episode per day on valid diary days during the 7-day micturition diary period prior to each visit. Population: FAS participants with available data were included in the analysis.
  urgency incontinence episodes
    number analyzed (Participants) | 415 | 407 | 405 | 414 | 823 | 822 | 3286
    (all) | 3.14 (3.23) | 3.00 (3.09) | 2.89 (3.31) | 3.23 (3.34) | 2.85 (2.81) | 2.80 (2.64) | 2.94 (3.00)
Number of urgency incontinence episodes/week [Mean (Standard Deviation); unit: urgency incontinence episodes] — The number of urgency incontinence episodes was number of times a participant recorded an urgency incontinence episode on valid diary days during the 7-day micturition diary period prior to each visit. Population: FAS participants with available data were included in the analysis.
  urgency incontinence episodes
    number analyzed (Participants) | 415 | 407 | 405 | 414 | 823 | 822 | 3286
    (all) | 21.7 (22.6) | 20.6 (21.4) | 19.8 (22.7) | 22.4 (23.3) | 19.5 (19.3) | 19.2 (18.2) | 20.3 (20.7)
Mean number of urgency episodes (Grade 3 or 4)/24 h [Mean (Standard Deviation); unit: urgency episodes] — An urgency episode (Grade 3 or 4) was defined as a complaint of a sudden, compelling desire to pass urine, which is difficult to defer; it was recorded when a micturition or incontinence episode was recorded and the severity of urinary urgency recorded was 3 (severe urgency) or 4 (urgency incontinence) according to the Patient Perception of Intensity of Urgency Scale (PPIUS). The mean number of urgency episodes per 24 hours was calculated from data recorded by the participant per day on valid diary days during the 7-day micturition diary period prior to each visit. Population: FAS participants with available data were included in the analysis.
  urgency episodes
    number analyzed (Participants) | 417 | 409 | 411 | 415 | 827 | 826 | 3305
    (all) | 6.52 (4.05) | 6.22 (3.89) | 6.46 (4.88) | 6.48 (3.88) | 6.22 (3.70) | 6.22 (3.56) | 6.32 (3.92)
Mean number of nocturia episodes/24 h [Mean (Standard Deviation); unit: nocturia episodes] — A nocturia episode was defined as waking at night 1 or more times to void (i.e., any voiding associated with sleep disturbance between the time the participant goes to bed with the intention to sleep until the time the patients gets up in the morning with the intention to stay awake). The mean number of nocturia episodes per 24hr was calculated from data recorded by the participant per day on valid diary days during the 7-day micturition diary period prior to each visit. Population: FAS participants with available data were included in the analysis.
  nocturia episodes
    number analyzed (Participants) | 368 | 344 | 356 | 352 | 710 | 704 | 2834
    (all) | 1.57 (1.06) | 1.53 (1.02) | 1.59 (1.09) | 1.59 (0.96) | 1.56 (1.07) | 1.52 (0.97) | 1.56 (1.03)
Number of nocturia episodes/week [Mean (Standard Deviation); unit: nocturia episode] — The number of nocturia episodes was calculated from sun of each nocturia episodes recorded by the participant per day on valid diary days during the 7-day micturition diary period prior to each visit. Population: FAS participants with available data were included in the analysis.
  nocturia episode
    number analyzed (Participants) | 368 | 344 | 356 | 352 | 710 | 704 | 2834
    (all) | 10.9 (7.4) | 10.6 (7.1) | 11.0 (7.6) | 11.0 (6.6) | 10.8 (7.4) | 10.5 (6.7) | 10.8 (7.2)
Mean number of pads used/24 h [Mean (Standard Deviation); unit: pads] — The mean number of pads used per 24 hours was calculated from data recorded by the participant per day on valid diary days during the 7-day micturition diary period prior to each visit. Population: FAS participants with available data were included in the analysis.
  pads
    number analyzed (Participants) | 256 | 252 | 251 | 262 | 513 | 511 | 2045
    (all) | 2.87 (2.99) | 2.86 (2.70) | 2.62 (3.18) | 2.87 (3.14) | 2.50 (2.58) | 2.58 (2.39) | 2.67 (2.76)
Number of pads used/week [Mean (Standard Deviation); unit: pads] — The number of pads used was calculated from sum of each record with a new pad checked on valid diary days during the 7-day micturition diary period prior to each visit. Population: FAS participants with available data were included in the analysis.
  pads
    number analyzed (Participants) | 256 | 252 | 251 | 262 | 513 | 511 | 2045
    (all) | 19.8 (20.9) | 19.6 (18.7) | 17.9 (21.7) | 19.9 (21.8) | 17.1 (17.7) | 17.7 (16.4) | 19.3 (19.0)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to End of Treatment (EoT) in Mean Number of Incontinence Episodes Per 24 Hours
Description: An incontinence episode was defined as the complaint of any involuntary leakage of urine. The mean number of incontinence episodes per 24 hours was calculated from data recorded by the participant per day on valid diary days during the 7-day micturition diary period.
Time Frame: Baseline and EoT (up to 12 weeks)
Population: FAS comprised all RAS patients who took ≥ 1 dose of double-blind treatment after randomization, reported ≥ 1 micturition in the baseline diary and ≥ 1 micturition postbaseline, reported ≥ 1 incontinence episode in the baseline diary and excluded participants from one site. Last observation carried forward (LOCF) was used for EoT.
Measure: Least Squares Mean (Standard Error); unit: incontinence episodes
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 412 | 409 | 406 | 413 | 823 | 816
incontinence episodes | -1.34 (0.10) | -1.70 (0.10) | -1.76 (0.10) | -1.79 (0.10) | -2.04 (0.07) | -1.98 (0.07)
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; Difference of the adjusted mean calculated by subtracting the adjusted mean of the solifenacin 5 mg monotherapy group from the adjusted mean of the combination group (solifenacin 5 mg + mirabegron 25 mg) based on the ANCOVA model with treatment group, sex, age group (< 65, ≥ 65 years), previous overactive bladder medication (yes, no) and geographic region as fixed factors and baseline value as a covariate; Test type: Superiority; p = 0.072, Stratified rank ANCOVA — Nominal p-value; No adjustment for multiplicity was needed for testing combination therapy vs. its 2 monotherapy components; Least squares mean difference = -0.25, 95% CI 2-sided [-0.49 to -0.01], Standard Error of Mean 0.12 — Adjustment for multiplicity across primary and the first secondary endpoint as well as across the 2 combination doses was made using a sequential Bonferroni-based testing procedure
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Difference of the adjusted mean calculated by subtracting the adjusted mean of the solifenacin 5 mg monotherapy group from the adjusted mean of the combination group (solifenacin 5 mg + mirabegron 50 mg) based on the ANCOVA model with treatment group, sex, age group (< 65, ≥ 65 years), previous overactive bladder medication (yes, no) and geographic region as fixed factors and baseline value as a covariate; Test type: Superiority; p = 0.033, Stratified rank ANCOVA — Nominal p-value; No adjustment for multiplicity was needed for testing combination therapy vs. its 2 monotherapy components; Least squares mean difference = -0.20, 95% CI 2-sided [-0.44 to 0.04], Standard Error of Mean 0.12 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Mirabegron 25 mg vs Solifenacin 5 mg + Mirabegron 25 mg; Difference of the adjusted mean calculated by subtracting the adjusted mean of the mirabegron 25 mg monotherapy group from the adjusted mean of the combination group (solifenacin 5 mg + mirabegron 25 mg) based on the ANCOVA model with treatment group, sex, age group (< 65, ≥ 65 years), previous overactive bladder medication (yes, no) and geographic region as fixed factors and baseline value as a covariate; Test type: Superiority; p = 0.001, Stratified rank ANCOVA; Least squares mean difference = -0.34, 95% CI 2-sided [-0.58 to -0.10], Standard Error of Mean 0.12 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Difference of the adjusted mean calculated by subtracting the adjusted mean of the mirabegron 50 mg monotherapy group from the adjusted mean of the combination group (solifenacin 5 mg + mirabegron 50 mg) based on the ANCOVA model with treatment group, sex, age group (< 65, ≥ 65 years), previous overactive bladder medication (yes, no) and geographic region as fixed factors and baseline value as a covariate; Test type: Superiority; p = 0.052, Stratified rank ANCOVA; No adjustment for multiplicity was needed for testing combination therapy vs. its 2 monotherapy components; Least squares mean difference = -0.23, 95% CI 2-sided [-0.47 to 0.01], Standard Error of Mean 0.12 — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Change From Baseline to EoT in Mean Number of Micturitions Per 24 Hours
Description: A micturition was defined as any voluntary micturition (excluding incontinence only episodes). The mean number of micturitions per 24 hours was calculated from data recorded by the participant per day on valid diary days during the 7-day micturition diary period.
Time Frame: Baseline and EoT (up to 12 weeks)
Population: FAS. LOCF was used for EoT.
Measure: Least Squares Mean (Standard Error); unit: micturitions
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 412 | 409 | 406 | 413 | 823 | 816
micturitions | -1.64 (0.12) | -2.00 (0.12) | -2.03 (0.12) | -2.20 (0.12) | -2.49 (0.08) | -2.59 (0.08)
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.040, ANCOVA — Nominal p-value; No adjustment for multiplicity was needed for testing combination therapy vs. its 2 monotherapy components; Least squares mean difference = -0.29, 95% CI 2-sided [-0.57 to -0.01], Standard Error of Mean 0.14 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.006, ANCOVA — Nominal p-value; No adjustment for multiplicity was needed for testing combination therapy vs. its 2 monotherapy components; Least squares mean difference = -0.39, 95% CI 2-sided [-0.67 to -0.11], Standard Error of Mean 0.14 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Mirabegron 25 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.001, ANCOVA — Nominal p-value; No adjustment for multiplicity was needed for testing combination therapy vs. its 2 monotherapy components; Least squares mean difference = -0.48, 95% CI 2-sided [-0.76 to -0.21], Standard Error of Mean 0.14 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p < 0.001, ANCOVA — Nominal p-value; No adjustment for multiplicity was needed for testing combination therapy vs. its 2 monotherapy components; Least squares mean difference = -0.56, 95% CI 2-sided [-0.84 to -0.28], Standard Error of Mean 0.14 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline to EoT in Mean Volume Voided Per Micturition
Description: The mean volume voided per micturition was calculated from the data recorded by the participant during 3 consecutive days with volume measurements during the 7-day micturition diary period.
Time Frame: Baseline and EoT (up to 12 weeks)
Population: FAS. LOCF was used for EoT.
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 413 | 407 | 408 | 411 | 821 | 821
mL | 8.44 (2.55) | 13.32 (2.57) | 21.99 (2.57) | 30.99 (2.56) | 34.84 (1.81) | 39.73 (1.81)
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.219, ANCOVA — Nominal p-value; No adjustment for multiplicity was needed for testing combination therapy vs. its 2 monotherapy components; Least squares mean difference = 3.85, 95% CI 2-sided [-2.29 to 10.00], Standard Error of Mean 3.13 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.005, ANCOVA — Nominal p-value; No adjustment for multiplicity was needed for testing combination therapy vs. its 2 monotherapy components; Least squares mean difference = 8.75, 95% CI 2-sided [2.61 to 14.89], Standard Error of Mean 3.13 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Mirabegron 25 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p < 0.001, ANCOVA — Nominal p-value; No adjustment for multiplicity was needed for testing combination therapy vs. its 2 monotherapy components; Least squares mean difference = 21.52, 95% CI 2-sided [15.35 to 27.68], Standard Error of Mean 3.14 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p < 0.001, ANCOVA — Nominal p-value; No adjustment for multiplicity was needed for testing combination therapy vs. its 2 monotherapy components; Least squares mean difference = 17.74, 95% CI 2-sided [11.58 to 23.90], Standard Error of Mean 3.14 — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Change From Baseline to EoT in Overactive Bladder Questionnaire (OAB-q) Symptom Bother Score
Description: The OAB-q was a self-reported questionnaire with items relating to symptom bother and health-related quality of life (HRQoL). The symptom bother portion consisted of 8 items, rated on a 6-point Likert scale (1 through 6). The total symptom bother score was calculated from the 8 answers and then transformed to range from 0 (least severity) to 100 (worst severity). A negative change from baseline indicates an improvement.
Time Frame: Baseline and EoT (up to 12 weeks)
Population: FAS. LOCF was used for EoT.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 400 | 392 | 398 | 399 | 800 | 795
units on a scale | -19.45 (0.98) | -23.93 (0.99) | -26.14 (0.98) | -26.44 (0.98) | -31.06 (0.69) | -32.24 (0.70)
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA; No adjustment for multiplicity was made for this comparison; Least squares mean difference = -4.63, 95% CI 2-sided [-6.98 to -2.27], Standard Error of Mean 1.20
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.001, ANCOVA; No adjustment for multiplicity was made for this comparison; Least squares mean difference = -5.80, 95% CI 2-sided [-8.17 to -3.44], Standard Error of Mean 1.21
Statistical Analysis 3: Comparison: Mirabegron 25 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p < 0.001, ANCOVA; No adjustment for multiplicity was made for this comparison; Least squares mean difference = -7.13, 95% CI 2-sided [-9.50 to -4.76], Standard Error of Mean 1.21
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p < 0.001, ANCOVA; No adjustment for multiplicity was made for this comparison; Least squares mean difference = -6.10, 95% CI 2-sided [-8.46 to -3.74], Standard Error of Mean 1.20

5. Secondary Outcome: Change From Baseline to EoT in Treatment Satisfaction-Visual Analogue Scale (TS-VAS)
Description: The TS-VAS was a visual analogue scale which asked participants to rate their satisfaction with the treatment by placing a vertical mark on a line that runs from 0 (No, not at all) on the left to 10 (Yes, completely) on the right. A positive change from baseline indicated improvement.
Time Frame: Baseline and EoT (up to 12 weeks)
Population: FAS. LOCF was used for EoT.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 399 | 391 | 398 | 399 | 798 | 794
units on a scale | 1.42 (0.11) | 2.16 (0.11) | 2.18 (0.11) | 2.28 (0.11) | 2.53 (0.08) | 2.55 (0.08)
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.077, ANCOVA; No adjustment for multiplicity was made for this comparison; Least squares mean difference = 0.25, 95% CI 2-sided [-0.03 to 0.52], Standard Error of Mean 0.14
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.050, ANCOVA; No adjustment for multiplicity was made for this comparison; Least squares mean difference = 0.27, 95% CI 2-sided [0.00 to 0.55], Standard Error of Mean 0.14
Statistical Analysis 3: Comparison: Mirabegron 25 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.008, ANCOVA; No adjustment for multiplicity was made for this comparison; Least squares mean difference = 0.37, 95% CI 2-sided [0.10 to 0.65], Standard Error of Mean 0.14
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.007, ANCOVA; No adjustment for multiplicity was made for this comparison; Least squares mean difference = 0.37, 95% CI 2-sided [0.10 to 0.65], Standard Error of Mean 0.14

6. Secondary Outcome: Number of Incontinence Episodes at Weeks 4, 8, 12 and EoT
Description: The number of incontinence episodes was calculated as the total number of incontinence episodes on valid diary days recorded during the 7-day micturition diary period.
Time Frame: Weeks 4, 8, 12 and EoT (up to 12 weeks)
Population: FAS participants with available data at each time point were included in the analysis. LOCF was used for EoT.
Measure: Mean (Standard Error); unit: incontinence episodes
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
incontinence episodes
  Week 4: number analyzed (Participants) | 406 | 406 | 402 | 402 | 817 | 810
  Week 4 | 18.09 (1.17) | 15.65 (1.08) | 12.90 (1.06) | 15.31 (1.11) | 12.51 (0.67) | 11.44 (0.70)
  Week 8: number analyzed (Participants) | 397 | 385 | 386 | 386 | 784 | 769
  Week 8 | 14.45 (1.12) | 12.84 (1.05) | 11.31 (1.09) | 12.19 (1.06) | 9.70 (0.65) | 9.33 (0.68)
  Week 12: number analyzed (Participants) | 374 | 369 | 369 | 379 | 754 | 750
  Week 12 | 14.06 (1.17) | 10.60 (0.98) | 9.50 (0.98) | 11.25 (1.03) | 7.62 (0.57) | 8.21 (0.68)
  End of treatment: number analyzed (Participants) | 412 | 409 | 406 | 413 | 823 | 816
  End of treatment | 13.70 (1.08) | 11.19 (0.95) | 9.79 (0.94) | 11.21 (0.98) | 8.02 (0.55) | 8.18 (0.64)
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; Rate ratio of number of incontinence episodes during the 7-day diary between the given combination group and the given monotherapy group calculated from a negative binomial regression model incl. treatment group, sex, age group (<65, ≥65 years), geographic region and previous OAB medication (yes, no) as factors, log(number of incontinence episodes used divided by number of valid diary days) at baseline included as a covariate and number of valid diary days at EoT as the offset variable; Test type: Superiority; p = 0.135, Negative binomial regression; Rate ratio = 0.87, 95% CI 2-sided [0.72 to 1.04], Standard Error of Mean 0.09
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.282, Negative binomial regression; Rate ratio = 0.90, 95% CI 2-sided [0.75 to 1.09], Standard Error of Mean 0.09
Statistical Analysis 3: Comparison: Mirabegron 25 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p < 0.001, Negative binomial regression; Rate ratio = 0.71, 95% CI 2-sided [0.59 to 0.85], Standard Error of Mean 0.09
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.172, Negative binomial regression; Rate ratio = 0.88, 95% CI 2-sided [0.73 to 1.06], Standard Error of Mean 0.10

7. Secondary Outcome: Change From Baseline to Weeks 4, 8, 12 and EoT in Number of Incontinence Episodes
Time Frame: Baseline and weeks 4, 8, 12 and EoT (up to 12 weeks)
Population: FAS participants with available data at each time point were included in the analysis. LOCF was used for EoT.
Measure: Least Squares Mean (Standard Error); unit: incontinence episodes
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
incontinence episodes
  Week 4: number analyzed (Participants) | 406 | 406 | 402 | 402 | 817 | 810
  Week 4 | -5.23 (0.66) | -7.59 (0.66) | -8.99 (0.67) | -8.92 (0.67) | -9.62 (0.47) | -10.51 (0.47)
  Week 8: number analyzed (Participants) | 397 | 385 | 386 | 386 | 784 | 769
  Week 8 | -8.79 (0.71) | -10.57 (0.72) | -10.97 (0.72) | -11.89 (0.72) | -12.53 (0.50) | -12.78 (0.51)
  Week 12: number analyzed (Participants) | 374 | 369 | 369 | 379 | 754 | 750
  Week 12 | -9.05 (0.72) | -12.33 (0.72) | -12.58 (0.72) | -12.75 (0.71) | -14.50 (0.51) | -13.94 (0.51)
  End of treatment: number analyzed (Participants) | 412 | 409 | 406 | 413 | 823 | 816
  End of treatment | -9.42 (0.68) | -11.93 (0.68) | -12.39 (0.68) | -12.65 (0.68) | -14.29 (0.48) | -13.98 (0.48)
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; Difference of the adjusted mean calculated by subtracting the adjusted mean of the solifenacin 5 mg monotherapy group from the adjusted mean of the combination group (solifenacin 5 mg + mirabegron 25 mg) based on the ANCOVA model with treatment group, sex, age group (<65, >=65 years), previous OAB medication (yes, no) and geographic region as fixed factors and baseline value as a covariate.offset variable; Test type: Superiority; p = 0.074, Stratified rank ANCOVA; least squares mean difference = -1.64, 95% CI 2-sided [-3.27 to -0.01], Standard Error of Mean 0.83
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Difference of the adjusted mean calculated by subtracting the adjusted mean of the solifenacin 5 mg monotherapy group from the adjusted mean of the combination group (solifenacin 5 mg + mirabegron 50 mg) based on the ANCOVA model with treatment group, sex, age group (<65, >=65 years), previous OAB medication (yes, no) and geographic region as fixed factors and baseline value as a covariate; Test type: Superiority; p = 0.025, Stratified rank ANCOVA; Least squares mean difference = -1.33, 95% CI 2-sided [-2.96 to 0.30], Standard Error of Mean 0.83
Statistical Analysis 3: Comparison: Mirabegron 25 mg vs Solifenacin 5 mg + Mirabegron 25 mg; Difference of the adjusted mean calculated by subtracting the adjusted mean of the mirabegron 25 mg monotherapy group from the adjusted mean of the combination group (solifenacin 5 mg + mirabegron 25 mg) based on the ANCOVA model with treatment group, sex, age group (<65, >=65 years), previous OAB medication (yes, no) and geographic region as fixed factors and baseline value as a covariate; Test type: Superiority; p < 0.001, Stratified rank ANCOVA; least square mean difference = -2.36, 95% CI 2-sided [-4.00 to -0.73], Standard Error of Mean 0.83
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Difference of the adjusted mean calculated by subtracting the adjusted mean of the mirabegron 50 mg monotherapy group from the adjusted mean of the combination group (solifenacin 5 mg + mirabegron 50 mg) based on the ANCOVA model with treatment group, sex, age group (<65, >=65 years), previous OAB medication (yes, no) and geographic region as fixed factors and baseline value as a covariate; Test type: Superiority; p = 0.024, Stratified rank ANCOVA; Least squares mean difference = -1.59, 95% CI 2-sided [-3.23 to 0.05], Standard Error of Mean 0.84

8. Secondary Outcome: Change From Baseline to Weeks 4, 8 and 12 in Mean Number of Incontinence Episodes Per 24 Hours
Time Frame: Baseline and weeks 4, 8 and 12
Population: FAS participants with available data at each time point were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: incontinence episodes
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
incontinence episodes
  Week 4: number analyzed (Participants) | 406 | 406 | 402 | 402 | 817 | 810
  Week 4 | -0.74 (0.10) | -1.07 (0.10) | -1.24 (0.10) | -1.24 (0.10) | -1.38 (0.07) | -1.50 (0.07)
  Week 8: number analyzed (Participants) | 397 | 385 | 386 | 386 | 784 | 769
  Week 8 | -1.20 (0.10) | -1.51 (0.10) | -1.57 (0.10) | -1.66 (0.10) | -1.79 (0.07) | -1.84 (0.07)
  Week 12: number analyzed (Participants) | 374 | 369 | 369 | 379 | 754 | 750
  Week 12 | -1.30 (0.11) | -1.76 (0.11) | -1.81 (0.11) | -1.80 (0.10) | -2.08 (0.07) | -1.98 (0.07)

9. Secondary Outcome: Change From Baseline to Weeks 4, 8 and 12 in Mean Number of Micturitions Per 24 Hours
Time Frame: Baseline and weeks 4, 8 and 12
Population: FAS participants with available data at each time point data were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: micturitions
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
micturitions
  Week 4: number analyzed (Participants) | 406 | 406 | 402 | 402 | 817 | 810
  Week 4 | -1.02 (0.11) | -1.46 (0.11) | -1.44 (0.11) | -1.39 (0.11) | -1.67 (0.08) | -1.91 (0.08)
  Week 8: number analyzed (Participants) | 397 | 385 | 386 | 386 | 784 | 769
  Week 8 | -1.43 (0.11) | -1.95 (0.12) | -1.89 (0.12) | -1.84 (0.12) | -2.23 (0.08) | -2.42 (0.08)
  Week 12: number analyzed (Participants) | 374 | 369 | 369 | 379 | 754 | 750
  Week 12 | -1.51 (0.12) | -2.01 (0.12) | -2.03 (0.12) | -2.22 (0.12) | -2.47 (0.08) | -2.60 (0.08)

10. Secondary Outcome: Change From Baseline to Weeks 4, 8 and 12 in Mean Volume Voided Per Micturition
Time Frame: Baseline and weeks 4, 8 and 12
Population: FAS participants with available data at each time point were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
mL
  Week 4: number analyzed (Participants) | 403 | 398 | 399 | 395 | 798 | 802
  Week 4 | 6.95 (2.13) | 10.08 (2.14) | 15.52 (2.14) | 24.23 (2.15) | 25.54 (1.51) | 28.99 (1.51)
  Week 8: number analyzed (Participants) | 395 | 382 | 380 | 387 | 770 | 771
  Week 8 | 9.00 (2.48) | 10.96 (2.52) | 17.73 (2.53) | 27.55 (2.50) | 32.94 (1.78) | 36.51 (1.77)
  Week 12: number analyzed (Participants) | 373 | 362 | 364 | 378 | 750 | 750
  Week 12 | 8.70 (2.70) | 12.88 (2.74) | 22.40 (2.73) | 31.89 (2.68) | 35.52 (1.90) | 41.28 (1.90)

11. Secondary Outcome: Change From Baseline to EoT in Corrected Micturition Frequency
Description: Corrected micturition frequency was defined as the mean number of micturitions per 24 hours that participants had at end of treatment if their fluid intake had remained unchanged since baseline.
Time Frame: Baseline and Week 12
Population: FAS. LOCF was used for EoT.
Measure: Least Squares Mean (Standard Error); unit: micturitions
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 412 | 409 | 406 | 413 | 823 | 816
micturitions | 0.15 (0.24) | -0.17 (0.24) | -0.97 (0.24) | -1.28 (0.24) | -1.10 (0.17) | -1.52 (0.17)
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; Difference of the adjusted mean calculated by subtracting the adjusted mean of the monotherapy group (solifenacin 5 mg) from the adjusted mean of the combination group (solifenacin 5 mg + mirabegron 25 mg) based on the ANCOVA model with with treatment group, sex, age group (<65, >=65 years), previous OAB medication (yes, no) and geographic region as fixed factors and baseline mean number of micturitions per 24 hours as a covariate; Test type: Superiority; p = 0.520, ANCOVA; Least squares mean difference = 0.19, 95% CI 2-sided [-0.39 to 0.76], Standard Error of Mean 0.29
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Difference of the adjusted mean calculated by subtracting the adjusted mean of the monotherapy group (solifenacin 5 mg) from the adjusted mean of the combination group (solifenacin 5 mg + mirabegron 50 mg) based on the ANCOVA model with with treatment group, sex, age group (<65, >=65 years), previous OAB medication (yes, no) and geographic region as fixed factors and baseline mean number of micturitions per 24 hours as a covariate; Test type: Superiority; p = 0.413, ANCOVA; Least squares mean difference = -0.24, 95% CI 2-sided [-0.82 to 0.34], Standard Error of Mean 0.29
Statistical Analysis 3: Comparison: Mirabegron 25 mg vs Solifenacin 5 mg + Mirabegron 25 mg; Difference of the adjusted mean calculated by subtracting the adjusted mean of the monotherapy group (mirabegron 25 mg) from the adjusted mean of the combination group (solifenacin 5 mg + mirabegron 25 mg) based on the ANCOVA model with with treatment group, sex, age group (<65, >=65 years), previous OAB medication (yes, no) and geographic region as fixed factors and baseline mean number of micturitions per 24 hours as a covariate; Test type: Superiority; p = 0.002, ANCOVA; Least squares mean difference = -0.92, 95% CI 2-sided [-1.50 to -0.34], Standard Error of Mean 0.29
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Difference of the adjusted mean calculated by subtracting the adjusted mean of the monotherapy group (mirabegron 50 mg) from the adjusted mean of the combination group (solifenacin 5 mg + mirabegron 50 mg) based on the ANCOVA model with with treatment group, sex, age group (<65, >=65 years), previous OAB medication (yes, no) and geographic region as fixed factors and baseline mean number of micturitions per 24 hours as a covariate; Test type: Superiority; p = 0.060, ANCOVA; Least squares mean diffrence = -0.56, 95% CI 2-sided [-1.13 to 0.02], Standard Error of Mean 0.30

12. Secondary Outcome: Number of Urgency Incontinence Episodes at Weeks 4, 8, 12 and EoT
Description: An urgency incontinence episode was defined as the involuntary leakage of urine accompanied by or immediately preceded by urgency. The number of urgency incontinence episodes was the number of times a participant recorded an urgency incontinence episode on valid diary days during the 7-day micturition diary period prior to each visit.
Time Frame: Weeks 4, 8, 12 and EoT (up to 12 weeks)
Population: FAS participants with available data at each time point were included in the analysis. LOCF was used for EoT. Only participants with ≥ 1 urgency incontinence episode at baseline were included in the analysis.
Measure: Mean (Standard Error); unit: urgency incontinence episodes
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
urgency incontinence episodes
  Week 4: number analyzed (Participants) | 403 | 404 | 396 | 401 | 813 | 806
  Week 4 | 15.76 (1.10) | 13.36 (0.99) | 11.46 (1.00) | 13.19 (1.06) | 10.22 (0.58) | 9.33 (0.58)
  Week 8: number analyzed (Participants) | 394 | 383 | 380 | 385 | 780 | 765
  Week 8 | 12.77 (1.07) | 10.65 (0.94) | 10.09 (1.02) | 10.41 (1.00) | 7.58 (0.53) | 7.31 (0.54)
  Week 12: number analyzed (Participants) | 371 | 367 | 363 | 378 | 750 | 746
  Week 12 | 12.00 (1.09) | 8.84 (0.89) | 8.32 (0.94) | 9.29 (0.96) | 5.86 (0.46) | 6.27 (0.49)
  End of treatment: number analyzed (Participants) | 409 | 407 | 400 | 412 | 819 | 812
  End of treatment | 11.69 (1.00) | 9.37 (0.86) | 8.63 (0.89) | 9.29 (0.91) | 6.25 (0.45) | 6.15 (0.47)
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; Rate ratio of number of urgency incontinence episodes during the 7-day diary bet. the given combination group & the given monotherapy group calculated from a negative binomial regression model incl. treatment group, sex, age group (<65,≥ 65 years), geographic region and previous OAB medication (yes, no) as factors, baseline log(number of urgency incontinence episodes used divided by number of valid diary days) included as a covariate & postbaseline number of valid diary days as offset variable; Test type: Superiority; p = 0.110, Negative binomial regression; Rate ratio = 0.85, 95% CI 2-sided [0.70 to 1.04], Standard Error of Mean 0.10
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 0.288, Negative binomial regression; Rate ratio = 0.90, 95% CI 2-sided [0.73 to 1.10], Standard Error of Mean 0.10
Statistical Analysis 3: Comparison: Mirabegron 25 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p < 0.001, Negative binomial regression; Rate ratio = 0.65, 95% CI 2-sided [0.53 to 0.79], Standard Error of Mean 0.10
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 0.084, Negative binomial regression; Rate ratio = 0.84, 95% CI 2-sided [0.68 to 1.02], Standard Error of Mean 0.10

13. Secondary Outcome: Change From Baseline to Weeks 4, 8, 12 and EoT in Number of Urgency Incontinence Episodes
Time Frame: Baseline and weeks 4, 8, 12 and EoT (up to 12 weeks)
Population: FAS participants with available data at each time point were included in the analysis. Only participants with ≥ 1 urgency incontinence episode at baseline were included in the analysis. LOCF was used for EoT.
Measure: Least Squares Mean (Standard Error); unit: urgency incontinence episodes
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
urgency incontinence episodes
  Week 4: number analyzed (Participants) | 403 | 404 | 396 | 401 | 813 | 806
  Week 4 | -5.49 (0.63) | -7.07 (0.63) | -8.39 (0.63) | -8.53 (0.63) | -9.44 (0.44) | -10.23 (0.44)
  Week 8: number analyzed (Participants) | 394 | 383 | 380 | 385 | 780 | 765
  Week 8 | -8.30 (0.66) | -9.93 (0.67) | -10.07 (0.67) | -11.10 (0.67) | -12.18 (0.47) | -12.18 (0.47)
  Week 12: number analyzed (Participants) | 371 | 367 | 363 | 378 | 750 | 746
  Week 12 | -8.96 (0.65) | -11.39 (0.66) | -11.66 (0.66) | -12.10 (0.65) | -13.87 (0.46) | -13.53 (0.46)
  End of treatment: number analyzed (Participants) | 409 | 407 | 400 | 412 | 819 | 812
  End of treatment | -9.26 (0.62) | -11.03 (0.62) | -11.44 (0.62) | -12.03 (0.62) | -13.64 (0.44) | -13.64 (0.44)
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; Difference of the adjusted mean calculated by subtracting the adjusted mean of the monotherapy group (solifenacin 5 mg) from the adjusted mean of the combination group (solifenacin 5 mg + mirabegron 25 mg) based on the ANCOVA model with treatment group, sex, age group (<65, >=65 years), previous OAB medication (yes, no) and geographic region as fixed factors and baseline value as a covariate; Test type: Superiority; p = 0.114, Stratified rank ANCOVA; Least squares mean difference = -1.61, 95% CI 2-sided [-3.09 to -0.13], Standard Error of Mean 0.76
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Difference of the adjusted mean calculated by subtracting the adjusted mean of the monotherapy group (solifenacin 5 mg) from the adjusted mean of the combination group (solifenacin 5 mg + mirabegron 50 mg) based on the ANCOVA model with treatment group, sex, age group (<65, >=65 years), previous OAB medication (yes, no) and geographic region as fixed factors and baseline value as a covariate; Test type: Superiority; p = 0.034, Stratified rank ANCOVA; Least squares mean difference = -1.62, 95% CI 2-sided [-3.10 to -0.13], Standard Error of Mean 0.76
Statistical Analysis 3: Comparison: Mirabegron 25 mg vs Solifenacin 5 mg + Mirabegron 25 mg; Difference of the adjusted mean calculated by subtracting the adjusted mean of the monotherapy group (mirabegron 25 mg) from the adjusted mean of the combination group (solifenacin 5 mg + mirabegron 25 mg) based on the ANCOVA model with treatment group, sex, age group (<65, >=65 years), previous OAB medication (yes, no) and geographic region as fixed factors and baseline value as a covariate; Test type: Superiority; p < 0.001, Stratified rank ANCOVA; Least squares mean difference = -2.61, 95% CI 2-sided [-4.09 to -1.12], Standard Error of Mean 0.76
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Difference of the adjusted mean calculated by subtracting the adjusted mean of the monotherapy group (mirabegron 50 mg) from the adjusted mean of the combination group (solifenacin 5 mg + mirabegron 50 mg) based on the ANCOVA model with treatment group, sex, age group (<65, >=65 years), previous OAB medication (yes, no) and geographic region as fixed factors and baseline value as a covariate; Test type: Superiority; p = 0.012, Stratified rank ANCOVA; Least squares mean difference = -2.21, 95% CI 2-sided [-3.70 to -0.71], Standard Error of Mean 0.76

14. Secondary Outcome: Change From Baseline to Weeks 4, 8, 12 and EoT in Mean Number of Urgency Incontinence Episodes Per 24 Hours
Description: The mean number of urgency incontinence episodes per 24 hours was calculated from data recorded by the participant per day on valid diary days during the 7-day micturition diary period prior to each visit.
Time Frame: Baseline and weeks 4, 8, 12 and EoT (up to 12 weeks)
Population: FAS participants with available data at each time point were included in the analysis. LOCF was used for EoT.
Measure: Least Squares Mean (Standard Error); unit: urgency incontinence episodes
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
urgency incontinence episodes
  Week 4: number analyzed (Participants) | 403 | 404 | 396 | 401 | 813 | 806
  Week 4 | -0.78 (0.09) | -1.00 (0.09) | -1.15 (0.09) | -1.19 (0.09) | -1.35 (0.06) | -1.47 (0.06)
  Week 8: number analyzed (Participants) | 394 | 383 | 380 | 385 | 780 | 765
  Week 8 | -1.15 (0.10) | -1.43 (0.10) | -1.44 (0.10) | -1.56 (0.10) | -1.74 (0.07) | -1.79 (0.07)
  Week 12: number analyzed (Participants) | 371 | 367 | 363 | 378 | 750 | 746
  Week 12 | -1.29 (0.10) | -1.63 (0.10) | -1.67 (0.10) | -1.72 (0.10) | -1.99 (0.07) | -1.93 (0.07)
  End of treatment: number analyzed (Participants) | 409 | 407 | 400 | 412 | 819 | 812
  End of treatment | -1.33 (0.09) | -1.58 (0.09) | -1.62 (0.09) | -1.71 (0.09) | -1.95 (0.06) | -1.94 (0.06)
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.134, Stratified rank ANCOVA; Least squares mean difference = -0.24, 95% CI 2-sided [-0.46 to -0.02], Standard Error of Mean 0.11
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 13, analysis 2]; Test type: Superiority; p = 0.043, Stratified rank ANCOVA; Least squares mean difference = -0.23, 95% CI 2-sided [-0.45 to -0.02], Standard Error of Mean 0.11
Statistical Analysis 3: Comparison: Mirabegron 25 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 13, analysis 3]; Test type: Superiority; p < 0.001, Stratified rank ANCOVA; Least squares mean diffeence = -0.37, 95% CI 2-sided [-0.59 to -0.15], Standard Error of Mean 0.11
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Difference of the adjusted mean calculated by subtracting the adjusted mean of the monotherapy group (mirabegron 50mg ) from the adjusted mean of the combination group (solifenacin 5 mg + mirabegron 50 mg) based on the ANCOVA model with treatment group, sex, age group (<65, >=65 years), previous OAB medication (yes, no) and geographic region as fixed factors and baseline value as a covariate; Test type: Superiority; p = 0.019, Stratified rank ANCOVA; Standard Error of the Mean = -0.32, 05% CI 2-sided [-0.54 to -0.10], Standard Error of Mean 0.11

15. Secondary Outcome: Change From Baseline to Weeks 4, 8, 12 and EoT in Mean Number of Urgency Episodes (Grade 3 or 4) Per 24 Hours
Description: An urgency episode was a complaint of a sudden, compelling desire to pass urine, which was difficult to defer; it was recorded when a micturition or incontinence episode was recorded and the severity of urinary urgency recorded was 3 (severe urgency) or 4 (urgency incontinence) according to the Patient Perception of Intensity of Urgency Scale (PPIUS). The mean number of urgency episodes per 24 hours was calculated from data recorded by the participant per day on valid diary days during the 7-day micturition diary period prior to each visit.
Time Frame: Baseline and weeks 4, 8, 12 and EoT (up to 12 weeks)
Population: FAS participants with available data at each time point were included in the analysis. LOCF was used for EoT. Only participants with ≥ 1 urgency episode at baseline were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: urgency episodes
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
urgency episodes
  Week 4: number analyzed (Participants) | 405 | 406 | 402 | 402 | 817 | 810
  Week 4 | -1.34 (0.15) | -1.95 (0.14) | -1.91 (0.15) | -2.14 (0.15) | -2.42 (0.10) | -2.66 (0.10)
  Week 8: number analyzed (Participants) | 396 | 385 | 386 | 386 | 784 | 769
  Week 8 | -1.85 (0.15) | -2.54 (0.15) | -2.43 (0.15) | -2.90 (0.15) | -3.13 (0.11) | -3.28 (0.11)
  Week 12: number analyzed (Participants) | 373 | 369 | 369 | 379 | 754 | 750
  Week 12 | -2.05 (0.16) | -2.85 (0.16) | -2.70 (0.16) | -3.11 (0.16) | -3.45 (0.11) | -3.50 (0.11)
  End of treatment: number analyzed (Participants) | 411 | 409 | 406 | 413 | 823 | 816
  End of treatment | -2.06 (0.15) | -2.74 (0.15) | -2.63 (0.15) | -3.05 (0.15) | -3.38 (0.11) | -3.51 (0.11)
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.074, ANCOVA; Least squares mean difference = -0.33, 95% CI 2-sided [-0.69 to 0.03], Standard Error of Mean 0.18
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 13, analysis 2]; Test type: Superiority; p = 0.014, ANCOVA; Least squares mean difference = -0.45, 95% CI 2-sided [-0.82 to -0.09], Standard Error of Mean 0.18
Statistical Analysis 3: Comparison: Mirabegron 25 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 13, analysis 3]; Test type: Superiority; p < 0.001, ANCOVA; Least squares mean difference = -0.65, 95% CI 2-sided [-1.01 to -0.28], Standard Error of Mean 0.18
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 13, analysis 4]; Test type: Superiority; p < 0.001, ANCOVA; Least squares mean difference = -0.87, 95% CI 2-sided [-1.24 to 0.51], Standard Error of Mean 0.19

16. Secondary Outcome: Number of Nocturia Episodes at Weeks 4, 8, 12 and EoT
Description: A nocturia episode was defined as waking at night 1 or more times to void (i.e., any voiding associated with sleep disturbance between the time the participant went to bed with the intention to sleep until the time the patients got up in the morning with the intention to stay awake). The number of nocturia episodes was the number of times a participant recorded a nocturia episode on valid diary days during the 7-day micturition diary period prior to each visit.
Time Frame: Weeks 4, 8, 12 and EoT (up to 12 weeks)
Population: FAS participants with available data at each time point were included in the analysis. LOCF was used for EoT. Only participants with ≥ 1 nocturia episode at baseline were included in the analysis.
Measure: Mean (Standard Error); unit: nocturia episodes
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
nocturia episodes
  Week 4: number analyzed (Participants) | 359 | 341 | 349 | 341 | 705 | 693
  Week 4 | 9.62 (0.43) | 8.46 (0.36) | 9.11 (0.47) | 9.22 (0.42) | 8.40 (0.25) | 8.09 (0.25)
  Week 8: number analyzed (Participants) | 349 | 327 | 336 | 329 | 676 | 655
  Week 8 | 8.99 (0.44) | 8.07 (0.34) | 8.61 (0.45) | 8.37 (0.38) | 7.63 (0.25) | 7.11 (0.24)
  Week 12: number analyzed (Participants) | 336 | 312 | 321 | 320 | 652 | 641
  Week 12 | 8.91 (0.43) | 7.99 (0.37) | 8.34 (0.48) | 8.17 (0.39) | 7.26 (0.24) | 6.67 (0.23)
  End of treatment: number analyzed (Participants) | 363 | 344 | 353 | 350 | 708 | 697
  End of treatment | 8.83 (0.42) | 7.79 (0.35) | 8.14 (0.45) | 8.12 (0.37) | 7.33 (0.24) | 6.67 (0.22)
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; Rate ratio of number of incontinence episodes during the 7-day diary between the given combination group and the given monotherapy group calculated from a negative binomial regression model incl. treatment group, sex, age group (<65, >=65 years), geographic region and previous OAB medication (yes, no) as factors, baseline log(number of nocturia episodes used divided by number of valid diary days) included as a covariate and postbaseline number of valid diary days as offset variable; Test type: Superiority; p = 0.006, Negative binomial regression; Rate ratio = 0.88, 95% CI 2-sided [0.81 to 0.96], Standard Error of Mean 0.05
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 16, analysis 1]; Test type: Superiority; p < 0.001, Negative binomial regression; Rate ratio = 0.81, 95% CI 2-sided [0.74 to 0.88], Standard Error of Mean 0.05
Statistical Analysis 3: Comparison: Mirabegron 25 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 16, analysis 1]; Test type: Superiority; p = 0.049, Negative binomial regression; Rate ratio = 0.91, 95% CI 2-sided [0.84 to 1.00], Standard Error of Mean 0.05
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 16, analysis 1]; Test type: Superiority; p = 0.001, Negative binomial regression; Rate ratio = 0.86, 95% CI 2-sided [0.79 to 0.94], Standard Error of Mean 0.05

17. Secondary Outcome: Change From Baseline to Weeks 4, 8, 12 and EoT in Number of Nocturia Episodes
Time Frame: Baseline and weeks 4, 8, 12, and EoT (up to 12 weeks)
Population: as for outcome 16
Measure: Least Squares Mean (Standard Error); unit: nocturia episodes
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
nocturia episodes
  Week 4: number analyzed (Participants) | 359 | 341 | 349 | 341 | 705 | 693
  Week 4 | -1.27 (0.27) | -2.25 (0.28) | -1.80 (0.27) | -1.79 (0.28) | -2.39 (0.19) | -2.50 (0.19)
  Week 8: number analyzed (Participants) | 349 | 327 | 336 | 329 | 676 | 655
  Week 8 | -1.94 (0.27) | -2.70 (0.28) | -2.41 (0.28) | -2.60 (0.28) | -3.13 (0.20) | -3.48 (0.20)
  Week 12: number analyzed (Participants) | 336 | 312 | 321 | 320 | 652 | 641
  Week 12 | -1.95 (0.29) | -2.77 (0.30) | -2.73 (0.29) | -2.89 (0.29) | -3.49 (0.21) | -3.96 (0.21)
  End of treatment: number analyzed (Participants) | 363 | 344 | 353 | 350 | 708 | 697
  End of treatment | -2.05 (0.27) | -2.91 (0.28) | -2.75 (0.28) | -2.81 (0.28) | -3.42 (0.20) | -3.96 (0.20)
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.073, ANCOVA; Least squares mean difference = -0.61, 95% CI 2-sided [-1.28 to 0.06], Standard Error of Mean 0.34
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 13, analysis 2]; Test type: Superiority; p = 0.001, ANCOVA; Least squares mean difference = -1.16, 95% CI 2-sided [-1.83 to -0.48], Standard Error of Mean 0.34
Statistical Analysis 3: Comparison: Mirabegron 25 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 13, analysis 3]; Test type: Superiority; p = 0.140, ANCOVA; Least squares mean difference = -0.51, 95% CI 2-sided [-1.18 to 0.17], Standard Error of Mean 0.34
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 13, analysis 4]; Test type: Superiority; p < 0.001, ANCOVA; Least squares mean difference = -1.21, 95% CI 2-sided [-1.88 to -0.54], Standard Error of Mean 0.34

18. Secondary Outcome: Change From Baseline to Weeks 4, 8, 12 and EoT in Mean Number of Nocturia Episodes Per 24 Hours
Description: The mean number of nocturia episodes per 24hr was calculated from data recorded by the participant per day on valid diary days during the 7-day micturition diary period prior to each visit.
Time Frame: Baseline and weeks 4, 8, 12 and EoT (up to 12 weeks)
Population: as for outcome 16
Measure: Least Squares Mean (Standard Error); unit: nocturia episodes
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
nocturia episodes
  Week 4: number analyzed (Participants) | 359 | 341 | 349 | 341 | 705 | 693
  Week 4 | -0.17 (0.04) | -0.31 (0.04) | -0.25 (0.04) | -0.24 (0.04) | -0.33 (0.03) | -0.35 (0.03)
  Week 8: number analyzed (Participants) | 349 | 327 | 336 | 329 | 676 | 655
  Week 8 | -0.27 (0.04) | -0.37 (0.04) | -0.35 (0.04) | -0.36 (0.04) | -0.44 (0.03) | -0.50 (0.03)
  Week 12: number analyzed (Participants) | 336 | 312 | 321 | 320 | 652 | 641
  Week 12 | -0.26 (0.04) | -0.38 (0.04) | -0.39 (0.04) | -0.41 (0.04) | -0.49 (0.03) | -0.56 (0.03)
  End of treatmemt: number analyzed (Participants) | 363 | 344 | 353 | 350 | 708 | 697
  End of treatmemt | -0.27 (0.04) | -0.40 (0.04) | -0.39 (0.04) | -0.39 (0.04) | -0.48 (0.03) | -0.56 (0.03)
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.065, ANCOVA; Least squares mean difference = -0.09, 95% CI 2-sided [-0.19 to 0.01], Standard Error of Mean 0.05
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 13, analysis 2]; Test type: Superiority; p = 0.001, ANCOVA; Least squares mean difference = -0.17, 95% CI 2-sided [-0.26 to -0.07], Standard Error of Mean 0.05
Statistical Analysis 3: Comparison: Mirabegron 25 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 13, analysis 3]; Test type: Superiority; p = 0.100, ANCOVA; Least squares mean difference = -0.08, 95% CI 2-sided [-0.18 to 0.02], Standard Error of Mean 0.05
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 13, analysis 4]; Test type: Superiority; p = 0.001, ANCOVA; Least squares mean difference = -0.17, 95% CI 2-sided [-0.26 to -0.07], Standard Error of Mean 0.05

19. Secondary Outcome: Number of Pads Used at Weeks 4, 8, 12 and EoT
Description: The number of pads used was the number of times a participant recorded a new pad used on valid diary days during the 7-day micturition diary period prior to each visit.
Time Frame: Weeks 4, 8 and 12 (up to 12 weeks)
Population: FAS participants with available data at each time point were included in the analysis. LOCF was used for EoT. Only participants with ≥ 1 pad used at baseline were included in the analysis.
Measure: Mean (Standard Error); unit: pads
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
pads
  Week 4: number analyzed (Participants) | 248 | 250 | 247 | 257 | 506 | 499
  Week 4 | 15.62 (1.33) | 13.46 (1.24) | 10.05 (1.21) | 11.41 (1.23) | 9.71 (0.70) | 9.34 (0.68)
  Week 8: number analyzed (Participants) | 239 | 237 | 240 | 243 | 485 | 472
  Week 8 | 12.75 (1.22) | 10.79 (1.05) | 9.53 (1.39) | 8.45 (1.03) | 8.07 (0.65) | 7.58 (0.62)
  Week 12: number analyzed (Participants) | 226 | 225 | 229 | 241 | 468 | 461
  Week 12 | 12.62 (1.21) | 9.65 (1.00) | 8.44 (1.26) | 8.21 (0.95) | 6.60 (0.58) | 6.64 (0.61)
  End of treatment: number analyzed (Participants) | 252 | 252 | 249 | 262 | 510 | 502
  End of treatment | 12.29 (1.11) | 10.15 (0.97) | 8.16 (1.17) | 8.53 (0.94) | 7.04 (0.56) | 6.80 (0.59)
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; Rate ratio of number of incontinence episodes during the 7-day diary between the given combination group and the given monotherapy group calculated from a negative binomial regression model incl. treatment group, sex, age group (<65, >=65 years), geographic region and previous OAB medication (yes, no) as factors, baseline log(number of pads used divided by number of valid diary days) included as a covariate and postbaseline number of valid diary days as offset variable; Test type: Superiority; p = 0.938, Negative binomial regression; Rate ratio = 1.01, 95% CI 2-sided [0.80 to 1.27], Standard Error of Mean 0.12
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 19, analysis 1]; Test type: Superiority; p = 0.967, Negative binomial regression; Rate ratio = 1.00, 95% CI 2-sided [0.79 to 1.25], Standard Error of Mean 0.12
Statistical Analysis 3: Comparison: Mirabegron 25 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 19, analysis 1]; Test type: Superiority; p = 0.008, Negative binomial regression; Standard Error of the Mean = 0.73, 95% CI 2-sided [0.58 to 0.92], Standard Error of Mean 0.12
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 19, analysis 1]; Test type: Superiority; p = 0.069, Negative binomial regression; Rate ratio = 0.80, 95% CI 2-sided [0.64 to 1.02], Standard Error of Mean 0.12

20. Secondary Outcome: Change From Baseline to Weeks 4, 8, 12 and EoT in Number of Pads Used
Time Frame: Baseline and weeks 4, 8, 12 and EOT (up to 12 weeks)
Population: as for outcome 19
Measure: Least Squares Mean (Standard Error); unit: pads
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
pads
  Week 4: number analyzed (Participants) | 248 | 250 | 247 | 257 | 506 | 499
  Week 4 | -3.69 (0.71) | -5.68 (0.71) | -7.83 (0.71) | -8.23 (0.70) | -7.61 (0.50) | -8.58 (0.50)
  Week 8: number analyzed (Participants) | 239 | 237 | 240 | 243 | 485 | 472
  Week 8 | -6.24 (0.77) | -8.44 (0.77) | -8.43 (0.76) | -10.67 (0.76) | -9.49 (0.54) | -10.59 (0.54)
  Week 12: number analyzed (Participants) | 226 | 225 | 229 | 241 | 468 | 461
  Week 12 | -6.29 (0.75) | -9.06 (0.75) | -9.41 (0.75) | -10.80 (0.73) | -10.66 (0.52) | -11.23 (0.53)
  End of treatment: number analyzed (Participants) | 252 | 252 | 249 | 262 | 510 | 502
  End of treatment | -6.60 (0.71) | -8.76 (0.71) | -9.80 (0.72) | -10.63 (0.70) | -10.67 (0.50) | -11.21 (0.50)
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.958, ANCOVA; Least squares mean difference = -0.04, 95% CI 2-sided [-1.73 to 1.64], Standard Error of Mean 0.86
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 13, analysis 2]; Test type: Superiority; p = 0.500, ANCOVA; Least squares mean difference = -0.58, 95% CI 2-sided [-2.27 to 1.11], Standard Error of Mean 0.86
Statistical Analysis 3: Comparison: Mirabegron 25 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 13, analysis 3]; Test type: Superiority; p = 0.028, ANCOVA; Least squares mean difference = -1.91, 95% CI 2-sided [-3.62 to -0.20], Standard Error of Mean 0.87
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 13, analysis 4]; Test type: Superiority; p = 0.108, ANCOVA; Least squares mean difference = -1.41, 95% CI 2-sided [-3.13 to 0.31], Standard Error of Mean 0.88

21. Secondary Outcome: Change From Baseline to Weeks 4, 8, 12 and EoT in Mean Number of Pads Used Per 24 Hours
Description: The mean number of pads used per 24 hours was calculated from data recorded by the participant per day on valid diary days during the 7-day micturition diary period prior to each visit.
Time Frame: Baseline and weeks 4, 8 and 12 (up to 12 weeks)
Population: as for outcome 19
Measure: Least Squares Mean (Standard Error); unit: pads
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
pads
  Week 4: number analyzed (Participants) | 248 | 250 | 247 | 257 | 506 | 499
  Week 4 | -0.52 (0.10) | -0.81 (0.10) | -1.12 (0.10) | -1.19 (0.10) | -1.09 (0.07) | -1.23 (0.07)
  Week 8: number analyzed (Participants) | 239 | 237 | 240 | 243 | 485 | 472
  Week 8 | -0.82 (0.11) | -1.20 (0.11) | -1.24 (0.11) | -1.53 (0.11) | -1.36 (0.08) | -1.51 (0.08)
  Week 12: number analyzed (Participants) | 226 | 225 | 229 | 241 | 468 | 461
  Week 12 | -0.92 (0.11) | -1.30 (0.11) | -1.37 (0.11) | -1.56 (0.11) | -1.54 (0.08) | -1.59 (0.08)
  End of treatment: number analyzed (Participants) | 252 | 252 | 249 | 262 | 510 | 502
  End of treatment | -0.94 (0.10) | -1.26 (0.10) | -1.41 (0.10) | -1.53 (0.10) | -1.53 (0.07) | -1.58 (0.07)
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.993, ANCOVA; Least squares mean difference = 0.00, 95% CI 2-sided [-0.25 to 0.25], Standard Error of Mean 0.13
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 13, analysis 2]; Test type: Superiority; p = 0.650, ANCOVA; Least squares mean difference = -0.06, 95% CI 2-sided [-0.30 to 0.19], Standard Error of Mean 0.13
Statistical Analysis 3: Comparison: Mirabegron 25 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 13, analysis 3]; Test type: Superiority; p = 0.035, ANCOVA; Least squares mean difference = -0.27, 95% CI 2-sided [-0.52 to -0.02], Standard Error of Mean 0.13
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 13, analysis 4]; Test type: Superiority; p = 0.169, ANCOVA; Least squares mean difference = -0.18, 95% CI 2-sided [-0.43 to 0.08], Standard Error of Mean 0.13

22. Secondary Outcome: Number of Incontinence-Free Days at Weeks 4, 8, 12 and EoT
Description: The number of incontinence-free days was the number of valid diary days during the 7-day micturition diary period with no incontinence episodes recorded.
Time Frame: Weeks 4, 8, 12 and EoT (up to 12 weeks)
Population: FAS participants with available data at each time point were included in the analysis. LOCF was used for EoT.
Measure: Mean (Standard Error); unit: incontinence-free days
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
incontinence-free days
  Week 4: number analyzed (Participants) | 406 | 406 | 402 | 402 | 817 | 810
  Week 4 | 2.25 (0.13) | 2.48 (0.13) | 2.98 (0.13) | 2.74 (0.14) | 3.08 (0.10) | 3.37 (0.10)
  Week 8: number analyzed (Participants) | 397 | 385 | 386 | 386 | 784 | 769
  Week 8 | 2.92 (0.14) | 3.17 (0.14) | 3.63 (0.15) | 3.31 (0.14) | 3.88 (0.10) | 4.01 (0.10)
  Week 12: number analyzed (Participants) | 374 | 369 | 369 | 379 | 754 | 750
  Week 12 | 3.19 (0.15) | 3.69 (0.15) | 3.96 (0.15) | 3.68 (0.14) | 4.33 (0.10) | 4.25 (0.10)
  End of treatment: number analyzed (Participants) | 412 | 409 | 406 | 413 | 823 | 816
  End of treatment | 3.16 (0.14) | 3.51 (0.14) | 3.89 (0.14) | 3.61 (0.14) | 4.20 (0.10) | 4.23 (0.10)
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; Odds ratio from a overdispersed binomial regression model (Williams' method) including treatment group, sex, age group (<65, >=65 years), previous OAB medication (yes, no) and geographic region as factors and baseline logarithm of mean number of incontinence episodes per 24 hours as a covariate; Test type: Superiority; p = 0.003, Overdispersed binomial regression; Odds Ratio (OR) = 1.37, 95% CI 2-sided [1.11 to 1.68]
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 22, analysis 1]; Test type: Superiority; p = 0.004, Overdispersed binomial regression; Odds Ratio (OR) = 1.36, 95% CI 2-sided [1.11 to 1.68]
Statistical Analysis 3: Comparison: Mirabegron 25 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 22, analysis 1]; Test type: Superiority; p < 0.001, Overdispersed binomial regression; Odds Ratio (OR) = 1.59, 95% CI 2-sided [1.29 to 1.95]
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 22, analysis 1]; Test type: Superiority; p = 0.004, Overdispersed binomial regression; Odds Ratio (OR) = 1.36, 95% CI 2-sided [1.10 to 1.68]

23. Secondary Outcome: Number of Days With < 8 Micturitions at Weeks 4, 8, 12 and EoT
Description: The number of days with < 8 micturitions was the number of valid diary days during the 7-day micturition diary period with less than 8 micturitions per day.
Time Frame: Weeks 4, 8,12 and EoT (up to 12 weeks)
Population: FAS participants with available data at each time point were included in the analysis. LOCF was used for EoT.
Measure: Mean (Standard Error); unit: days
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
days
  Week 4: number analyzed (Participants) | 406 | 406 | 402 | 402 | 817 | 810
  Week 4 | 1.49 (0.10) | 1.74 (0.10) | 1.55 (0.10) | 1.86 (0.11) | 2.07 (0.08) | 2.11 (0.08)
  Week 8: number analyzed (Participants) | 397 | 385 | 386 | 386 | 784 | 769
  Week 8 | 1.69 (0.10) | 2.08 (0.12) | 1.99 (0.11) | 2.22 (0.12) | 2.59 (0.09) | 2.70 (0.09)
  Week 12: number analyzed (Participants) | 374 | 369 | 369 | 379 | 754 | 750
  Week 12 | 1.76 (0.11) | 2.31 (0.13) | 2.25 (0.12) | 2.49 (0.13) | 2.87 (0.09) | 2.95 (0.10)
  End of treatment: number analyzed (Participants) | 412 | 409 | 406 | 413 | 823 | 816
  End of treatment | 1.80 (0.11) | 2.28 (0.12) | 2.22 (0.12) | 2.49 (0.12) | 2.84 (0.09) | 2.92 (0.09)
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; Odds ratio from a overdispersed binomial regression model (Williams' method) including treatment group, sex, age group (<65, >=65 years), previous OAB medication (yes, no) and geographic region as factors and baseline mean number of micturitions per 24 hours as a covariate; Test type: Superiority; p = 0.039, Overdispersed binomial regression; Odds Ratio (OR) = 1.23, 95% CI 2-sided [1.01 to 1.50]
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 23, analysis 1]; Test type: Superiority; p = 0.009, Overdispersed binomial regression; Odds Ratio (OR) = 1.30, 95% CI 2-sided [1.07 to 1.59]
Statistical Analysis 3: Comparison: Mirabegron 25 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 23, analysis 1]; Test type: Superiority; p < 0.001, overdispersed binomial regression; Odds Ratio (OR) = 1.45, 95% CI 2-sided [1.19 to 1.77]
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 23, analysis 1]; Test type: Superiority; p < 0.001, Overdispersed binomial regression; Odds Ratio (OR) = 1.50, 95% CI 2-sided [1.23 to 1.84]

24. Secondary Outcome: Number of Incontinence-Free Days With < 8 Micturitions at Weeks 4, 8, 12 and EoT
Description: The number of incontinence-free days with < 8 micturitions per day was the number of valid diary days during the 7-day micturition diary period with no incontinence episodes recorded and with < 8 micturitions per day.
Time Frame: Weeks 4, 8, 12 and EoT (up to 12 weeks)
Population: FAS participants with available data at each time point were included in the analysis. LOCF was used for EoT.
Measure: Mean (Standard Error); unit: days
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
days
  Week 4: number analyzed (Participants) | 406 | 406 | 402 | 402 | 817 | 810
  Week 4 | 0.64 (0.07) | 0.84 (0.08) | 0.87 (0.08) | 0.91 (0.08) | 1.21 (0.07) | 1.32 (0.07)
  Week 8: number analyzed (Participants) | 397 | 385 | 386 | 386 | 784 | 769
  Week 8 | 0.85 (0.08) | 1.20 (0.10) | 1.23 (0.10) | 1.31 (0.10) | 1.75 (0.08) | 1.89 (0.08)
  Week 12: number analyzed (Participants) | 374 | 369 | 369 | 379 | 754 | 750
  Week 12 | 0.98 (0.09) | 1.47 (0.11) | 1.50 (0.11) | 1.60 (0.11) | 2.12 (0.09) | 2.15 (0.09)
  End of treatment: number analyzed (Participants) | 412 | 409 | 406 | 413 | 823 | 816
  End of treatment | 1.01 (0.08) | 1.40 (0.10) | 1.47 (0.10) | 1.59 (0.10) | 2.04 (0.08) | 2.12 (0.09)
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 23, analysis 1]; Test type: Superiority; p = 0.011, Overdispersed binomial regression; Odds Ratio (OR) = 1.32, 95% CI 2-sided [1.07 to 1.64]
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 23, analysis 1]; Test type: Superiority; p = 0.002, Overdispersed binomial regression; Odds Ratio (OR) = 1.41, 95% CI 2-sided [1.14 to 1.75]
Statistical Analysis 3: Comparison: Mirabegron 25 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 23, analysis 1]; Test type: Superiority; p < 0.001, Overdispersed binomial regression; Odds Ratio (OR) = 1.65, 95% CI 2-sided [1.32 to 2.06]
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 23, analysis 1]; Test type: Superiority; p < 0.001, Overdispersed binomial regression; Odds Ratio (OR) = 1.66, 95% CI 2-sided [1.33 to 2.07]

25. Secondary Outcome: Change From Baseline to Weeks 4, 8, 12 and EoT in Patient Perception of Bladder Condition Questionnaire (PPBC)
Description: The PPBC was a validated, global assessment tool using a 6-point Likert scale on which participants rated their subjective impression of their current bladder condition. Participants assessed their bladder condition using this scale: 1. Does not cause me any problems at all; 2. Causes me some very minor problems; 3. Causes me some minor problems; 4. Causes me (some) moderate problems; 5. Causes me severe problems; 6. Causes me many severe problems.
Time Frame: Baseline and weeks 4, 8, 12, EoT (up to 12 weeks)
Population: FAS participants with available data at each time point were included in the analysis. LOCF was used for EoT .
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
units on a scale
  Week 4: number analyzed (Participants) | 397 | 388 | 393 | 394 | 791 | 791
  Week 4 | -0.54 (0.06) | -0.72 (0.06) | -0.83 (0.06) | -0.81 (0.06) | -0.99 (0.04) | -1.07 (0.04)
  Week 8: number analyzed (Participants) | 381 | 372 | 380 | 385 | 758 | 761
  Week 8 | -0.80 (0.06) | -1.07 (0.06) | -1.12 (0.06) | -1.18 (0.06) | -1.32 (0.04) | -1.48 (0.04)
  Week 12: number analyzed (Participants) | 371 | 362 | 366 | 375 | 739 | 735
  Week 12 | -0.95 (0.06) | -1.23 (0.06) | -1.34 (0.06) | -1.32 (0.06) | -1.57 (0.04) | -1.72 (0.04)
  End of treatment: number analyzed (Participants) | 400 | 393 | 398 | 399 | 801 | 795
  End of treatment | -0.91 (0.06) | -1.18 (0.06) | -1.31 (0.06) | -1.27 (0.06) | -1.53 (0.04) | -1.66 (0.04)
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA; Least squares mean difference = -0.26, 95% CI 2-sided [-0.41 to -0.11], Standard Error of Mean 0.07
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 13, analysis 2]; Test type: Superiority; p < 0.001, ANCOVA; Least squares mean difference = -0.39, 95% CI 2-sided [-0.54 to -0.25], Standard Error of Mean 0.07
Statistical Analysis 3: Comparison: Mirabegron 25 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 13, analysis 3]; Test type: Superiority; p < 0.001, ANCOVA; Least squares mean difference = -0.35, 95% CI 2-sided [-0.50 to -0.20], Standard Error of Mean 0.07
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 13, analysis 4]; Test type: Superiority; p < 0.001, ANCOVA; Least squares mean difference = -0.35, 95% CI 2-sided [-0.50 to -0.20], Standard Error of Mean 0.07

26. Secondary Outcome: Change From Baseline to Weeks 4, 8 and 12 in the OAB-q Symptom Bother Score
Description: The OAB-q was a self-reported questionnaire with items relating to symptom bother and health-related quality of life (HRQoL). The symptom bother portion in the OAB-q (seen in this outcome measure) consisted of 8 items, rated on a 6-point Likert scale (1 through 6). The total symptom bother score was calculated from the 8 answers and then transformed to range from 0 (least severity) to 100 (worst severity). A negative change from baseline indicated an improvement.
Time Frame: Baseline and weeks 4, 8 and 12
Population: FAS participants with available data at each time point were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
units on a scale
  Week 4: number analyzed (Participants) | 397 | 388 | 392 | 394 | 790 | 789
  Week 4 | -13.84 (0.92) | -17.05 (0.93) | -18.98 (0.93) | -19.53 (0.93) | -23.46 (0.65) | -25.19 (0.65)
  Week 8: number analyzed (Participants) | 381 | 370 | 380 | 385 | 757 | 761
  Week 8 | -17.35 (0.98) | -22.79 (0.99) | -23.54 (0.98) | -24.69 (0.97) | -29.10 (0.69) | -30.04 (0.69)
  Week 12: number analyzed (Participants) | 371 | 362 | 366 | 374 | 738 | 734
  Week 12 | -19.94 (1.01) | -24.44 (1.02) | -26.80 (1.02) | -26.72 (1.01) | -31.70 (0.72) | -33.15 (0.72)

27. Secondary Outcome: Change From Baseline to Weeks 4, 8, 12 and EoT in OAB-q Health-Related Quality of Life Questionnaire (HRQL) Total Score
Description: The OAB-q was a self-reported questionnaire with items relating to symptom bother and health-related quality of life (HRQoL). The HRQoL portion in the OAB-q (seen in this outcome measure) consisted of 25 HRQL items comprising 4 HRQL subscales (Coping, Concern, Sleep, and Social Interaction), scored 1-6. The total HRQoL score was calculated by adding the 4 HRQoL subscale scores and transforming to a scale from 0 to 100, with higher scores indicating better quality of life. A positive change from baseline indicated an improvement.
Time Frame: Baseline and weeks 4, 8, 12 and EoT (up to 12 weeks)
Population: FAS participants with available data at each time point were included in the analysis. LOCF was used for EoT.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
units on a scale
  Week 4: number analyzed (Participants) | 397 | 388 | 392 | 394 | 790 | 789
  Week 4 | 10.16 (0.83) | 13.54 (0.83) | 15.28 (0.83) | 14.78 (0.83) | 17.46 (0.58) | 17.95 (0.59)
  Week 8: number analyzed (Participants) | 381 | 370 | 380 | 385 | 757 | 761
  Week 8 | 14.51 (0.88) | 17.95 (0.89) | 18.54 (0.88) | 18.57 (0.88) | 22.30 (0.62) | 22.45 (0.62)
  Week 12: number analyzed (Participants) | 371 | 362 | 366 | 374 | 738 | 734
  Week 12 | 15.76 (0.92) | 19.59 (0.93) | 21.48 (0.92) | 20.54 (0.91) | 24.63 (0.65) | 24.93 (0.65)
  End of treatment: number analyzed (Participants) | 400 | 392 | 398 | 399 | 800 | 795
  End of treatment | 15.37 (0.88) | 18.94 (0.89) | 21.00 (0.89) | 20.15 (0.89) | 23.96 (0.63) | 24.30 (0.63)
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA; Least squares mean difference = 3.81, 95% CI 2-sided [1.69 to 5.94], Standard Error of Mean 1.08
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 13, analysis 2]; Test type: Superiority; p < 0.001, ANCOVA; Least squares mean difference = 4.16, 95% CI 2-sided [2.03 to 6.29], Standard Error of Mean 1.09
Statistical Analysis 3: Comparison: Mirabegron 25 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 13, analysis 3]; Test type: Superiority; p < 0.001, ANCOVA; Least squares mean difference = 5.02, 95% CI 2-sided [2.88 to 7.15], Standard Error of Mean 1.09
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 13, analysis 4]; Test type: Superiority; p = 0.002, ANCOVA; Least squares mean difference = 3.30, 95% CI 2-sided [1.17 to 5.43], Standard Error of Mean 1.09

28. Secondary Outcome: Change From Baseline to Weeks 4, 8, 12 and EoT in OAB-q HRQL Subscale Score: Coping
Description: The Coping score was calculated by adding 8 response scores and transforming to a scale from 0 to 100, with higher scores indicating better quality of life. A positive change from baseline indicated an improvement.
Time Frame: Baseline and weeks 4, 8, 12 and EoT (up to 12 weeks)
Population: FAS participants with available data at each time point were included in the analysis. LOCF was used for EoT.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
units on a scale
  Week 4: number analyzed (Participants) | 397 | 388 | 392 | 394 | 790 | 789
  Week 4 | 11.74 (0.99) | 14.87 (1.00) | 17.68 (1.00) | 16.52 (1.00) | 19.31 (0.70) | 20.36 (0.70)
  Week 8: number analyzed (Participants) | 381 | 370 | 380 | 385 | 757 | 761
  Week 8 | 16.13 (1.04) | 20.64 (1.05) | 21.52 (1.04) | 21.69 (1.03) | 25.49 (0.74) | 25.85 (0.73)
  Week 12: number analyzed (Participants) | 371 | 362 | 366 | 374 | 738 | 734
  Week 12 | 18.17 (1.09) | 22.04 (1.10) | 24.94 (1.10) | 23.67 (1.09) | 28.32 (0.77) | 29.03 (0.78)
  End of treatment: number analyzed (Participants) | 400 | 392 | 398 | 399 | 800 | 795
  End of treatment | 17.73 (1.05) | 21.28 (1.06) | 24.32 (1.05) | 23.25 (1.05) | 27.37 (0.74) | 28.12 (0.75)
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.001, ANCOVA; Least squares mean difference = 4.12, 95% CI 2-sided [1.60 to 6.65], Standard Error of Mean 1.29
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 13, analysis 2]; Test type: Superiority; p < 0.001, ANCOVA; Lest squares mean difference = 4.87, 95% CI 2-sided [2.34 to 7.40], Standard Error of Mean 1.29
Statistical Analysis 3: Comparison: Mirabegron 25 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 13, analysis 3]; Test type: Superiority; p < 0.001, ANCOVA; Least squares mean difference = 6.09, 95% CI 2-sided [3.55 to 8.63], Standard Error of Mean 1.30
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 13, analysis 4]; Test type: Superiority; p = 0.003, ANCOVA; Least squares mean difference = 3.80, 95% CI 2-sided [1.27 to 6.33], Standard Error of Mean 1.29

29. Secondary Outcome: Change From Baseline to Weeks 4, 8, 12 and EoT in OAB-q HRQL Subscale Score: Concern
Description: The Concern score was calculated by adding 7 response scores and transforming to a scale from 0 to 100, with higher scores indicating better quality of life. A positive change from baseline indicated an improvement.
Time Frame: Baseline and weeks 4, 8, 12 and EoT (up to 12 weeks)
Population: FAS participants with available data at each time point were included in the analysis. LOCF was used for EoT.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
units on a scale
  Week 4: number analyzed (Participants) | 397 | 388 | 392 | 394 | 790 | 789
  Week 4 | 11.24 (0.95) | 15.89 (0.96) | 17.39 (0.95) | 17.18 (0.95) | 20.48 (0.67) | 21.09 (0.67)
  Week 8: number analyzed (Participants) | 381 | 370 | 380 | 385 | 757 | 761
  Week 8 | 16.10 (0.99) | 20.63 (1.01) | 20.55 (1.00) | 20.96 (0.99) | 25.26 (0.71) | 25.65 (0.70)
  Week 12: number analyzed (Participants) | 371 | 362 | 366 | 374 | 738 | 734
  Week 12 | 17.53 (1.03) | 22.37 (1.04) | 23.62 (1.04) | 23.19 (1.03) | 27.53 (0.73) | 28.24 (0.73)
  End of treatment: number analyzed (Participants) | 400 | 392 | 398 | 399 | 800 | 795
  End of treatment | 16.98 (1.00) | 21.55 (1.01) | 23.07 (1.00) | 22.65 (1.00) | 26.89 (0.71) | 27.47 (0.71)
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.001, ANCOVA; Least squares mean difference = 4.24, 95% CI 2-sided [1.84 to 6.63], Standard Error of Mean 1.22
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 13, analysis 2]; Test type: Superiority; p < 0.001, ANCOVA; Least squares mean difference = 4.82, 95% CI 2-sided [2.42 to 7.22], Standard Error of Mean 1.22
Statistical Analysis 3: Comparison: Mirabegron 25 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 13, analysis 3]; Test type: Superiority; p < 0.001, ANCOVA; Least squares mean difference = 5.34, 95% CI 2-sided [2.93 to 7.75], Standard Error of Mean 1.23
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 13, analysis 4]; Test type: Superiority; p < 0.001, ANCOVA; Least squares mean difference = 4.41, 95% CI 2-sided [2.01 to 6.81], Standard Error of Mean 1.22

30. Secondary Outcome: Change From Baseline to Weeks 4, 8, 12 and EoT in OAB-q HRQL Subscale Score: Sleep
Description: The Sleep score was calculated by adding 5 response scores and transforming to a scale from 0 to 100, with higher scores indicating better quality of life. A positive change from baseline indicated an improvement.
Time Frame: Baseline and weeks 4, 8, 12 and EoT (up to 12 weeks)
Population: FAS participants with available data at each time point were included in the analysis. LOCF was used for EoT.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
units on a scale
  Week 4: number analyzed (Participants) | 397 | 388 | 392 | 394 | 790 | 789
  Week 4 | 9.28 (0.95) | 12.70 (0.96) | 13.80 (0.96) | 13.08 (0.96) | 15.97 (0.68) | 16.66 (0.68)
  Week 8: number analyzed (Participants) | 381 | 370 | 380 | 385 | 757 | 761
  Week 8 | 13.58 (1.03) | 16.39 (1.05) | 17.33 (1.03) | 16.43 (1.03) | 20.29 (0.73) | 20.49 (0.73)
  Week 12: number analyzed (Participants) | 371 | 362 | 366 | 374 | 738 | 734
  Week 12 | 14.40 (1.05) | 18.04 (1.06) | 19.16 (1.06) | 18.35 (1.05) | 22.97 (0.74) | 22.76 (0.75)
  End of treatment: number analyzed (Participants) | 400 | 392 | 398 | 399 | 800 | 795
  End of treatment | 14.17 (1.01) | 17.51 (1.02) | 19.11 (1.02) | 17.97 (1.01) | 22.39 (0.72) | 22.39 (0.72)
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA; Least squares mean difference = 4.42, 95% CI 2-sided [1.98 to 6.85], Standard Error of Mean 1.24
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 13, analysis 2]; Test type: Superiority; p < 0.001, ANCOVA; Least squares mean difference = 4.42, 95% CI 2-sided [1.98 to 6.86], Standard Error of Mean 1.24
Statistical Analysis 3: Comparison: Mirabegron 25 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 13, analysis 3]; Test type: Superiority; p < 0.001, ANCOVA; Least squares mean difference = 4.87, 95% CI 2-sided [2.42 to 7.32], Standard Error of Mean 1.25
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 13, analysis 4]; Test type: Superiority; p = 0.008, ANCOVA; Least squares mean difference = 3.28, 95% CI 2-sided [0.84 to 5.72], Standard Error of Mean 1.24

31. Secondary Outcome: Change From Baseline to Weeks 4, 8, 12 and EoT in OAB-q HRQL Subscale Score: Social
Description: The Social score was calculated by adding 5 response scores and transforming to a scale from 0 to 100, with higher scores indicating better quality of life. A positive change from baseline indicated an improvement.
Time Frame: Weeks 4, 8, 12 and EoT (up to 12 weeks)
Population: FAS participants with available data at each time point were included in the analysis. LOCF was used for EoT.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
units on a scale
  Week 4: number analyzed (Participants) | 397 | 388 | 392 | 394 | 790 | 789
  Week 4 | 7.07 (0.78) | 9.04 (0.79) | 10.19 (0.78) | 9.89 (0.78) | 11.55 (0.55) | 11.25 (0.55)
  Week 8: number analyzed (Participants) | 381 | 370 | 380 | 385 | 757 | 761
  Week 8 | 10.65 (0.82) | 11.50 (0.83) | 12.34 (0.82) | 12.02 (0.81) | 14.89 (0.58) | 14.73 (0.58)
  Week 12: number analyzed (Participants) | 371 | 362 | 366 | 374 | 738 | 734
  Week 12 | 10.84 (0.83) | 13.43 (0.84) | 15.35 (0.84) | 13.74 (0.83) | 16.16 (0.59) | 16.08 (0.59)
  End of treatment: number analyzed (Participants) | 400 | 392 | 398 | 399 | 800 | 795
  End of treatment | 10.56 (0.81) | 13.04 (0.81) | 14.87 (0.81) | 13.57 (0.81) | 15.84 (0.57) | 15.82 (0.57)
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.022, ANCOVA; Least squares mean difference = 2.27, 95% CI 2-sided [0.33 to 4.21], Standard Error of Mean 0.99
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 13, analysis 2]; Test type: Superiority; p = 0.023, ANCOVA; Least squares mean difference = 2.25, 95% CI 2-sided [0.31 to 4.19], Standard Error of Mean 0.99
Statistical Analysis 3: Comparison: Mirabegron 25 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 13, analysis 3]; Test type: Superiority; p = 0.005, ANCOVA; Least squares mean difference = 2.80, 95% CI 2-sided [0.85 to 4.74], Standard Error of Mean 0.99
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 13, analysis 4]; Test type: Superiority; p = 0.337, ANCOVA; Least squares mean difference = 0.95, 95% CI 2-sided [-0.99 to 2.89], Standard Error of Mean 0.99

32. Secondary Outcome: Patient's Global Impression of Change (PGIC) Scale: Impression in Bladder Symptoms at Week 12 and EoT
Description: The PGIC was a 2-part questionnaire, assessing both the change in the patient's overall condition and change in bladder condition since the start of the study (from very much worse to very much improved).
Time Frame: Week 12 and EoT (up to 12 weeks)
Population: FAS participants with available data were included in the analysis. LOCF was used for EoT.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
percentage of participants
  Week 12: Very much improved | 8.4 | 13.9 | 15.1 | 13.5 | 19.8 | 27.1
  Week 12: Much improved | 29.7 | 32.9 | 34.8 | 40.5 | 39.8 | 34.0
  Week 12: Minimally improved | 29.7 | 26.8 | 26.5 | 25.8 | 22.2 | 20.7
  Week 12: No change | 17.5 | 12.9 | 9.7 | 8.9 | 7.7 | 7.3
  Week 12: Minimally worse | 4.1 | 1.5 | 2.2 | 1.7 | 0.8 | 0.8
  Week 12: Much worse | 1.0 | 1.0 | 1.2 | 0.5 | 0.2 | 0
  Week 12: Very much worse | 0.5 | 0.5 | 0.7 | 0.5 | 0.2 | 0.5
  EoT: Very much improved | 8.4 | 13.9 | 15.1 | 13.5 | 20.0 | 27.1
  EoT: Much improved | 30.4 | 33.2 | 34.8 | 41.0 | 40.0 | 34.6
  EoT: Minimally improved | 29.9 | 26.8 | 27.0 | 26.3 | 22.6 | 21.3
  EoT: No change | 18.2 | 13.4 | 10.2 | 9.6 | 7.9 | 7.4
  EoT: Minimally worse | 4.1 | 1.5 | 2.2 | 1.7 | 0.8 | 0.8
  EoT: Much worse | 1.0 | 1.0 | 1.2 | 0.7 | 0.4 | 0
  EoT: Very much worse | 0.5 | 0.5 | 0.7 | 0.5 | 0.2 | 0.6

33. Secondary Outcome: PGIC Scale: Impression in General Health at Week 12 and EoT
Description: as for outcome 32
Time Frame: Week 12 and EoT (up to 12 weeks)
Population: FAS participants with available data were included in the analysis. LOCF was used for EoT.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
percentage of participants
  Week 12: Very much improved | 4.8 | 8.0 | 7.3 | 7.7 | 10.3 | 14.6
  Week 12: Much improved | 23.9 | 28.0 | 29.2 | 31.8 | 33.4 | 30.2
  Week 12: Minimally improved | 23.9 | 21.5 | 22.4 | 24.1 | 20.1 | 20.9
  Week 12: No change | 31.8 | 27.8 | 27.5 | 25.3 | 23.9 | 21.6
  Week 12: Minimally worse | 4.3 | 2.9 | 2.2 | 1.4 | 2.5 | 2.2
  Week 12: Much worse | 1.7 | 0.7 | 1.2 | 0.5 | 0.5 | 0.1
  Week 12: Very much worse | 0.2 | 0.5 | 0.5 | 0.5 | 0.2 | 0.6
  End of treatment: Very much improved | 4.8 | 8.0 | 7.3 | 7.7 | 10.3 | 14.6
  End of treatment: Much improved | 24.2 | 28.0 | 29.2 | 31.8 | 33.6 | 30.4
  End of treatment: Minimally improved | 24.4 | 21.5 | 22.9 | 24.1 | 20.2 | 21.3
  End of treatment:No change | 32.3 | 28.3 | 27.7 | 26.5 | 24.3 | 21.9
  End of treatment: Minimally worse | 4.3 | 2.9 | 2.4 | 1.9 | 2.8 | 2.7
  End of treatment: Much worse | 1.9 | 0.7 | 1.2 | 0.5 | 0.5 | 0.2
  End of treatment: Very much worse | 0.5 | 0.7 | 0.5 | 0.7 | 0.2 | 0.7

34. Secondary Outcome: Change From Baseline to EoT in European Quality of Life in 5 Dimensions (EQ-5D) Questionnaire Subscale Score: Mobility
Description: The EQ-5D questionnaire was an international, standardized, nondisease specific instrument for describing and valuing health status, and has 5 dimensions: Mobility, Self-care, Usual Activities, Pain/Discomfort, and Anxiety/Depression. Each dimension had 5 response levels ranging from level 1 (no problem or none) to level 5 (unable to perform activity).
Time Frame: Baseline and EoT (up to 12 weeks)
Population: FAS participants with available data were included in the analysis. LOCF was used for EoT.
Measure: Number; unit: participants
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
participants
  No problems -> no problems | 204 | 239 | 225 | 227 | 449 | 452
  No problems -> slight problems | 16 | 20 | 25 | 22 | 41 | 38
  No problems -> moderate problems | 11 | 12 | 9 | 8 | 20 | 10
  No problems -> severe problems | 1 | 3 | 3 | 1 | 1 | 2
  No problems -> unable to walk about | 0 | 1 | 0 | 0 | 0 | 1
  No problems -> no data | 2 | 4 | 5 | 4 | 6 | 9
  Slight problems -> no problems | 33 | 35 | 35 | 30 | 76 | 60
  Slight problems -> slight problems | 27 | 20 | 24 | 19 | 40 | 49
  Slight problems -> moderate problems | 11 | 6 | 4 | 6 | 19 | 9
  Slight problems -> severe problems | 5 | 0 | 3 | 1 | 2 | 2
  Slight problems -> unable to walk about | 0 | 0 | 0 | 0 | 0 | 0
  Slight problems -> no data | 2 | 3 | 0 | 0 | 0 | 2
  Moderate problems -> no problems | 17 | 7 | 25 | 18 | 31 | 46
  Moderate problems -> slight problems | 18 | 10 | 10 | 22 | 24 | 25
  Moderate problems -> moderate problems | 21 | 12 | 10 | 13 | 33 | 35
  Moderate problems -> severe problems | 10 | 5 | 4 | 2 | 8 | 10
  Moderate problems -> unable to walk about | 0 | 0 | 0 | 1 | 1 | 1
  Moderate problems -> no data | 1 | 1 | 0 | 1 | 0 | 2
  Severe problems -> no problems | 3 | 5 | 9 | 7 | 12 | 17
  Severe problems -> slight problems | 6 | 7 | 3 | 4 | 13 | 8
  Severe problems -> moderate problems | 5 | 4 | 8 | 8 | 15 | 15
  Severe problems -> severe problems | 8 | 5 | 1 | 8 | 11 | 13
  Severe problems -> unable to walk about | 0 | 0 | 0 | 0 | 0 | 0
  Severe problems -> no data | 0 | 0 | 2 | 1 | 1 | 0
  Unable to walk about -> no problems | 0 | 0 | 0 | 2 | 2 | 0
  Unable to walk about -> slight problems | 1 | 0 | 0 | 0 | 0 | 0
  Unable to walk about -> moderate problems | 1 | 0 | 0 | 0 | 0 | 1
  Unable to walk about -> severe problems | 1 | 0 | 0 | 0 | 0 | 0
  Unable to walk about -> unable to walk about | 0 | 0 | 0 | 0 | 0 | 0
  Unable to walk about -> no data | 0 | 0 | 0 | 0 | 0 | 0
  No data -> no problems | 12 | 7 | 3 | 6 | 15 | 16
  No data -> slight problems | 1 | 0 | 1 | 2 | 4 | 2
  No data -> moderate problems | 0 | 3 | 1 | 0 | 0 | 2
  No data -> severe problems | 0 | 1 | 0 | 2 | 2 | 0
  No data -> unable to walk about | 0 | 0 | 0 | 0 | 0 | 0
  No data -> no data | 1 | 0 | 1 | 0 | 1 | 0

35. Secondary Outcome: Change From Baseline to EoT in EQ-5D Questionnaire Subscale Score: Self-Care
Description: as for outcome 34
Time Frame: Baseline and EoT (up to 12 weeks)
Population: FAS participants with available data were included in the analysis. LOCF was used for EoT.
Measure: Number; unit: participants
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
participants
  No problems -> no problems | 311 | 324 | 336 | 319 | 652 | 647
  No problems -> slight problems | 21 | 17 | 9 | 20 | 22 | 26
  No problems -> moderate problems | 9 | 5 | 6 | 3 | 12 | 4
  No problems -> severe problems | 0 | 0 | 1 | 1 | 1 | 1
  No problems -> unable to wash/dress myself | 1 | 0 | 1 | 0 | 0 | 0
  No problems -> no data | 4 | 8 | 6 | 5 | 6 | 12
  Slight problems -> no problems | 17 | 13 | 16 | 25 | 35 | 33
  Slight problems -> slight problems | 10 | 10 | 12 | 12 | 22 | 26
  Slight problems -> moderate problems | 2 | 4 | 1 | 2 | 3 | 7
  Slight problems -> severe problems | 2 | 0 | 0 | 0 | 1 | 2
  Slight problems -> unable to wash/dress myself | 0 | 0 | 0 | 0 | 0 | 0
  Slight problems -> no data | 1 | 0 | 0 | 1 | 1 | 0
  Moderate problems -> no problems | 6 | 8 | 3 | 2 | 17 | 18
  Moderate problems -> slight problems | 3 | 1 | 8 | 3 | 9 | 7
  Moderate problems -> moderate problems | 9 | 1 | 2 | 6 | 8 | 9
  Moderate problems -> severe problems | 0 | 0 | 0 | 0 | 2 | 1
  Moderate problems -> unable to wash/dress myself | 0 | 0 | 0 | 0 | 0 | 0
  Moderate problems -> no data | 0 | 0 | 0 | 0 | 0 | 1
  Severe problems -> no problems | 2 | 2 | 2 | 1 | 3 | 4
  Severe problems -> slight problems | 1 | 0 | 0 | 3 | 3 | 3
  Severe problems -> moderate problems | 1 | 2 | 0 | 0 | 7 | 3
  Severe problems -> severe problems | 3 | 3 | 0 | 1 | 1 | 0
  Severe problems -> unable to wash/dress myself | 0 | 0 | 0 | 0 | 0 | 0
  Severe problems -> no data | 0 | 0 | 1 | 0 | 0 | 0
  Unable to wash/dress myself -> no problems | 0 | 1 | 1 | 0 | 0 | 3
  Unable to wash/dress myself -> slight problems | 0 | 0 | 0 | 0 | 0 | 0
  Unable to wash/dress myself -> moderate problems | 1 | 0 | 0 | 0 | 0 | 0
  Unable to wash/dress myself -> severe problems | 0 | 0 | 0 | 0 | 0 | 0
  Unable to wash/dress myself -> unable to w/d | 0 | 0 | 0 | 1 | 0 | 0
  Unable to wash/dress myself -> no data | 0 | 0 | 0 | 0 | 0 | 0
  No data -> no problems | 13 | 8 | 3 | 8 | 20 | 18
  No data -> slight problems | 0 | 2 | 2 | 1 | 1 | 0
  No data -> moderate problems | 0 | 1 | 0 | 1 | 0 | 2
  No data -> severe problems | 0 | 0 | 0 | 0 | 0 | 0
  No data -> unable to wash/dress myself | 0 | 0 | 0 | 0 | 0 | 0
  No data -> no data | 1 | 0 | 1 | 0 | 1 | 0

36. Secondary Outcome: Change From Baseline to EoT in EQ-5D Questionnaire Subscale Score: Usual Activities
Description: as for outcome 34
Time Frame: Baseline and EoT (up to 12 weeks)
Population: FAS participants with available data were included in the analysis. LOCF was used for EoT.
Measure: Number; unit: participants
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
participants
  No problems -> No problems | 196 | 228 | 219 | 223 | 434 | 451
  No problems -> Slight problems | 37 | 25 | 28 | 25 | 37 | 48
  No problems -> Moderate problems | 9 | 5 | 9 | 8 | 13 | 11
  No problems -> Severe problems | 2 | 0 | 1 | 0 | 1 | 1
  No problems -> unable to do usual activities | 0 | 0 | 0 | 0 | 1 | 1
  No problems -> no data | 2 | 5 | 4 | 3 | 5 | 8
  Slight problems -> no problems | 45 | 41 | 52 | 52 | 98 | 95
  Slight problems -> slight problems | 28 | 29 | 23 | 25 | 64 | 56
  Slight problems -> moderate problems | 15 | 9 | 3 | 8 | 18 | 12
  Slight problems -> severe problems | 2 | 0 | 2 | 0 | 2 | 3
  Slight problems ->unable to do usual activities | 0 | 0 | 0 | 0 | 0 | 0
  Slight problems -> no data | 2 | 2 | 0 | 3 | 2 | 4
  Moderate problems -> no problems | 14 | 13 | 15 | 13 | 44 | 26
  Moderate problems -> slight problems | 12 | 9 | 16 | 14 | 29 | 30
  Moderate problems -> moderate problems | 15 | 11 | 9 | 12 | 25 | 17
  Moderate problems -> severe problems | 1 | 3 | 0 | 1 | 3 | 3
  Moderate problems ->unable to do usual activities | 0 | 0 | 0 | 0 | 0 | 1
  Moderate problems -> no data | 1 | 1 | 2 | 0 | 0 | 1
  Severe problems -> no problems | 7 | 3 | 7 | 6 | 7 | 11
  Severe problems -> slight problems | 3 | 4 | 6 | 2 | 8 | 8
  Severe problems -> moderate problems | 6 | 7 | 5 | 6 | 9 | 7
  Severe problems -> severe problems | 4 | 1 | 1 | 3 | 2 | 9
  Severe problems -> unable to do usual activities | 0 | 1 | 0 | 0 | 0 | 0
  Severe problems -> no data | 0 | 0 | 1 | 0 | 0 | 0
  Unable to do usual activities -> no problems | 0 | 1 | 0 | 0 | 0 | 2
  Unable to do usual activities -> slight problems | 1 | 0 | 0 | 0 | 1 | 1
  Unable to do usual activities -> moderate problems | 2 | 1 | 1 | 0 | 1 | 1
  Unable to do usual activities -> severe problems | 0 | 0 | 1 | 0 | 0 | 0
  Unable to do usual activities -> unable to do usu. | 0 | 0 | 0 | 1 | 1 | 0
  Unable to do usual activities -> no data | 0 | 0 | 0 | 0 | 0 | 0
  No data -> no problems | 12 | 7 | 2 | 7 | 18 | 15
  No data -> slight problems | 1 | 2 | 3 | 1 | 1 | 3
  No data -> moderate problems | 0 | 2 | 0 | 2 | 2 | 2
  No data -> severe problems | 0 | 0 | 0 | 0 | 0 | 0
  No data -> unable to do usual activities | 0 | 0 | 0 | 0 | 0 | 0
  No data -> no data | 1 | 0 | 1 | 0 | 1 | 0

37. Secondary Outcome: Change From Baseline to EoT in EQ-5D Questionnaire Subscale Score: Pain/Discomfort
Description: as for outcome 34
Time Frame: Baseline and EoT (up to 12 weeks)
Population: FAS participants with available data were included in the analysis. LOCF was used for EoT.
Measure: Number; unit: participants
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
participants
  No pain/discomfort -> no pain/discomfort | 131 | 175 | 153 | 154 | 290 | 317
  No pain/discomfort -> slight pain/discomfort | 38 | 29 | 37 | 33 | 74 | 51
  No pain/discomfort -> moderate pain/discomfort | 10 | 9 | 17 | 13 | 19 | 20
  No pain/discomfort -> severe pain/discomfort | 0 | 0 | 3 | 3 | 3 | 1
  No pain/discomfort -> extreme pain/discomfort | 0 | 0 | 0 | 0 | 1 | 0
  No pain/discomfort -> no data | 2 | 3 | 4 | 2 | 3 | 8
  Slight pain/discomfort -> no pain/discomfort | 53 | 51 | 44 | 46 | 117 | 105
  Slight pain/discomfort -> slight pain/discomfort | 54 | 49 | 45 | 47 | 94 | 101
  Slight pain/discomfort -> moderate pain/discomfort | 12 | 11 | 14 | 18 | 15 | 19
  Slight pain/discomfort -> severe pain/discomfort | 3 | 0 | 2 | 0 | 6 | 3
  Slight pain/discomfort -> exteme pain/discomfort | 2 | 0 | 1 | 0 | 0 | 0
  Slight pain/discomfort -> no data | 2 | 5 | 2 | 2 | 2 | 4
  Moderate pain/discomfort -> no pain/discomfort | 20 | 14 | 24 | 23 | 45 | 46
  Moderate pain/discomfort -> slight pain/discomfort | 23 | 15 | 20 | 22 | 46 | 45
  Moderate pain/discomfort -> moderate pain/discomf | 31 | 13 | 16 | 15 | 34 | 40
  Moderate pain/discomfort -> severe pain/discomfort | 4 | 5 | 3 | 1 | 4 | 6
  Moderate pain/discomfort -> extreme pain/discomf | 0 | 0 | 0 | 0 | 1 | 0
  Moderate pain/discomfort -> no data | 1 | 0 | 0 | 1 | 1 | 1
  Severe pain/discomfort -> no pain/discomfort | 2 | 4 | 3 | 1 | 8 | 12
  Severe pain/discomfort -> slight pain/discomfort | 3 | 4 | 6 | 4 | 11 | 7
  Severe pain/discomfort -> moderate pain/discomfort | 8 | 4 | 6 | 11 | 15 | 11
  Severe pain/discomfort -> severe pain/discomfort | 4 | 3 | 1 | 4 | 7 | 8
  Severe pain/discomfort -> extreme pain/discomfort | 0 | 1 | 1 | 0 | 1 | 0
  Severe pain/discomfort -> no data | 0 | 0 | 1 | 0 | 1 | 0
  Extreme pain/discomfort -> no pain/discomfort | 0 | 0 | 0 | 0 | 1 | 0
  Extreme pain/discomfort -> slight pain/discomfort | 1 | 0 | 0 | 2 | 1 | 1
  Extreme pain/discomfort -> moderate pain/discom. | 0 | 2 | 1 | 0 | 1 | 1
  Extreme pain/discomfort -> severe pain/discomfort | 0 | 2 | 1 | 2 | 3 | 0
  Extreme pain/discomfort -> extreme pain/discomfort | 0 | 0 | 0 | 0 | 1 | 0
  Extreme pain/discomfort -> no data | 0 | 0 | 0 | 1 | 0 | 0
  No data -> no pain/discomfort | 11 | 5 | 3 | 6 | 14 | 14
  No data -> slight pain/discomfort | 2 | 2 | 2 | 2 | 6 | 3
  No data -> moderate pain/discomfort | 0 | 4 | 0 | 2 | 1 | 3
  No data -> severe pain/discomfort | 0 | 0 | 0 | 0 | 0 | 0
  No data -> extreme pain/discomfort | 0 | 0 | 0 | 0 | 0 | 0
  No data -> no data | 1 | 0 | 1 | 0 | 1 | 0

38. Secondary Outcome: Change From Baseline to EoT in EQ-5D Questionnaire Subscale Score: Anxiety/Depression
Description: as for outcome 34
Time Frame: Baseline and EoT (up to 12 weeks)
Population: FAS participants with available data were included in the analysis. LOCF was used for EoT.
Measure: Number; unit: participants
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
participants
  Not anxious -> not anxious | 157 | 176 | 187 | 166 | 360 | 370
  Not anxious -> slightly anxious | 42 | 27 | 25 | 29 | 45 | 50
  Not anxious -> moderately anxious | 7 | 6 | 6 | 8 | 13 | 11
  Not anxious -> severely anxious | 0 | 2 | 5 | 1 | 2 | 1
  Not anxious -> extremely anxious | 0 | 0 | 1 | 0 | 0 | 1
  Not anxious -> no data | 2 | 3 | 2 | 1 | 3 | 6
  Slightly anxious -> not anxious | 42 | 60 | 54 | 59 | 122 | 134
  Slightly anxious -> slightly anx | 49 | 40 | 45 | 40 | 79 | 65
  Slightly anxious -> moderately anxious | 17 | 16 | 12 | 17 | 18 | 16
  Slightly anxious -> severely anxious | 4 | 2 | 2 | 2 | 5 | 5
  Slightly anxious -> extremely anxious | 0 | 0 | 0 | 0 | 1 | 0
  Slightly anxious -> no data | 2 | 3 | 2 | 5 | 3 | 4
  Moderately anxious -> not anxious | 12 | 13 | 12 | 22 | 42 | 35
  Moderately anxious -> slightly anxious | 19 | 17 | 19 | 14 | 43 | 41
  Moderately anxious -> moderately anxious | 17 | 7 | 11 | 10 | 18 | 23
  Moderately anxious -> severely anxious | 2 | 3 | 0 | 1 | 8 | 7
  Moderately anxious -> extremely anxious | 0 | 1 | 0 | 0 | 1 | 1
  Moderately anxious -> no data | 1 | 1 | 2 | 0 | 1 | 3
  Severely anxious -> not anxious | 7 | 5 | 6 | 6 | 12 | 8
  Severely anxious -> slightly anxious | 3 | 3 | 4 | 5 | 11 | 6
  Severely anxious -> moderately anxious | 5 | 7 | 2 | 6 | 6 | 7
  Severely anxious -> severely anxious | 10 | 1 | 2 | 5 | 5 | 2
  Severely anxious -> extremely anxious | 1 | 0 | 0 | 1 | 0 | 3
  Severely anxious -> no data | 0 | 1 | 1 | 0 | 0 | 0
  Extremely anxious -> not anxious | 2 | 1 | 0 | 0 | 2 | 1
  Extremely anxious -> slightly anxious | 2 | 2 | 1 | 2 | 2 | 3
  Extremely anxious -> moderately anxious | 1 | 1 | 1 | 1 | 2 | 1
  Extremely anxious -> severely anxious | 0 | 1 | 1 | 3 | 0 | 1
  Extremely anxious -> extremely anxious | 0 | 0 | 2 | 1 | 1 | 2
  Extremely anxious -> no data | 0 | 0 | 0 | 0 | 0 | 0
  No data -> not anxious | 9 | 8 | 3 | 6 | 13 | 14
  No data -> slightly anxious | 4 | 1 | 2 | 2 | 6 | 3
  No data -> moderately anxious | 0 | 2 | 0 | 2 | 1 | 2
  No data -> severely anxious | 0 | 0 | 0 | 0 | 0 | 1
  No data -> extremely anxious | 0 | 0 | 0 | 0 | 1 | 0
  No data -> no data | 1 | 0 | 1 | 0 | 1 | 0

39. Secondary Outcome: Change From Baseline to Week 12 and EoT in Work Productivity and Activity Impairment: Specific Health Problem Questionnaire (WPAI:SHP) Score: Percent Work Time Missed
Description: The WPAI:SHP was a self-administered questionnaire with 6 questions (Q1=Employment status; Q2=Hours absent from work due to the bladder condition; Q3=Hours absent from work due to other reasons; Q4=Hours actually worked; Q5=Impact of the bladder condition on productivity while working; Q6=Impact of the bladder condition on productivity while doing regular daily activities other than work) and a 1-week recall period. WPAI outcomes were expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity, i.e., worse outcomes. A negative change from baseline indicated improvement.
Time Frame: Baseline and week 12 and EoT (up to 12 weeks)
Population: FAS participants with available data at each time point were included in the analysis. LOCF was used for EoT. Only participants with both baseline and post-baseline values were included in the analysis.
Measure: Mean (Standard Deviation); unit: percentage of work time missed
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
percentage of work time missed
  Week 12: number analyzed (Participants) | 128 | 127 | 139 | 130 | 274 | 244
  Week 12 | -2.98 (21.70) | -0.33 (22.03) | -1.72 (18.70) | -2.47 (14.13) | -2.06 (20.93) | -2.59 (19.65)
  End of treatment: number analyzed (Participants) | 129 | 127 | 140 | 132 | 277 | 247
  End of treatment | -2.96 (21.61) | -0.33 (22.03) | -1.71 (18.64) | -2.44 (14.03) | -1.48 (21.95) | -2.55 (19.54)

40. Secondary Outcome: Change From Baseline to Week 12 and EoT in WPAI:SHP Score: Percent Impairment While Working
Time Frame: Baseline and week 12 and EoT (up to 12 weeks)
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: percentage of impairment while working
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
percentage of impairment while working
  Week 12: number analyzed (Participants) | 126 | 122 | 138 | 130 | 271 | 241
  Week 12 | -11.27 (25.36) | -14.96 (26.21) | -12.25 (25.06) | -10.85 (25.58) | -14.69 (26.99) | -13.07 (27.35)
  End of treatment: number analyzed (Participants) | 127 | 122 | 139 | 132 | 273 | 244
  End of treatment | -11.18 (25.28) | -14.96 (26.21) | -12.37 (25.01) | -10.98 (25.68) | -14.58 (26.92) | -12.87 (27.31)

41. Secondary Outcome: Change From Baseline to Week 12 and EoT in WPAI:SHP Score: Percent Overall Work Impairment
Time Frame: Baseline and week 12 and EoT (up to 12 weeks)
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: percentage of overall work impairment
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
percentage of overall work impairment
  Week 12: number analyzed (Participants) | 126 | 122 | 138 | 130 | 271 | 241
  Week 12 | -12.23 (25.66) | -15.70 (26.54) | -12.92 (26.71) | -12.31 (26.91) | -16.31 (29.06) | -13.97 (29.30)
  End of treatment: number analyzed (Participants) | 127 | 122 | 139 | 132 | 273 | 244
  End of treatment | -12.14 (25.58) | -15.70 (26.54) | -13.05 (26.65) | -12.42 (26.98) | -16.07 (29.12) | -13.76 (29.25)

42. Secondary Outcome: Change From Baseline to Week 12 and EoT in WPAI:SHP Score: Percent Activity Impairment
Time Frame: Baseline and week 12 and EoT (up to 12 weeks)
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: percentage of activity impairment
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
percentage of activity impairment
  Week 12: number analyzed (Participants) | 368 | 358 | 365 | 373 | 730 | 731
  Week 12 | -11.49 (27.31) | -16.89 (27.57) | -14.99 (27.81) | -16.19 (29.16) | -19.60 (28.80) | -18.92 (29.47)
  End of treatment: number analyzed (Participants) | 375 | 361 | 368 | 380 | 736 | 743
  End of treatment | -11.55 (27.19) | -16.72 (27.82) | -15.05 (27.95) | -16.05 (28.95) | -19.45 (28.80) | -18.76 (29.33)

43. Secondary Outcome: Change From Baseline to Weeks 4, 8 and 12 in TS-VAS
Description: as for outcome 5
Time Frame: Baseline and week 4, 8 and 12
Population: FAS participants with available data at each time point were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
units on a scale
  Week 4: number analyzed (Participants) | 395 | 386 | 391 | 394 | 788 | 788
  Week 4 | 1.14 (0.12) | 1.68 (0.12) | 1.77 (0.12) | 1.82 (0.12) | 2.06 (0.08) | 2.13 (0.08)
  Week 8: number analyzed (Participants) | 380 | 369 | 380 | 385 | 754 | 756
  Week 8 | 1.50 (0.11) | 2.16 (0.12) | 2.09 (0.11) | 2.20 (0.11) | 2.48 (0.08) | 2.48 (0.08)
  Week 12: number analyzed (Participants) | 370 | 361 | 366 | 373 | 736 | 732
  Week 12 | 1.47 (0.12) | 2.24 (0.12) | 2.23 (0.12) | 2.32 (0.12) | 2.58 (0.08) | 2.63 (0.08)

44. Secondary Outcome: Percentage of Participants With Zero Incontinence Episodes Per 24 Hours Using the Last 3 Diary Days at Weeks 4, 8, 12 and EoT
Description: The percentage of participants with zero incontinence episodes per 24 hours postbaseline in the last 3 days prior to weeks 4, 8, 12 and EoT.
Time Frame: Weeks 4, 8, 12 and EoT (up to 12 weeks)
Population: FAS participants with available data at each time point were included in the analysis. LOCF was used for EoT.
Measure: Number; unit: percentage of particpants
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
percentage of particpants
  Week 4: number analyzed (Participants) | 406 | 406 | 402 | 402 | 817 | 810
  Week 4 | 23.2 | 24.9 | 27.6 | 28.9 | 35.1 | 37.3
  Week 8: number analyzed (Participants) | 397 | 385 | 386 | 386 | 784 | 769
  Week 8 | 28.7 | 35.3 | 40.7 | 38.3 | 45.3 | 48.2
  Week 12: number analyzed (Participants) | 374 | 369 | 369 | 379 | 754 | 750
  Week 12 | 38.0 | 42.5 | 47.4 | 42.7 | 52.3 | 52.7
  End of treatment: number analyzed (Participants) | 412 | 409 | 406 | 413 | 823 | 816
  End of treatment | 37.6 | 40.6 | 46.3 | 42.9 | 50.7 | 52.2
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; Odds ratio from a logistic regression model including treatment group, sex, age group (<65, >=65 years), previous OAB medication (yes, no) and geographic region as factors and baseline mean number of incontinence episodes per 24 hours during the last 3 days as a covariate; Test type: Superiority; p = 0.035, Logistic regression; Odds Ratio (OR) = 1.31, 95% CI 2-sided [1.02 to 1.69]
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 44, analysis 1]; Test type: Superiority; p = 0.009, Logistic regression; Odds Ratio (OR) = 1.40, 95% CI 2-sided [1.09 to 1.81]
Statistical Analysis 3: Comparison: Mirabegron 25 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 44, analysis 1]; Test type: Superiority; p = 0.002, Logistic regression; Odds Ratio (OR) = 1.50, 95% CI 2-sided [1.16 to 1.93]
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 44, analysis 1]; Test type: Superiority; p = 0.023, Logistic regression; Odds Ratio (OR) = 1.34, 95% CI 2-sided [1.04 to 1.73]

45. Secondary Outcome: Percentage of Participants With ≥ 10 Points Improvement From Baseline in the OAB-q Symptom Bother Score at Weeks 4, 8, 12 and EoT
Description: The percentage of participants with ≥ 10 points improvement from baseline to each visit (weeks 4, 8, 12 and EoT).
Time Frame: Weeks 4, 8, 12 and EoT (up to 12 weeks)
Population: FAS participants with available data at each time point were included in the analysis. LOCF was used for EoT.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
percentage of participants
  Week 4: number analyzed (Participants) | 397 | 388 | 392 | 394 | 790 | 789
  Week 4 | 56.4 | 62.6 | 69.9 | 73.9 | 73.9 | 75.8
  Week 8: number analyzed (Participants) | 381 | 370 | 380 | 385 | 757 | 761
  Week 8 | 62.2 | 71.6 | 73.4 | 79.2 | 83.9 | 82.8
  Week 12: number analyzed (Participants) | 371 | 362 | 366 | 374 | 738 | 734
  Week 12 | 66.0 | 72.1 | 78.4 | 82.4 | 83.5 | 85.1
  End of treatment: number analyzed (Participants) | 400 | 392 | 398 | 399 | 800 | 795
  End of treatment | 65.3 | 71.2 | 77.1 | 81.2 | 82.8 | 84.3
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; Odds ratio from a logistic regression model including treatment group, sex, age group (<65, >=65 years), previous OAB medication (yes, no) and geographic region as factors and baseline OAB-q subscale as a covariate; Test type: Superiority; p = 0.224, Logistic regression; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.88 to 1.69]
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 45, analysis 1]; Test type: Superiority; p = 0.037, Logistic regression; Odds Ratio (OR) = 1.42, 95% CI 2-sided [1.02 to 1.96]
Statistical Analysis 3: Comparison: Mirabegron 25 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 45, analysis 1]; Test type: Superiority; p < 0.001, Logistic regression; Odds Ratio (OR) = 1.98, 95% CI 2-sided [1.47 to 2.67]
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 45, analysis 1]; Test type: Superiority; p = 0.002, Logistic regression; Odds Ratio (OR) = 1.65, 95% CI 2-sided [1.21 to 2.26]

46. Secondary Outcome: Percentage of Participants With ≥ 10 Points Improvement From Baseline in HRQL Total Score at Weeks 4, 8, 12 and EoT
Description: The percentage of participants with ≥ 10 points improvement from baseline to each visit (weeks 4, 8, 12 and EoT).
Time Frame: Weeks 4, 8, 12 and EoT (up to 12 weeks)
Population: FAS participants with available data at each time point were included in the analysis. LOCF was used for EoT.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
percentage of participants
  Week 4: number analyzed (Participants) | 397 | 388 | 392 | 394 | 790 | 789
  Week 4 | 45.3 | 52.8 | 59.7 | 61.7 | 62.9 | 61.3
  Week 8: number analyzed (Participants) | 381 | 370 | 380 | 385 | 757 | 761
  Week 8 | 51.2 | 62.2 | 65.3 | 66.2 | 71.5 | 69.3
  Week 12: number analyzed (Participants) | 371 | 362 | 366 | 374 | 738 | 734
  Week 12 | 57.7 | 62.4 | 69.1 | 71.7 | 76.3 | 71.8
  End of treatment: number analyzed (Participants) | 400 | 392 | 398 | 399 | 800 | 795
  End of treatment | 56.8 | 61.0 | 68.3 | 71.2 | 74.5 | 71.1
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 45, analysis 1]; Test type: Superiority; p = 0.077, Logistic regression; Odds Ratio (OR) = 1.29, 95% CI 2-sided [0.97 to 1.72]
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Odds ratio from a logistic regression model treatment group, sex, age group (<65, >=65 years), previous OAB medication (yes, no) and geographic region as factors and baseline OAB-q subscale as a covariate; Test type: Superiority; p = 0.321, Logistic regression; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.87 to 1.53]
Statistical Analysis 3: Comparison: Mirabegron 25 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 45, analysis 1]; Test type: Superiority; p < 0.001, Logistic regression; Odds Ratio (OR) = 1.92, 95% CI 2-sided [1.46 to 2.53]
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 45, analysis 1]; Test type: Superiority; p = 0.294, Logistic regression; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.88 to 1.53]

47. Secondary Outcome: Percentage of Participants With 50% Reduction in Mean Number of Incontinence Episodes Per 24 Hours at Weeks 4, 8, 12 and EoT
Description: The percentage of participants with ≥ 50% decrease from baseline in mean number of incontinence episodes per 24 hours at each time point (weeks 4, 8, 12 and EoT).
Time Frame: Weeks 4, 8, 12 and EoT (up to 12 weeks)
Population: FAS participants with available data at each time point were included in the analysis. LOCF was used for EoT.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
percentage of participants
  Week 4: number analyzed (Participants) | 406 | 406 | 402 | 402 | 817 | 810
  Week 4 | 41.1 | 45.3 | 56.7 | 53.2 | 57.2 | 60.6
  Week 8: number analyzed (Participants) | 397 | 385 | 386 | 386 | 784 | 769
  Week 8 | 54.9 | 61.8 | 63.7 | 65.3 | 69.8 | 70.6
  Week 12: number analyzed (Participants) | 374 | 369 | 369 | 379 | 754 | 750
  Week 12 | 58.6 | 66.4 | 70.2 | 71.0 | 75.9 | 76.1
  End of treatment: number analyzed (Participants) | 412 | 409 | 406 | 413 | 823 | 816
  End of treatment | 59.5 | 64.5 | 69.0 | 70.5 | 74.5 | 75.7
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 44, analysis 1]; Test type: Superiority; p = 0.251, Logistic regression; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.89 to 1.53]
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 44, analysis 1]; Test type: Superiority; p = 0.107, Logistic regression; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.95 to 1.64]
Statistical Analysis 3: Comparison: Mirabegron 25 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 44, analysis 1]; Test type: Superiority; p < 0.001, Logistic regression; Odds Ratio (OR) = 1.59, 95% CI 2-sided [1.23 to 2.07]
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 44, analysis 1]; Test type: Superiority; p = 0.012, Logistic regression; Odds Ratio (OR) = 1.41, 95% CI 2-sided [1.08 to 1.85]

48. Secondary Outcome: Percentage of Participants for Micturition Frequency Normalization at Weeks 4, 8, 12 and EoT
Description: The percentage of participants with micturition frequency normalization was defined as any participant who had ≥ 8 micturitions/24 hours at baseline and < 8 micturitions/24 h postbaseline at weeks 4, 8, 12 and EoT.
Time Frame: Weeks 4, 8 , 12 and EoT (up to 12 weeks)
Population: FAS participants with available data at each time point were included in the analysis. LOCF was used for EoT.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
percentage of participants
  Week 4: number analyzed (Participants) | 406 | 406 | 402 | 402 | 817 | 810
  Week 4 | 24.1 | 30.8 | 25.4 | 31.1 | 36.0 | 37.7
  Week 8: number analyzed (Participants) | 397 | 385 | 386 | 386 | 784 | 769
  Week 8 | 28.7 | 37.9 | 34.5 | 37.0 | 45.3 | 49.0
  Week 12: number analyzed (Participants) | 374 | 369 | 369 | 379 | 754 | 750
  Week 12 | 29.7 | 42.3 | 40.7 | 44.9 | 50.8 | 53.1
  End of treatment: number analyzed (Participants) | 412 | 409 | 406 | 413 | 823 | 816
  End of treatment | 31.1 | 42.1 | 40.1 | 45.0 | 51.3 | 52.6
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; Odds ratio from a logistic regression model including treatment group, sex, age group (<65, >=65 years), previous OAB medication (yes, no) and geographic region as factors and baseline mean number of micturitions per 24 hours as a covariate; Test type: Superiority; p = 0.044, Logistic regression; Odds Ratio (OR) = 1.30, 95% CI 2-sided [1.01 to 1.67]
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 48, analysis 1]; Test type: Superiority; p = 0.006, Logistic regression; Odds Ratio (OR) = 1.43, 95% CI 2-sided [1.11 to 1.84]
Statistical Analysis 3: Comparison: Mirabegron 25 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 48, analysis 1]; Test type: Superiority; p = 0.004, Logistic regression; Odds Ratio (OR) = 1.47, 95% CI 2-sided [1.13 to 1.90]
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 48, analysis 1]; Test type: Superiority; p < 0.001, Logistic regression; Odds Ratio (OR) = 1.60, 95% CI 2-sided [1.23 to 2.08]

49. Secondary Outcome: Percentage of Participants With Zero Incontinence Episodes Per 24 Hours Using the Last 7 Diary Days at Weeks 4, 8, 12 and EoT
Description: The percentage of participants with zero incontinence episodes per 24 hours postbaseline in the last 7 days prior to weeks 4, 8, 12 and EoT.
Time Frame: Weeks 4, 8, 12 and EoT (up to 12 weeks)
Population: FAS participants with available data at each time point were included in the analysis. LOCF was used for EoT.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
percentage of participants
  Week 4: number analyzed (Participants) | 406 | 406 | 402 | 402 | 817 | 810
  Week 4 | 12.8 | 13.1 | 16.7 | 17.7 | 23.9 | 26.0
  Week 8: number analyzed (Participants) | 397 | 385 | 386 | 386 | 784 | 769
  Week 8 | 19.1 | 24.4 | 29.8 | 28.2 | 36.6 | 38.4
  Week 12: number analyzed (Participants) | 374 | 369 | 369 | 379 | 754 | 750
  Week 12 | 29.1 | 32.2 | 35.0 | 31.9 | 42.4 | 43.7
  End of treatment: number analyzed (Participants) | 412 | 409 | 406 | 413 | 823 | 816
  End of treatment | 28.6 | 30.6 | 34.0 | 31.5 | 40.9 | 43.1
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; Odds ratio from a logistic regression model including treatment group, sex, age group (<65, >=65 years), previous OAB medication (yes, no) and geographic region as factors and baseline mean number of incontinence episodes per 24 hours as a covariate; Test type: Superiority; p = 0.004, Logistic regression; Odds Ratio (OR) = 1.47, 95% CI 2-sided [1.13 to 1.92]
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 49, analysis 1]; Test type: Superiority; p < 0.001, Logistic regression; Odds Ratio (OR) = 1.62, 95% CI 2-sided [1.24 to 2.11]
Statistical Analysis 3: Comparison: Mirabegron 25 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 49, analysis 1]; Test type: Superiority; p = 0.001, Logistic regression; Odds Ratio (OR) = 1.59, 95% CI 2-sided [1.22 to 2.07]
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 49, analysis 1]; Test type: Superiority; p = 0.001, Logistic regression; Odds Ratio (OR) = 1.57, 95% CI 2-sided [1.21 to 2.04]

50. Secondary Outcome: Percentage of Participants With ≥ 1 Point Improvement From Baseline in PPBC at Weeks 4, 8, 12 and EoT
Description: The percentage of participants with ≥ 1 point improvement from baseline in PPBC at weeks 4, 8, 12 and EoT.
Time Frame: Weeks 4, 8, 12 and EoT (up to 12 weeks)
Population: FAS participants with available data at each time point were included in the analysis. LOCF was used for EoT.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
percentage of participants
  Week 4: number analyzed (Participants) | 397 | 388 | 393 | 394 | 791 | 791
  Week 4 | 48.9 | 52.8 | 60.3 | 58.1 | 63.1 | 62.7
  Week 8: number analyzed (Participants) | 381 | 372 | 380 | 385 | 758 | 761
  Week 8 | 56.4 | 65.3 | 69.7 | 72.7 | 71.6 | 75.4
  Week 12: number analyzed (Participants) | 371 | 362 | 366 | 375 | 739 | 735
  Week 12 | 59.8 | 66.9 | 73.8 | 74.1 | 76.6 | 80.0
  End of treaetment: number analyzed (Participants) | 400 | 393 | 398 | 399 | 801 | 795
  End of treaetment | 59.8 | 65.4 | 72.4 | 71.9 | 75.7 | 78.4
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; Odds ratio from a logistic regression model including treatment group, sex, age group (<65, >=65 years), previous OAB medication (yes, no) and geographic region as factors and baseline PPBC as a covariate; Test type: Superiority; p = 0.065, Logistic regression; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.98 to 1.78]
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 50, analysis 1]; Test type: Superiority; p = 0.001, Logistic regression; Odds Ratio (OR) = 1.68, 95% CI 2-sided [1.24 to 2.27]
Statistical Analysis 3: Comparison: Mirabegron 25 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 50, analysis 1]; Test type: Superiority; p < 0.001, Logistic regression; Odds Ratio (OR) = 1.76, 95% CI 2-sided [1.32 to 2.36]
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 50, analysis 1]; Test type: Superiority; p = 0.007, Logistic regression; Odds Ratio (OR) = 1.51, 95% CI 2-sided [1.12 to 2.04]

51. Secondary Outcome: Percentage of Participants With Major (≥ 2 Points) Improvement From Baseline in PPBC at Weeks 4, 8, 12 and EoT
Description: The percentage of participants with a major (≥ 2 points) improvement from baseline in PPBC at weeks 4, 8, 12 and EoT.
Time Frame: Weeks 4, 8, 12 and EoT (up to 12 weeks)
Population: FAS participants with available data at each time point were included in the analysis. LOCF was used for EoT.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
percentage of participants
  Week 4: number analyzed (Participants) | 397 | 388 | 393 | 384 | 791 | 791
  Week 4 | 15.9 | 20.6 | 22.4 | 27.4 | 31.1 | 31.1
  Week 8: number analyzed (Participants) | 381 | 372 | 380 | 385 | 758 | 761
  Week 8 | 27.0 | 33.3 | 35.0 | 40.5 | 42.7 | 46.4
  Week 12: number analyzed (Participants) | 371 | 362 | 366 | 375 | 739 | 735
  Week 12 | 29.6 | 39.0 | 42.3 | 44.5 | 50.7 | 52.9
  End of treatment: number analyzed (Participants) | 400 | 393 | 398 | 399 | 801 | 795
  End of treatment | 29.5 | 37.2 | 40.7 | 42.6 | 49.7 | 51.2
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 50, analysis 1]; Test type: Superiority; p = 0.007, Logistic regression; Odds Ratio (OR) = 1.44, 95% CI 2-sided [1.11 to 1.87]
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 50, analysis 1]; Test type: Superiority; p < 0.001, Logistic regression; Odds Ratio (OR) = 1.67, 95% CI 2-sided [1.28 to 2.17]
Statistical Analysis 3: Comparison: Mirabegron 25 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 50, analysis 1]; Test type: Superiority; p < 0.001, Logistic regression; Odds Ratio (OR) = 1.76, 95% CI 2-sided [1.34 to 2.30]
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 50, analysis 1]; Test type: Superiority; p < 0.001, Logistic regression; Odds Ratio (OR) = 1.68, 95% CI 2-sided [1.29 to 2.19]

52. Secondary Outcome: Percentage of Participants Who Were Double Responders (50% Reduction in Mean Number of Incontinence Episodes Per 24 Hours and at Least 10 Points Improvement on OAB-q Symptom Bother Scale) at Weeks 4, 8, 12 and EoT
Description: The percentage of participants considered as double responders, defined as participants with 50% reduction in mean number of incontinence episodes per 24 hours compared to baseline and minimal important difference reached (improvement by ≥ 10 points) on the OAB-q Symptom Bother score at weeks 4, 8, 12 and EoT.
Time Frame: Weeks 4, 8, 12 and EoT (up to 12 weeks)
Population: FAS participants with available data at each time point were included in the analysis. LOCF was used for EoT.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
percentage of participants
  Week 4: number analyzed (Participants) | 388 | 385 | 387 | 385 | 784 | 778
  Week 4 | 28.6 | 34.8 | 45.7 | 44.9 | 47.8 | 52.3
  Week 8: number analyzed (Participants) | 374 | 366 | 375 | 372 | 750 | 742
  Week 8 | 39.8 | 50.0 | 51.5 | 56.5 | 63.1 | 63.5
  Week 12: number analyzed (Participants) | 360 | 350 | 355 | 363 | 727 | 721
  Week 12 | 45.0 | 55.7 | 59.4 | 63.1 | 66.7 | 69.5
  End of treatment: number analyzed (Participants) | 396 | 391 | 395 | 398 | 798 | 790
  End of treatment | 45.2 | 54.0 | 58.2 | 62.6 | 65.2 | 68.2
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; Odds ratio from a logistic regression model including treatment group, sex, age group (<65, >=65 years), previous OAB medication (yes, no) and geographic region as factors, and baseline mean number of incontinence episodes per 24 hours and baseline OAB-q symptom bother scale as covariates; Test type: Superiority; p = 0.381, Logistic regression; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.87 to 1.45]
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 52, analysis 1]; Test type: Superiority; p = 0.040, Logistic regression; Odds Ratio (OR) = 1.31, 95% CI 2-sided [1.01 to 1.70]
Statistical Analysis 3: Comparison: Mirabegron 25 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 52, analysis 1]; Test type: Superiority; p = 0.001, Logistic regression; Odds Ratio (OR) = 1.56, 95% CI 2-sided [1.21 to 2.00]
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 52, analysis 1]; Test type: Superiority; p = 0.001, Logistic regression; Odds Ratio (OR) = 1.57, 95% CI 2-sided [1.21 to 2.03]

53. Secondary Outcome: Percentage of Participants Who Were Double Responders (50% Reduction in Mean Number of Incontinence Episodes Per 24 Hours and at Least 10 Points Improvement on OAB-q HRQL Total Score) at Weeks 4, 8, 12 and EoT
Description: The percentage of participants considered as double responders, defined as participants with 50% reduction in mean number of incontinence episodes per 24 hours compared to baseline and minimal important difference reached (improvement by ≥ 10 points) on the OAB-q HRQL total score at weeks 4, 8, 12 and EoT.
Time Frame: Weeks 4, 8, 12 and EoT (up to 12 weeks)
Population: FAS participants with available data at each time point were included in the analysis. LOCF was used for EoT.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
percentage of participants
  Week 4: number analyzed (Participants) | 388 | 385 | 387 | 385 | 784 | 778
  Week 4 | 23.2 | 28.3 | 39.8 | 37.7 | 40.4 | 40.5
  Week 8: number analyzed (Participants) | 374 | 366 | 375 | 372 | 750 | 742
  Week 8 | 32.9 | 43.2 | 46.1 | 48.4 | 54.1 | 53.0
  Week 12: number analyzed (Participants) | 360 | 350 | 355 | 363 | 727 | 721
  Week 12 | 39.2 | 48.3 | 53.5 | 54.8 | 61.6 | 59.2
  End of treatment: number analyzed (Participants) | 396 | 391 | 395 | 398 | 798 | 790
  End of treatment | 39.1 | 46.0 | 52.9 | 54.0 | 59.0 | 58.2
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; Odds ratio from a logistic regression model including treatment group, sex, age group (<65, >=65 years), previous OAB medication (yes, no) and geographic region as factors, and baseline mean number of incontinence episodes per 24 hours and baseline OAB-q HRQL total score as covariates; Test type: Superiority; p = 0.095, Logistic regression; Odds Ratio (OR) = 1.24, 95% CI 2-sided [0.96 to 1.59]
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 53, analysis 1]; Test type: Superiority; p = 0.073, Logistic regression; Odds Ratio (OR) = 1.26, 95% CI 2-sided [0.98 to 1.62]
Statistical Analysis 3: Comparison: Mirabegron 25 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 53, analysis 1]; Test type: Superiority; p < 0.001, Logistic regression; Odds Ratio (OR) = 1.66, 95% CI 2-sided [1.29 to 2.13]
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 53, analysis 1]; Test type: Superiority; p = 0.067, Logistic regression; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.98 to 1.63]

54. Secondary Outcome: Percentage of Participants Who Were Double Responders (50% Reduction in Mean Number of Incontinence Episodes Per 24 Hours and at Least 1 Point Improvement on PPBC) at Weeks 4, 8, 12 and EoT
Description: The percentage of participants considered as double responders, defined as participants with 50% reduction in mean number of incontinence episodes per 24 hours compared to baseline and ≥ 1 point improvement from baseline in PPBC at weeks 4, 8, 12 and EoT.
Time Frame: Weeks 4, 8, 12 and EoT (up to 12 weeks)
Population: FAS participants with available data at each time point were included in the analysis. LOCF was used for EoT.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
percentage of participants
  Week 4: number analyzed (Participants) | 388 | 384 | 387 | 385 | 785 | 780
  Week 4 | 23.2 | 27.9 | 37.7 | 34.5 | 39.9 | 42.9
  Week 8: number analyzed (Participants) | 374 | 367 | 375 | 372 | 751 | 742
  Week 8 | 35.6 | 44.7 | 50.1 | 51.3 | 53.8 | 57.7
  Week 12: number analyzed (Participants) | 360 | 350 | 355 | 364 | 728 | 722
  Week 12 | 40.6 | 51.7 | 54.9 | 56.9 | 62.0 | 65.4
  End of treatment: number analyzed (Participants) | 396 | 392 | 395 | 398 | 799 | 790
  End of treatment | 40.9 | 48.5 | 53.9 | 56.0 | 59.9 | 63.8
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; Odds ratio from a logistic regression model including treatment group, sex, age group (<65, >=65 years), previous OAB medication (yes, no) and geographic region as factors, and baseline mean number of lncontinence episodes per 24 hours and baseline PPBC as covariates; Test type: Superiority; p = 0.210, Logistic regression; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.91 to 1.52]
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 54, analysis 1]; Test type: Superiority; p = 0.004, Logistic regression; Odds Ratio (OR) = 1.46, 95% CI 2-sided [1.13 to 1.89]
Statistical Analysis 3: Comparison: Mirabegron 25 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 54, analysis 1]; Test type: Superiority; p < 0.001, Logistic regression; Odds Ratio (OR) = 1.59, 95% CI 2-sided [1.23 to 2.06]
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 54, analysis 1]; Test type: Superiority; p < 0.001, Logistic regression; Odds Ratio (OR) = 1.59, 95% CI 2-sided [1.23 to 2.05]

55. Secondary Outcome: Percentage of Participants Who Were Triple Responders (50% Reduction in Mean Number of Incontinence Episodes Per 24 Hours, at Least 10 Points Improvement on OAB-q Symptom Bother Scale and at Least 1 Point Improvement on PPBC) at Weeks 4, 8, 12 and EoT
Description: The percentage of participants considered as triple responders, defined as participants with 50% reduction in mean number of incontinence episodes per 24 hours compared to baseline, minimal important difference reached (improvement by ≥ 10 points) on the OAB-q Symptom Bother score, and ≥ 1 point improvement from baseline in PPBC at weeks 4, 8, 12 and EoT.
Time Frame: Weeks 4, 8, 12 and EoT (up to 12 weeks)
Population: FAS participants with available data at each time point were included in the analysis. LOCF was used for EoT.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
percentage of participants
  Week 4: number analyzed (Participants) | 388 | 384 | 387 | 385 | 784 | 778
  Week 4 | 17.8 | 24.0 | 33.6 | 31.4 | 37.5 | 40.2
  Week 8: number analyzed (Participants) | 374 | 366 | 375 | 372 | 750 | 742
  Week 8 | 29.7 | 41.3 | 43.2 | 47.8 | 51.6 | 54.7
  Week 12: number analyzed (Participants) | 360 | 350 | 355 | 363 | 727 | 721
  Week 12 | 35.8 | 47.7 | 49.6 | 54.5 | 58.2 | 62.0
  End of treatment: number analyzed (Participants) | 396 | 391 | 395 | 398 | 798 | 790
  End of treatment | 36.1 | 45.0 | 48.4 | 53.3 | 56.3 | 60.3
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; Odds ratio from a logistic regression model including treatment group, sex, age group (<65, >=65 years), previous OAB medication (yes, no) and geographic region as factors, and baseline mean number of incontinence episodes per 24 hours, baseline OAB-q symptom bother scale and baseline PPBC as covariates; Test type: Superiority; p = 0.335, Logistic regression; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.88 to 1.46]
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 55, analysis 1]; Test type: Superiority; p = 0.009, Logistic regression; Odds Ratio (OR) = 1.40, 95% CI 2-sided [1.09 to 1.81]
Statistical Analysis 3: Comparison: Mirabegron 25 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 55, analysis 1]; Test type: Superiority; p = 0.001, Logistic regression; Odds Ratio (OR) = 1.56, 95% CI 2-sided [1.21 to 2.02]
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 55, analysis 1]; Test type: Superiority; p < 0.001, Logistic regression; Odds Ratio (OR) = 1.71, 95% CI 2-sided [1.33 to 2.21]

56. Secondary Outcome: Percentage of Participants Who Were Triple Responders (50% Reduction in Mean Number of Incontinence Episodes Per 24 Hours, at Least 10 Points Improvement on OAB-q HRQL Total Score and at Least 1 Point Improvement on PPBC) at Weeks 4, 8, 12 and EoT
Description: The percentage of participants considered as triple responders, defined as participants with 50% reduction in mean number of incontinence episodes per24 hours compared to baseline, minimal important difference reached (improvement by ≥ 10 points) on the HRQL total score, and ≥ 1 point improvement from baseline in PPBC at weeks 4, 8, 12 and EoT.
Time Frame: Weeks 4, 8, 12 and EoT (up to 12 weeks)
Population: FAS participants with available data at each time point were included in the analysis. LOCF was used for EoT.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 418 | 410 | 411 | 415 | 827 | 827
percentage of participants
  Week 4: number analyzed (Participants) | 388 | 384 | 387 | 385 | 784 | 778
  Week 4 | 15.2 | 20.6 | 30.0 | 28.6 | 32.7 | 33.4
  Week 8: number analyzed (Participants) | 374 | 366 | 375 | 372 | 750 | 742
  Week 8 | 24.9 | 36.9 | 38.9 | 43.0 | 46.3 | 46.8
  Week 12: number analyzed (Participants) | 360 | 350 | 355 | 363 | 727 | 721
  Week 12 | 33.3 | 42.0 | 45.6 | 49.9 | 54.5 | 54.2
  End of treatment: number analyzed (Participants) | 396 | 391 | 395 | 398 | 798 | 790
  End of treatment | 33.3 | 39.1 | 44.8 | 49.2 | 51.6 | 52.8
Statistical Analysis 1: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 25 mg; Odds ratio from a logistic regression model including treatment group, sex, age group (<65, >=65 years), previous OAB medication (yes, no) and geographic region as factors, and baseline mean number of incontinence episodes per 24 hours, baseline OAB-q HRQL total score and baseline PPBC as covariates; Test type: Superiority; p = 0.416, Logistic regression; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.86 to 1.43]
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 56, analysis 1]; Test type: Superiority; p = 0.105, Logistic regression; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.96 to 1.59]
Statistical Analysis 3: Comparison: Mirabegron 25 mg vs Solifenacin 5 mg + Mirabegron 25 mg; [analysis description as in outcome 56, analysis 1]; Test type: Superiority; p < 0.001, Logistic regression; Odds Ratio (OR) = 1.66, 95% CI 2-sided [1.28 to 2.16]
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 56, analysis 1]; Test type: Superiority; p = 0.005, Logistic regression; Odds Ratio (OR) = 1.45, 95% CI 2-sided [1.12 to 1.87]

57. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: A TEAE refered to an adverse event (AE; defined as any untoward medical occurrence in a participant administered a study drug or who had undergone study procedures and did not necessarily have a causal relationship with this treatment) which started or worsened in the period from first double-blind medication intake until 14 days after the last double-blind medication intake. Serious TEAEs with a start date reported until 30 days after the last double-blind medication intake were also summarized as TEAEs, and also included serious TEAEs upgraded by the sponsor based on review of the sponsor's list of Always Serious terms if any upgrade was done. Drug-related TEAEs may be possible or probable, as assessed by the investigator, or records where relationship is missing.
Time Frame: From first dose of double-blind study drug up to 30 days after last dose of double-blind study drug (up to 16 weeks)
Population: Safety Analysis Set (SAF), which comprised all randomized participants who received ≥ 1 dose of double-blind treatment and excluded participants from one site.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 429 | 423 | 422 | 423 | 853 | 848
Participants
  Any TEAE | 145 | 135 | 147 | 149 | 345 | 314
  Drug-related TEAEs | 45 | 37 | 52 | 63 | 157 | 150
  Deaths | 0 | 0 | 0 | 0 | 0 | 0
  Serious TEAEs | 8 | 6 | 5 | 3 | 12 | 19
  Drug-related serious TEAEs | 0 | 1 | 1 | 0 | 2 | 3
  TEAEs leading to discontinuation | 9 | 7 | 10 | 7 | 20 | 22
  Drug-related TEAEs leading to discontinuation | 7 | 4 | 6 | 5 | 17 | 19

58. Secondary Outcome: Change From Baseline to Weeks 4, 8, 12 and EoT in Postvoid Residual (PVR) Volume
Description: PVR volume was assessed by ultrasonography or a bladder scanner.
Time Frame: Baseline and weeks 4, 8, 12 and EoT (up to 12 weeks)
Population: SAF participants with available data at each time point were included in the analysis. LOCF was used for EoT.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 429 | 423 | 422 | 423 | 853 | 848
mL
  Week 4: number analyzed (Participants) | 408 | 397 | 398 | 412 | 815 | 812
  Week 4 | -0.8 (29.9) | 1.6 (28.0) | -2.1 (29.7) | 5.8 (35.6) | 7.2 (47.7) | 10.6 (51.1)
  Week 8: number analyzed (Participants) | 393 | 378 | 383 | 393 | 779 | 784
  Week 8 | -1.9 (28.6) | -0.4 (29.8) | -0.6 (34.4) | 5.4 (35.2) | 7.0 (37.4) | 9.9 (46.0)
  Week 12: number analyzed (Participants) | 382 | 376 | 370 | 383 | 766 | 763
  Week 12 | -1.0 (29.9) | 1.0 (29.8) | 0.0 (30.1) | 4.7 (33.1) | 7.9 (44.4) | 9.6 (50.1)
  End of treatment: number analyzed (Participants) | 410 | 401 | 404 | 414 | 821 | 815
  End of treatment | -1.0 (29.4) | 0.7 (29.1) | -0.8 (30.0) | 4.8 (33.3) | 9.0 (55.0) | 11.0 (54.9)

59. Secondary Outcome: Change From Baseline to Weeks 4, 12 and EoT in Mean 24-hours, Mean Daytime and Mean Nighttime Systolic Blood Pressure (SBP)
Description: Vital signs (blood pressure and pulse rate) were monitored using an ambulatory blood pressure monitoring (ABPM) device placed on the upper arm followed by intake of the double-blind study medication and worn for at least 24 hours.
Time Frame: Baseline and weeks 4, 12 and EoT (up to 12 weeks)
Population: ABPM analysis set (ABPMAS), which consisted of all participants in the SAF for whom at least 1 ABPM variable could be calculated at baseline and postbaseline visit. Participants with data available at each time point were included in the analysis. LOCF was used for EoT.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 92 | 85 | 87 | 86 | 176 | 189
mmHg
  Week 4: 24-hour mean: number analyzed (Participants) | 76 | 66 | 67 | 72 | 141 | 157
  Week 4: 24-hour mean | -1.00 (1.22) | -2.04 (1.31) | 0.96 (1.30) | 1.03 (1.26) | -0.85 (0.90) | 0.31 (0.85)
  Week 4: mean daytime: number analyzed (Participants) | 72 | 60 | 62 | 60 | 129 | 147
  Week 4: mean daytime | -1.55 (1.22) | -1.19 (1.33) | -0.67 (1.31) | -1.13 (1.34) | -1.63 (0.91) | -0.53 (0.85)
  Week 4: mean nighttime: number analyzed (Participants) | 82 | 74 | 75 | 72 | 147 | 161
  Week 4: mean nighttime | -0.51 (1.38) | -1.14 (1.46) | 1.42 (1.44) | 0.41 (1.47) | 1.14 (1.03) | 0.54 (0.98)
  Week 12: 24-hour mean: number analyzed (Participants) | 67 | 62 | 63 | 60 | 121 | 139
  Week 12: 24-hour mean | -1.97 (1.37) | -2.70 (1.42) | -1.75 (1.41) | 0.40 (1.45) | -0.71 (1.02) | 0.40 (0.95)
  Week 12: mean daytime: number analyzed (Participants) | 65 | 56 | 55 | 53 | 106 | 116
  Week 12: mean daytime | -2.22 (1.37) | -2.53 (1.46) | -2.14 (1.48) | -2.09 (1.50) | -0.39 (1.06) | -0.71 (1.02)
  Week 12: mean nighttime: number analyzed (Participants) | 75 | 64 | 71 | 65 | 132 | 146
  Week 12: mean nighttime | -1.03 (1.64) | -2.81 (1.77) | -0.77 (1.68) | 1.31 (1.76) | 0.11 (1.23) | 0.79 (1.17)
  End of treatment: 24-hour mean: number analyzed (Participants) | 80 | 73 | 76 | 78 | 150 | 168
  End of treatment: 24-hour mean | -1.73 (1.24) | -3.44 (1.29) | -1.14 (1.27) | 0.37 (1.25) | -0.52 (0.90) | -0.08 (0.85)
  End of treatment: mean daytime: number analyzed (Participants) | 78 | 67 | 69 | 69 | 137 | 153
  End of treatment: mean daytime | -2.01 (1.22) | -3.29 (1.31) | -1.92 (1.30) | -2.17 (1.30) | -0.68 (0.92) | -1.28 (0.87)
  End of treatment: mean nighttime: number analyzed (Participants) | 88 | 80 | 82 | 82 | 160 | 175
  End of treatment: mean nighttime | -1.00 (1.47) | -3.48 (1.54) | -0.60 (1.52) | 1.42 (1.52) | 0.41 (1.09) | 0.91 (1.04)

60. Secondary Outcome: Change From Baseline to Weeks 4, 12 and EoT in Mean 24-h, Mean Daytime and Mean Nighttime Diastolic Blood Pressure (DBP)
Description: Vital signs (blood pressure and pulse rate) were monitored using ABPM device placed on the upper arm followed by intake of the double-blind study medication and worn for at least 24 hours.
Time Frame: Baseline and weeks 4, 12 and EoT (up to 12 weeks)
Population: ABPMAS participants with available data at each time point were included in the analysis. LOCF was used for EoT.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 92 | 85 | 87 | 86 | 176 | 189
mmHg
  Week 4: 24-hour mean: number analyzed (Participants) | 76 | 66 | 67 | 72 | 141 | 157
  Week 4: 24-hour mean | -0.70 (0.50) | -0.86 (0.54) | 0.22 (0.54) | 0.25 (0.52) | 0.03 (0.37) | 0.38 (0.35)
  Week 4: mean daytime: number analyzed (Participants) | 72 | 60 | 62 | 60 | 129 | 147
  Week 4: mean daytime | -1.25 (0.53) | -0.36 (0.58) | -0.33 (0.57) | -0.77 (0.58) | -0.40 (0.40) | 0.07 (0.37)
  Week 4: mean nighttime: number analyzed (Participants) | 82 | 74 | 75 | 72 | 147 | 161
  Week 4: mean nighttime | -0.12 (0.59) | -0.97 (0.62) | 0.40 (0.62) | 0.48 (0.63) | 0.93 (0.44) | 0.47 (0.42)
  Week 12: 24-hour mean: number analyzed (Participants) | 67 | 62 | 63 | 60 | 121 | 139
  Week 12: 24-hour mean | -0.80 (0.56) | -0.93 (0.58) | -0.19 (0.57) | 0.43 (0.59) | -0.37 (0.41) | 0.31 (0.39)
  Week 12: mean daytime: number analyzed (Participants) | 65 | 56 | 55 | 53 | 106 | 116
  Week 12: mean daytime | -0.85 (0.60) | -0.54 (0.64) | -0.40 (0.65) | -0.33 (0.66) | -0.06 (0.46) | -0.18 (0.44)
  Week 12: mean nighttime: number analyzed (Participants) | 75 | 64 | 71 | 65 | 132 | 146
  Week 12: mean nighttime | -0.49 (0.66) | -1.39 (0.71) | -0.03 (0.68) | 0.92 (0.71) | 0.23 (0.49) | 0.49 (0.47)
  End of treatment: 24-hour mean: number analyzed (Participants) | 80 | 73 | 76 | 78 | 150 | 168
  End of treatment: 24-hour mean | -0.96 (0.51) | -1.41 (0.53) | -0.11 (0.52) | 0.05 (0.52) | -0.02 (0.37) | 0.25 (0.35)
  End of treatment: mean daytime: number analyzed (Participants) | 78 | 67 | 69 | 69 | 137 | 153
  End of treatment: mean daytime | -1.17 (0.53) | -0.98 (0.58) | -0.69 (0.57) | -0.79 (0.57) | -0.18 (0.40) | -0.36 (0.38)
  End of treatment: mean nighttime: number analyzed (Participants) | 88 | 80 | 82 | 82 | 160 | 175
  End of treatment: mean nighttime | -0.41 (0.60) | -2.00 (0.63) | 0.08 (0.63) | 0.71 (0.63) | 0.56 (0.45) | 0.61 (0.43)

61. Secondary Outcome: Change From Baseline to Weeks 4, 12 and EoT in Mean 24-h, Mean Daytime and Mean Nighttime Pulse Rate (PR)
Description: Vital signs (blood pressure and pulse rate) were monitored using an ABPM device placed on the upper arm followed by intake of the double-blind study medication and worn for at least 24 hours.
Time Frame: Baseline and weeks 4, 12 and EoT (up to 12 weeks)
Population: ABPMAS participants with available data at each time point were included in the analysis. LOCF was used for EoT.
Measure: Least Squares Mean (Standard Error); unit: beats per minute (bpm)
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 92 | 85 | 87 | 86 | 176 | 189
beats per minute (bpm)
  Week 4: 24-hour mean: number analyzed (Participants) | 76 | 66 | 67 | 72 | 141 | 157
  Week 4: 24-hour mean | -0.83 (0.63) | 1.14 (0.68) | 2.32 (0.67) | 0.36 (0.65) | 0.40 (0.46) | 0.69 (0.44)
  Week 4: mean daytime: number analyzed (Participants) | 72 | 60 | 62 | 60 | 129 | 147
  Week 4: mean daytime | -0.70 (0.73) | 1.19 (0.79) | 3.52 (0.78) | 0.37 (0.80) | -0.05 (0.54) | 0.61 (0.51)
  Week 4: mean nighttime: number analyzed (Participants) | 82 | 74 | 75 | 72 | 147 | 161
  Week 4: mean nighttime | -0.72 (0.68) | 0.98 (0.71) | 1.77 (0.70) | 1.09 (0.72) | 0.86 (0.50) | 0.86 (0.48)
  Week 12: 24-hour mean: number analyzed (Participants) | 67 | 62 | 63 | 60 | 121 | 139
  Week 12: 24-hour mean | 0.70 (0.72) | 0.38 (0.74) | 1.19 (0.74) | 0.12 (0.76) | 0.94 (0.53) | 1.44 (0.50)
  Week 12: mean daytime: number analyzed (Participants) | 65 | 56 | 55 | 53 | 106 | 116
  Week 12: mean daytime | 0.89 (0.82) | 0.25 (0.88) | 2.12 (0.89) | -0.13 (0.90) | 0.84 (0.64) | 1.36 (0.61)
  Week 12: mean nighttime: number analyzed (Participants) | 75 | 64 | 71 | 65 | 132 | 146
  Week 12: mean nighttime | 0.34 (0.71) | 0.21 (0.77) | 0.19 (0.73) | 0.06 (0.76) | 0.76 (0.53) | 1.52 (0.51)
  End of treatment: 24-hour mean: number analyzed (Participants) | 80 | 73 | 76 | 78 | 150 | 168
  End of treatment: 24-hour mean | 0.41 (0.65) | 0.63 (0.68) | 1.67 (0.67) | 0.02 (0.66) | 0.85 (0.47) | 1.52 (0.45)
  End of treatment: mean daytime: number analyzed (Participants) | 78 | 67 | 69 | 69 | 137 | 153
  End of treatment: mean daytime | 0.45 (0.74) | 0.37 (0.80) | 2.64 (0.79) | -0.07 (0.79) | 0.32 (0.56) | 1.24 (0.53)
  End of treatment: mean nighttime: number analyzed (Participants) | 88 | 80 | 82 | 82 | 160 | 175
  End of treatment: mean nighttime | 0.39 (0.66) | 0.82 (0.69) | 0.75 (0.68) | 0.45 (0.68) | 1.21 (0.49) | 1.64 (0.47)

62. Secondary Outcome: Change From Baseline to Weeks 4, 12 and EoT in Mean SBP in the Time to Maximum Concentration (Tmax) Window
Description: Vital signs (blood pressure and pulse rate) were monitored using an ABPM device placed on the upper arm followed by intake of the double-blind study medication and worn for at least 24 hours. Tmax (time to maximum concentration) window of mirabegron and solifenacin was from 4-6 hours postdose.
Time Frame: Baseline and weeks 4, 12 and EoT (up to 12 weeks)
Population: ABPMAS participants with available data at each time point were included in the analysis. LOCF was used for EoT.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 92 | 85 | 87 | 86 | 176 | 189
mmHg
  Week 4: number analyzed (Participants) | 77 | 63 | 73 | 72 | 142 | 160
  Week 4 | -2.71 (1.68) | 0.34 (1.86) | -1.03 (1.72) | -1.77 (1.74) | -1.55 (1.23) | -1.47 (1.17)
  Week 12: number analyzed (Participants) | 72 | 60 | 64 | 59 | 130 | 131
  Week 12 | -4.86 (1.78) | -2.13 (1.95) | -1.64 (1.88) | -3.15 (1.96) | -0.26 (1.32) | 0.60 (1.32)
  End of treatment: number analyzed (Participants) | 83 | 75 | 79 | 78 | 157 | 169
  End of treatment | -4.40 (1.60) | -2.19 (1.68) | -1.94 (1.64) | -3.64 (1.65) | -0.61 (1.16) | -0.98 (1.12)

63. Secondary Outcome: Change From Baseline to Weeks 4, 12 and EoT in Mean DBP in the Tmax Window
Description: Vital signs (blood pressure and pulse rate) were monitored using an ABPM device placed on the upper arm followed by intake of the double-blind study medication and worn for at least 24 hours. Tmax window of mirabegron and solifenacin was from 4-6 hours postdose.
Time Frame: Baseline and weeks 4, 12 and EoT (up to 12 weeks)
Population: ABPMAS participants with available data at each time point were included in the analysis. LOCF was used for EoT.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 92 | 85 | 87 | 86 | 176 | 189
mmHg
  Week 4: number analyzed (Participants) | 77 | 63 | 73 | 72 | 142 | 160
  Week 4 | -1.24 (0.84) | 0.09 (0.93) | -0.65 (0.86) | -0.48 (0.87) | -0.22 (0.62) | -0.71 (0.58)
  Week 12: number analyzed (Participants) | 72 | 60 | 64 | 59 | 130 | 131
  Week 12 | -1.74 (0.92) | -0.45 (1.00) | -0.31 (0.97) | -1.49 (1.01) | 0.48 (0.68) | -0.03 (0.68)
  End of treatment: number analyzed (Participants) | 83 | 75 | 79 | 78 | 157 | 169
  End of treatment | -1.85 (0.84) | -0.71 (0.88) | -0.71 (0.85) | -1.22 (0.86) | 0.44 (0.61) | -0.80 (0.59)

64. Secondary Outcome: Change From Baseline to Weeks 4, 12 and EoT in Mean PR in the Tmax Window
Description: as for outcome 63
Time Frame: Baseline and weeks 4, 12 and EoT (up to 12 weeks)
Population: ABPMAS participants with available data at each time point were included in the analysis. LOCF was used for EoT.
Measure: Least Squares Mean (Standard Error); unit: bpm
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 92 | 85 | 87 | 86 | 176 | 189
bpm
  Week 4: number analyzed (Participants) | 77 | 63 | 73 | 72 | 142 | 160
  Week 4 | 0.02 (1.08) | 2.39 (1.19) | 3.68 (1.10) | 0.47 (1.11) | -0.91 (0.79) | 0.67 (0.75)
  Week 12: number analyzed (Participants) | 72 | 60 | 64 | 59 | 130 | 131
  Week 12 | 0.10 (1.10) | 1.22 (1.20) | 1.87 (1.16) | 0.37 (1.21) | 0.15 (0.81) | 1.39 (0.81)
  End of treatment: number analyzed (Participants) | 83 | 75 | 79 | 78 | 157 | 169
  End of treatment | -0.43 (1.05) | 0.82 (1.10) | 3.41 (1.07) | -1.25 (1.08) | 0.34 (0.76) | 1.25 (0.73)

65. Secondary Outcome: Maximum 1-hour Change From Time-matched Baseline in SBP at Weeks 4, 12 and EoT
Description: Vital signs (blood pressure and pulse rate) were monitored using an ABPM device placed on the upper arm followed by intake of the double-blind study medication and worn for at least 24 hours. The maximum 1 hour change from time-matched baseline was calculated as the maximum difference between the post-baseline hourly means and the time-matched baseline hourly means.
Time Frame: Baseline and weeks 4, 12 and EoT (up to 12 weeks)
Population: ABPMAS participants with available data at each time point were included in the analysis. Only participants with an increase (i.e., maximum 1-hour change from time-matched baseline ≥ 0 mmHg) were included in the analysis. LOCF was used for EoT.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 92 | 85 | 87 | 86 | 176 | 189
mmHg
  Week 4: number analyzed (Participants) | 76 | 66 | 67 | 72 | 141 | 157
  Week 4 | 34.05 (2.06) | 31.14 (2.20) | 38.20 (2.19) | 35.16 (2.11) | 32.88 (1.51) | 32.80 (1.43)
  Week 12: number analyzed (Participants) | 67 | 62 | 63 | 60 | 121 | 139
  Week 12 | 33.21 (2.30) | 30.68 (2.38) | 32.88 (2.36) | 35.11 (2.42) | 33.53 (1.70) | 32.82 (1.59)
  End of treatment: number analyzed (Participants) | 80 | 73 | 76 | 78 | 150 | 168
  End of treatment | 34.98 (2.11) | 30.65 (2.20) | 33.53 (2.16) | 34.95 (2.14) | 34.70 (1.54) | 32.55 (1.45)

66. Secondary Outcome: Maximum 1-hour Change From Time-matched Baseline in DBP at Weeks 4, 12 and EoT
Description: Vital signs (blood pressure and pulse rate) were monitored using an ABPM device placed on the upper arm followed by intake of the double-blind study medication and worn for at least 24 hours. Tmax window of mirabegron and solifenacin was from 4-6 hours postdose. The maximum 1 hour change from time-matched baseline was calculated as the maximum difference between the post-baseline hourly means and the time-matched baseline hourly means.
Time Frame: Baseline and weeks 4, 12 and EoT (up to 12 weeks)
Population: as for outcome 65
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 92 | 85 | 87 | 86 | 176 | 189
mmHg
  Week 4: number analyzed (Participants) | 76 | 66 | 67 | 72 | 141 | 157
  Week 4 | 18.78 (1.27) | 19.15 (1.36) | 20.41 (1.35) | 20.02 (1.31) | 20.74 (0.93) | 20.27 (0.88)
  Week 12: number analyzed (Participants) | 67 | 62 | 63 | 60 | 121 | 139
  Week 12 | 19.68 (1.23) | 19.52 (1.28) | 20.41 (1.27) | 21.18 (1.30) | 19.26 (0.92) | 20.01 (0.85)
  End of treatment: number analyzed (Participants) | 80 | 73 | 76 | 78 | 150 | 168
  End of treatment | 20.29 (1.16) | 19.29 (1.22) | 20.71 (1.19) | 20.47 (1.18) | 20.29 (0.85) | 20.36 (0.80)

67. Secondary Outcome: Maximum 1-hour Change From Time-matched Baseline in PR at Weeks 4, 12 and EoT
Description: as for outcome 66
Time Frame: Baseline and weeks 4, 12 and EoT (up to 12 weeks)
Population: as for outcome 65
Measure: Least Squares Mean (Standard Error); unit: bpm
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 92 | 85 | 87 | 86 | 176 | 189
bpm
  Week 4: number analyzed (Participants) | 76 | 66 | 67 | 72 | 141 | 157
  Week 4 | 22.34 (1.35) | 23.86 (1.44) | 25.12 (1.43) | 24.28 (1.38) | 21.48 (0.99) | 21.80 (0.94)
  Week 12: number analyzed (Participants) | 67 | 62 | 63 | 60 | 121 | 139
  Week 12 | 22.63 (1.42) | 23.54 (1.47) | 26.03 (1.46) | 23.52 (1.50) | 22.60 (1.05) | 24.08 (0.98)
  End of treatment: number analyzed (Participants) | 80 | 73 | 76 | 78 | 150 | 168
  End of treatment | 23.01 (1.31) | 24.12 (1.37) | 26.23 (1.34) | 23.33 (1.33) | 22.66 (0.96) | 24.14 (0.90)

68. Secondary Outcome: Change From Baseline to Weeks 4, 12 and EoT in SBP Peak/Trough Difference
Description: Vital signs (blood pressure and pulse rate) were monitored using an ABPM device placed on the upper arm followed by intake of the double-blind study medication and worn for at least 24 hours. Peak/trough difference was defined as the difference between the highest 1-h to lowest 1-h average per participant per visit.
Time Frame: Baseline and weeks 4, 12 and EoT (up to 12 weeks)
Population: ABPMAS participants with available data at each time point were included in the analysis. LOCF was used for EoT.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 92 | 85 | 87 | 86 | 176 | 189
mmHg
  Week 4: number analyzed (Participants) | 76 | 66 | 67 | 72 | 141 | 157
  Week 4 | -0.71 (1.86) | 0.14 (1.99) | -0.69 (1.98) | 0.85 (1.91) | -1.61 (1.36) | 0.41 (1.29)
  Week 12: number analyzed (Participants) | 67 | 62 | 63 | 60 | 121 | 139
  Week 12 | 1.18 (1.98) | -2.45 (2.05) | -4.55 (2.03) | -1.63 (2.08) | 0.68 (1.47) | 0.62 (1.37)
  End of treatment: number analyzed (Participants) | 80 | 73 | 76 | 78 | 150 | 168
  End of treatment | 1.15 (1.83) | -1.38 (1.91) | -2.30 (1.87) | -0.97 (1.85) | 0.25 (1.33) | 0.68 (1.26)

69. Secondary Outcome: Change From Baseline to Weeks 4, 12 and EoT in DBP Peak/Trough Difference
Description: as for outcome 68
Time Frame: Baseline and weeks 4, 12 and EoT (up to 12 weeks)
Population: ABPMAS participants with available data at each time point were included in the analysis. LOCF was used for EoT.
Measure: Least Squares Mean (Standard Error); unit: nnHg
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 92 | 85 | 87 | 86 | 176 | 189
nnHg
  Week 4: number analyzed (Participants) | 76 | 66 | 67 | 72 | 141 | 157
  Week 4 | -0.76 (1.31) | -1.08 (1.40) | -0.20 (1.39) | -1.60 (1.34) | 0.39 (0.96) | -0.56 (0.91)
  Week 12: number analyzed (Participants) | 67 | 62 | 63 | 60 | 121 | 139
  Week 12 | 0.53 (1.30) | 0.15 (1.34) | -1.90 (1.33) | -0.66 (1.36) | -1.24 (0.96) | 0.46 (0.90)
  End of treatment: number analyzed (Participants) | 80 | 73 | 76 | 78 | 150 | 168
  End of treatment | 0.87 (1.23) | 0.27 (1.28) | -0.96 (1.26) | -1.67 (1.24) | -0.98 (0.89) | 0.52 (0.85)

70. Secondary Outcome: Change From Baseline to Weeks 4, 12 and EoT in PR Peak/Trough Difference
Description: as for outcome 68
Time Frame: Baseline and weeks 4, 12 and EoT (up to 12 weeks)
Population: ABPMAS participants with available data at each time point were included in the analysis. LOCF was used for EoT.
Measure: Least Squares Mean (Standard Error); unit: bpm
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 92 | 85 | 87 | 86 | 176 | 189
bpm
  Week 4: number analyzed (Participants) | 76 | 66 | 67 | 72 | 141 | 157
  Week 4 | 1.16 (1.38) | 0.46 (1.48) | 1.54 (1.46) | 0.78 (1.41) | -0.68 (1.01) | -0.51 (0.96)
  Week 12: number analyzed (Participants) | 67 | 62 | 63 | 60 | 121 | 139
  Week 12 | 3.35 (1.45) | -0.04 (1.50) | 1.15 (1.49) | 3.49 (1.53) | -0.53 (1.07) | 1.48 (1.00)
  End of treatment: number analyzed (Participants) | 80 | 73 | 76 | 78 | 150 | 168
  End of treatment | 2.48 (1.32) | 0.45 (1.37) | 1.14 (1.35) | 3.16 (1.33) | -0.02 (0.96) | 1.80 (0.91)

ADVERSE EVENTS:
Time Frame: From first dose of double-blind study drug up to 30 days after last dose of double-blind study drug (up to 16 weeks).
Arm/Group | Placebo | Mirabegron 25 mg | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
All-Cause Mortality (participants affected / at risk) | 0/429 | 0/423 | 0/422 | 0/423 | 0/853 | 0/848
Serious Adverse Events (participants affected / at risk) | 8/429 | 6/423 | 5/422 | 3/423 | 12/853 | 19/848
Other Adverse Events (participants affected / at risk) | 8/429 | 17/423 | 14/422 | 25/423 | 72/853 | 60/848
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=429) | Mirabegron 25 mg (N=423) | Mirabegron 50 mg (N=422) | Solifenacin 5 mg (N=423) | Solifenacin 5 mg + Mirabegron 25 mg (N=853) | Solifenacin 5 mg + Mirabegron 50 mg (N=848)
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Post procedural infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Scrub typhus (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cerebrovascular disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Radiculopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0 | 0
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 2
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hepatitis toxic (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Otorrhoea (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Renal stone removal (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=429) | Mirabegron 25 mg (N=423) | Mirabegron 50 mg (N=422) | Solifenacin 5 mg (N=423) | Solifenacin 5 mg + Mirabegron 25 mg (N=853) | Solifenacin 5 mg + Mirabegron 50 mg (N=848)
Dry mouth (Gastrointestinal disorders) | 8 | 17 | 14 | 25 | 72 | 60

LIMITATIONS AND CAVEATS:
Due to lack of data integrity, one site's data was not included in the efficacy and safety analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript at least 45 days prior to publication for review and comment. Sponsor may delay the publication temporarily to seek patent protection or permanently withhold the publication.